Replication of the RECOVER-II Anticoagulant Trial in Healthcare Claims

Data NCT04735523

January 25, 2021

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Treatment of Acute Venous Thromboembolism with Dabigatran or Warfarin (RECOVER II)

#### 1.2 Intended aim(s)

To compare the risk of symptomatic, recurrent venous thromboembolism (VTE) in patients with symptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE) for dabigatran 150 mg versus warfarin.

### 1.3 Primary endpoint for replication

The primary outcome of the study was symptomatic, recurrent VTE or death related to VTE

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a primary event rate of 2% at 6 months follow-up and with a noninferiority margin of 2.75, it was determined that 2,550 patients would be needed to capture at least 46 events and achieve 90% power to conclude noninferiority of dabigatran over standard therapy at one-sided alpha level of 0.025.

### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; RR= 0.69 (95% CI 0.36-1.32)

### 1.6 Trial estimate

RR = 1.08 (95% CI 0.64-1.80) comparing dabigatran vs warfarin (Schulman et al., 2014)

## 2. Person responsible for implementation of replication in Aetion

Dureshahwar Jawaid, MPH implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum, MarketScan, Medicare

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.



#### 5. Cohort Identification

### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing dabigatran to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of dabigatran to warfarin (index date). We will restrict the analyses to patients with a diagnosis of proximal DVT or PE.

### 5.2 Important steps for cohort formation

New use of dabigatran, exposure, and warfarin, comparator, is defined as no use in 180 days prior to index date.

#### 5.2.1 Eligible cohort entry dates

Market availability of dabigatran in the U.S. for treatment of deep vein thrombosis and pulmonary embolism started on April 7, 2014

- For Medicare: April 7, 2014 December 31, 2017 (end of available data)
- For Marketscan: April 7, 2014 December 31, 2018 (end of available data)
- For Optum: April 7, 2014 March 31, 2020 (end of available data)

## 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date.

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining Patients |
| All patients | | 77,673,639 | | 200,203,908 | | 6,886,908 |
| Did not meet cohort entry criteria | -<br>77,124,704 | 548,935 | -<br>199,725,626 | 478,282 | -4,396,002 | 2,490,906 |

| Excluded due to insufficient enrollment | -67,201 | 481,734 | -36,281 | 442,001 | -52,122 | 2,438,784 |
|---|---|---|---|---|---|---|
| Excluded due to prior use of referent | -378,710 | 103,024 | -331,731 | 110,270 | -1,924,222 | 514,562 |
| Excluded due to prior use of exposure | -30,781 | 72,243 | -35,333 | 74,937 | -163,530 | 351,032 |
| Excluded because patient qualified in >1 exposure category | -3 | 72,240 | -1 | 74,936 | -9 | 351,023 |
| Excluded based on Age (<65 - Medicare only) | - | - | - | - | -36484 | 314,539 |
| Excluded based on Age (Missing) | 0 | 72,240 | 0 | 74,936 | -105 | 314,434 |
| Excluded based on Gender | 0 | 72,240 | 0 | 74,936 | 0 | 314,434 |
| Excluded based on Use of other NOACs ( Rivaroxaban, Apixaban, edoxaban) | -4,797 | 67,443 | -3163 | 71,773 | -17983 | 296,451 |
| Excluded based on Inclusion # 1 - Age <= 18 | -41 | 67,402 | -76 | 71,697 | 0 | 296,451 |
| Excluded based on Inclusion # 2 - VTE | -49,506 | 17,896 | -48,049 | 23,648 | -211,430 | 85,021 |
| Excluded based on Exclusion # 2 | -618 | 17,278 | -389 | 23,259 | -2,123 | 82,898 |
| Excluded based on Exclusion # 3 - caval filter | -257 | 17,021 | -294 | 22,965 | -971 | 81,927 |
| Excluded based on Exclusion # 4 - major bleeding | -1,096 | 15,925 | -836 | 22,129 | -3836 | 78,091 |
| Excluded based on Exclusion # 5 - Anemia | -886 | 15,039 | -952 | 21,177 | -4,786 | 73,305 |
| Excluded based on Exclusion # 7 - unstable CVD | -385 | 14,654 | -221 | 20,956 | -1,015 | 72,290 |
| Excluded based on Exclusion # 9 - End-stage liver disease | -370 | 14,284 | -315 | 20,641 | -1,037 | 71,253 |
| Excluded based on Exclusion # 10 - Severe renal impairment | -1,088 | 13,196 | -741 | 19,900 | -3,745 | 67,508 |
| Excluded based on Exclusion # 11d - Active infective endocarditis | -2 | 13,194 | -1 | 19,899 | -4 | 67,504 |
| Excluded based on Exclusion # 11e - Heart valve | -17 | 13,177 | -78 | 19,821 | -202 | 67,302 |
| Excluded based on Exclusion # 12 - Pregnancy | -32 | 13,145 | -58 | 19,763 | -2 | 67,300 |
| Excluded based on Exclusion # 13 - drug induced liver disease | 0 | 13,145 | 0 | 19,763 | 0 | 67,300 |
| Excluded based on Exclusion # 14a - alcohol/drug abuse | -138 | 13,007 | -113 | 19,650 | -198 | 67,102 |
| Excluded based on CCI (180 days)- ICD9 and ICD10 v2 | -41 | 12,966 | -23 | 19,627 | -73 | 67,029 |
| Final cohort | | 12,966 | | 19,627 | | 67,029 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### 6. Variables

### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of dabigatran. New initiation will be defined by no use of dabigatran or warfarin in the prior 6 months before treatment initiation (washout period).

#### Comparator:

New initiators of warfarin, defined by no use of dabigatran or warfarin in the prior 6 months.

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest: (definitions provided in **Appendix A**):

Primary Outcome: VTE and cause-specific mortality

Secondary Outcome: Individual components

- Hospital admission for VTE (principal diagnosis position)
- Cause-specific mortality
  - Inpatient mortality identified using discharge status codes from hospitalization for VTE

### Safety outcome of interest:

1. Major bleeding

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of dabigatran and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (dabigatran and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from dabigatran to rivaroxaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 180 days.

## 7. Initial Feasibility Analysis

### Aetion report name:

For dabigatran vs. warfarin

Optum- https://bwh-dope.aetion.com/projects/details/1500/results/62528/result/0

MarketScan- https://bwh-dope.aetion.com/projects/details/1501/results/62529/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/1499/results/63197/result/0

Date conducted: 12/9/2020 (Medicare 12/23/20)

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population FEASIBILITY- FOR STUDY OUTCOME
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

## Aetion report name:

For dabigatran vs. warfarin

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1500/results/62531/result/0">https://bwh-dope.aetion.com/projects/details/1500/results/62531/result/0</a>

 $Market S can- \underline{https://bwh-dope.aetion.com/projects/details/1501/results/62532/result/0}$ 

Medicare- https://bwh-dope.aetion.com/projects/details/1499/results/63198/result/0

Date conducted: 12/9/2020 (Medicare 12/23/20)

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 11/18/2020 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 11/29/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

### **Aetion report links:**

Optum: https://bwh-dope.aetion.com/projects/details/1500/results/62793/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/1501/results/62794/result/0
Medicare: https://bwh-dope.aetion.com/projects/details/1499/results/63201/result/0

Date conducted: 12/16/20 (Medicare 12/23/20)

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 47 (0.88%) | 24 (0.90%) | 23 (0.86%) |
| Death | 91 (1.70%) | 54 (2.02%) | 37 (1.38%) |
| Start of an additional exposure | 105 (1.96%) | 18 (0.67%) | 87 (3.25%) |
| End of index exposure | 3,523 (65.85%) | 1,724 (64.45%) | 1,799 (67.25%) |
| Specified date reached | 562 (10.50%) | 269 (10.06%) | 293 (10.95%) |
| End of patient enrollment | 217 (4.06%) | 109 (4.07%) | 108 (4.04%) |
| Switch to NOACs + nursing home admission | 805 (15.05%) | 477 (17.83%) | 328 (12.26%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Marketscan Medicare | | | |
| Overall Patient Population | 84 [38-176] | 88.5 [38-163] | 84 [38-164] |
| Referent | 79 [38-156] | 82 [38-160] | 89 [38-168] |
| Exposure | 93 [38-188] | 92 [38-171] | 77[38-157] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 8.11 | 14.8 | 19.67 | 17.19 |

### 10. Final Power Assessment

## Date conducted: 12/16/20

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

### o Pooled

| © 10012G | |
|----------------------------|-------------|
| Non-inferiority Analysis | |
| Number of patients matched | |
| Reference | 2,675 |
| Exposed | 2,675 |
| Risk per 1,000 patients | 17.19 |
| HR from RCT | 1.08 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2.75 |
| Number of events expected | 91.9665 |
| Power | 0.994158797 |

o Optum

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| Reference | 387 |
| Exposed | 387 |
| Risk per 1,000 patients | 8.11 |
| HR from RCT | 1.08 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2.75 |
| Number of events expected | 6.27714 |
| Power | 0.215017932 |

### Marketscan

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| Reference | 711 |
| Exposed | 711 |
| Risk per 1,000 patients | 14.80 |
| HR from RCT | 1.08 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2.75 |
| Number of events expected | 21.0456 |
| Power | 0.572949662 |

## Medicare

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Non-inferiority Analysis | |
|----------------------------|------------|
| Number of patients matched | |
| Reference | 1,577 |
| Exposed | 1,577 |
| Risk per 1,000 patients | 19.67 |
| HR from RCT | 1.08 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2.75 |
| Number of events expected | 62.03918 |
| Power | 0.95736364 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 12/24/2020 |
|-------------------------|--------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 01/18/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <a href="Google Form">Google Form</a>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study

Effectiveness research with Real World Data to support FDA's regulatory decision making

variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

## 12. Register study protocol on clinicalTrials.gov

### Date conducted:

• Register the study on clinicalTrials.gov and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

## **14. Requested Results**

## 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

## 14.2 Table 2: Follow-up time

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

## 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

## 14.4 Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

## 14.5 <u>Table 5: Results from secondary analyses;</u>

Effectiveness research with Real World Data to support FDA's regulatory decision making

## 15. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Schulman S, Kakkar AK, Goldhaber SZ, et al. Treatment of Acute Venous Thromboembolism With Dabigatran or Warfarin and Pooled Analysis. Circulation. 2014;129:764–772

| | # RE-COVER II trial definitions | | Implementation in routine care | References | Notes | Color coding |
|---|---|---|---|---|---|---|
| F | | | ; Unintended S with label change | | | Can be replicated in claims Using dummy definitions for measuring in claims |
| F | | EXPOSURE v kxed doses of dabigatran (150 mg twice daily) vs. adjusted-dose warfarin | Exposure | | | |
| | C | oncomitant Medications: Low molecular weight heparin (89%), fondaparinux (2%), and aspirin (9%) | dabigatran Referent | | | |
| F | _ | | warfarin | | | Can't be measured in claims Can't be measured in claims but not important |
| F | - | PRIMAR | Y OUTCOME | | | for the analysis |
| | fr | ecurrent Symptomatic Venous Thromboembolism (VTE) and Deaths Related to VTE [ Time Frame: For statistical analysis 1 om randomisation to end of post treatment period (ptp), planned to be up to day 224. For statistical analysis 2: from indomisation to 6 months (up to day 180) ] | Measured 1 day after drug initiation in primary diagnosis position inpatient care setting VTE codes (see excel sheet RECOVER outcome VTE) | Fang MC, Fan D, Sung SH, et al. Validity of Using Inpatient and<br>Outpatient Administrative Codes to Identify Acute Venous<br>Thromboembolism: The CVRN VTE Study, Med Care. 2017;55(12):e137-<br>e143. Codes for pregnancy-related VTE and superficial thrombophlebitis were<br>not included. | | |
| - | - | INCLUSI | N CRITERIA Measured on the day of drug initiation | | | |
| | 1 A | ge ≥18 years | Measured on the day of orug initiation Age >18 | | | |
| | 2 <sup>a</sup> | cute deep vein thrombosis (DVT) of the leg involving proximal veins, and/or pulmonary embolism (PE) lin patients for whon<br>I least 6 months of anticoagulant therapy is considered appropriate. E and DVT were objectively verified by: Compression ultrasonography, Venography of legs, V/Q scanning, Angiography or CT<br>ngiography | micasured so days derive the day or drug initiation any diagnosis position | | | |
| L | 3 W | /ritten informed consent | N/A | | | |
| H | - | EXCLUSI | ON CRITERIA | | | |
| | 10 | vert symptoms of VTE for longer than 2 weeks prior to enrolment | N/A | | | |
| | | vert symptoms of VTE for longer than 2 weeks prior to enrolment E satisfying at least one of the following criteria: | N/A Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism ICD-9 diagnosis: 415.1x (already in inclusion criteria 2) | | The inclusion and exclusion criteria were the same as previously described [RECOVER I] except that baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal for patients to be excluded. "Schulman S, Kakkar AK, Goldhaber SZ, et al. Treatment of Acute Venous Thromboembolism with Dablgatran or Warfaria and Poole Analysis. Circulation. 2014;129:764-772 Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the oriteria described in RECOVER I to construct our list of criteria for trial emulation. | |
| 22 | 2 P | | Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism | | baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal<br>for patients to be excluded. "Schulman S, Kalkar AK, Goldhaber SZ, et al. Treatment of Acute Venous<br>Thromboembolism With Dabgarran or Warfarin and Pooled Analysis. Circulation. 2014;129:764–772<br>Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the | |
| 2a | 2 Pl | E satisfying at least one of the following criteria: | Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism ICD-9 diagnosis: 415.1x (already in inclusion criteria 2) | | baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal<br>for patients to be excluded. "Schulman S, Kalkar AK, Goldhaber SZ, et al. Treatment of Acute Venous<br>Thromboembolism With Dabgarran or Warfarin and Pooled Analysis. Circulation. 2014;129:764–772<br>Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the | |
| 22 2h | 2 Pl | E satisfying at least one of the following criteria: aemodynamic instability, | Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism ICD-9 diagnosis: 415.1x (already in inclusion criteria 2) N/A (mostly captured by the criteria 2b-2c and 3) Thrombactomy. ICD-9 procedure: 39.74 ICD-9 procedure: 39.74 ICD-9 procedure: 30.632Z, 03G64ZZ, 03G64ZZ, 03G4ZZ, 03G4ZZ, 03G63ZZ, 03GAZZ, 0 | | baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal<br>for patients to be excluded. "Schulman S, Kalkar AK, Goldhaber SZ, et al. Treatment of Acute Venous<br>Thromboembolism With Dabgarran or Warfarin and Pooled Analysis. Circulation. 2014;129:764–772<br>Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the | |
| 28 | 2 Pl | E satisfying at least one of the following criteria: semodynamic instability, R Embolectomy is indicated or performed, | Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism ICD-9 diagnosis: 415.1x (already in inclusion criteria 2) N/A (mostly captured by the criteria 2b-2c and 3) Thrombectomy. ICD-9 procedure: 39.74 ICD-10 procedure: 39.74 ICD-10 procedure: 30.73 ICD-1 | | baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal for patients to be excluded." Schulman S, Kalkar AK, Goldber SZ, et al. Teatment of Acute Venous Thromboembolism With Dablgaran or Warfarin and Pooled Analysis. Circulation. 2014;129:764-772 Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the oriteria described in RECOVER 1 to construct our list of criteria for trial emulation. Not indicated by FDA for PE: Reteplase (Returase) Terrencetplase (TRIASE) | |
| 2 t | 2 Pl | E satisfying at least one of the following criteria: semodynamic instability, R Embolectomy is indicated or performed, | Measured 30 days before the day of drug initiation any diagnosis position Pulmonary embolism ICD-9 diagnosis: 415.1x (already in inclusion criteria 2) N/A (mostly captured by the criteria 2b-2c and 3) Thrombectomy. ICD-9 procedure: 39.74 ICD-9 procedure: 39.74 ICD-10 procedure: 39.73 ICD-10 procedure: 39.73 ICD-10 procedure: 39.73 ICD-10 procedure: 39.73 ICD-10 procedure: 39.73 ICD-10 procedure: 39.74 ICD-10 procedure: 39.73 ICD-10 procedure: 39.73 ICD-10 procedure: 39.74 ICD | | baseline aminotransferases had to exceed 3 times rather than 2 times the local upper limit of the normal for patients to be excluded." Schulman S, Kalkar AK, Goldber SZ, et al. Teatment of Acute Venous Thromboembolism With Dablgaran or Warfarin and Pooled Analysis. Circulation. 2014;129:764-772 Seeing as the exclusion criteria were declared to be the same for the two trials, we also referred to the oriteria described in RECOVER 1 to construct our list of criteria for trial emulation. Not indicated by FDA for PE: Reteplase (Returase) Terrencetplase (TRIASE) | |

| | | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting | | |
|---|---|---|---|---|
| 5 | Known anaemia | Anemia (non-deficiency/neoplastic/chemotherapy/hemorrhagic assoicated) | | |
| | | ICD-9 diagnosis: 282.x, 283.x, 284.x, 285.x<br>ICD-10 diagnosis: D55 - D62, D63.0 | | |
| 6 | Need of anticoagulant treatment for disorders other than VTE | N/A | | |
| | | Measured 30 days before the day of drug initiation any diagnosis position and inpatient or outpatient care setting | | |
| | | Unstable angina:<br>ICD-9: 411.x | | |
| 7 | Recent unstable cardiovascular disease | ICD-10: I24.1x, I20.0x, I25.1x, I25.7x, I24.0x, I24.8x, I24.9x | | |
| | | MI<br>ICD-9: 410.x except 410.x2<br>Stroke | | |
| | | (CD-9: 430.xx, 431.xx, 433.x1, 434.xx, 436.x<br>IIIA<br>ICD-9: 435.xx | | |
| | | ICD-9: 435.xx | | |
| 8 | Elevated AST or ALT > 3x ULN | N/A | | |
| | | | "A coding algorithm combining ICD-9-CM codes for cirrhosis and hepatic decompensation events, with or without ICD-9-CM codes for a chronic liver disease, can identify patients with end-stage liver disease" | |
| | | Measured 180 days before the day of drug initiation any diagnosis position and inpatient or outpatient care setting | Goldberg D, Lewis J, Halpern S, Weiner M, Lo Re V 3rd. Validation of three coding algorithms to identify patients with end-stage liver disease | |
| | | Model for end-stage liver disease: | Jul;21(7):765-769. doi: 10.1002/pds.3290. Epub 2012 Jul 4. PMID: | |
| | | Cirrhosis: | 22674685; PMCID: PMC4267226. | |
| 1 | | ICD-9 codes: 571.2 (alcoholic cirrhosis), 571.5 (cirrhosis without mention of alcohol, 571.6 (billiary cirrhosis). | | |
| 9 | Liver disease expected to have any potential impact on survival (severe liver conditions) | Hepatic decompensation:<br>ICD-9 codes: 456.0, 456.20 (esophageal varices with bleeding); 456.1, 456.21 (esophageal varices without bleeding); 789.5,<br>789.59 (ascites); 572.2 (hepatic coma)) 567.0, 567.2, 567.21, 567.21, | | |
| | | 567.29, 567.8, 567.89, 567.9 (peritonitis); 572.4 (hepatorenal syndrome) | | |
| | | HCC and other malignant liver cancers: ICD-9 codes: 155.x | | |
| | | ICD-10 codes: C22.x | | |
| | | Measured 180 days before the day of drug initiation any diagnosis position and inpatient or outpatient care setting | | |
| | | CKD stage 4/5/ESRD:<br>ICD-9: 585.4x, 585.5x, 585.6x | | |
| 10 | Severe renal impairment | ICD-10: N18.4x, N18.5x, N18.6x | | |
| | | Dalysis/ Renal transplant:<br>codes are in the sheet "Dialysis and Renal Transplant" | | |
| 11 | Contraindications to anticoagulant therapy (not specified) | mostly captured in criteria 4 | | |
| 11a | Recent or active major bleeding | see criteria 4 | | |
| 11b | Recent brain, eye, or spinal cord injury or surgery; | see criteria 4 | | |
| 11c | malignant or severe, uncontrolled hypertension | see criteria 4 | | |
| | | Measured 45 days prior to drug initiation in any diagnosis setting, any position: | | |
| 11d | Active infective endocarditis | Infective endocarditis ICD-9 codes: 421.x | | |
| | | ICD-10 codes: I33.x | | |
| | | Measured 90 days prior to drug initiation in in patient, inpatient setting, any position | | |
| | | Heart Valve<br>ICD-9 codes: | | |
| | | V42.2 (heart valve replaced by transplant) V43.3 (heart valve replaced by a mechanical device/prosthesis) | | |
| | | CPT codes: | | |
| | | 33660-33665 (atrioventricular valve repair) 33400-33403 (aortic valve valvuloplasty) | | |
| 11e | Mechanical prosthetic heart valve (recently implanted - RE-ALIGN trial) | 33405 (Replacement, aortic valve, with cardiopulmonary bypass; with prosthetic valve other than homograft or stentless valve) | | |
| | | 33420-33430 (mitral valve repair/valvuloplasty/replacement) 33460 (valvectomy, tricuspid valve, with cardiopulmonary bypass) | | |
| | | 33463-33468 (tricuspid valve repair/valvuloplasty/replacement) 33475 (replacement, pulmonary valve) 33496 (prosthetic valve dysfunction repair) | | |
| | | 33496 (prosthetic valve dystrunction repair) 0257T (implantation of catheter-delivered prosthetic aortic heart valve; open thoracic approach) 0258T (transthoracic cardiac exposure for catheter-delivered aortic valve replacement without cardiopulmonary bypass) | | |
| | | 102-bit (transtronacic caroiac exposure for catheter-oeilwerea aortic valve replacement; without carolopulmonary dypass) 0259T (transtronacic caroiac exposure for catheter-delilvered aortic valve replacement; with cathopulmonary bypass) 0262T (implantation of catheter-delilvered prosthetic pulmonary valve, endovascular approach) | | |
| <u> </u> | | ococi (impanitution oi cataccet-uenvereu prostrette printiniary varve, enauvascular approach) | | |
| 12 | Women who are pregnant, nursing, or of childbearing potential who refuse to use a medically acceptable form of contraception | see excel "Pregnancy" | | |
| | | | 1 | 1 |

| 13 Patients who have developed transaminase elevations upon exposure to ximelagatran | Measured 30 days before the day of drug initiation any diagnosis position <u>Drus: induced liver disease</u> AND <u>ximelagatran</u> (CD-10: K71.9 - Toxic liver disease (drug induced disorder of liver) |
|---|---|
| 14 Patients considered unsuitable for inclusion by the investigator | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting CCI >= 10. (life expectancy less than the expected duration of the trial) or Alcohol abuse or dependence (any position any setting) ICD 9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x (CMS has not released mapping for new ICDIO for this code), 171.3x ICD-10 diagnosis: F10.x, ICDx, G62.1, 142.6, 099.31x Unus abuse or dependence (any position, any setting) 1292.xx, 301.xx, 302.xx, 303.xx, 868.3x 965.0x, 967.xx, 969.4x-969.6x, 969.72-969.79, 970.81 CD-10 diagnosis: F11.xx, F12.xx, F13.xx, F13.xx, F13.xx, F13.xx, G62.0x, 969.32x Unus abuse or dependence (any position, any setting) |
| 15 Patients who in the investigators opinion should not be treated with warfarin | |
| 16 Allergy to heparins or other alternate approved therapy used for initial treatment, warfarin or dabigatran, or to one of the excipients included in these medications | |
| 17 Participation in another clinical trial with an investigational drug during the last 30 days or previous participation in this stu | dy |

| <u>Trial ID</u> | |
|---|---|
| Trial Name (with web links) | <u>RE-COVER II</u> |
| Trial Name (with pdf links) | |
| <u>NCT</u> | NCT00680186 |
| Therapeutic Area | Cardiology/Vascular Diseases |
| <u>Study Batch</u> | NOACs |
| <u>Brand Name</u> | Pradaxa |
| <u>Generic Name</u> | dabigatran etexilate |
| <u>Year</u> | 2013 |
| Measurable Endpoint | recurrent venous thromboembolism |
| <u>Exposure</u> | dabigatran etexilate |
| <u>Comparator</u> | warfarin |
| <u>Population</u> | |
| <u>Trial Finding</u> | 1.08 (95% CI 0.64–1.80) |
| No. of Patients | Dabigatran (n=1280) |
| | Warfarin (n=1288) |
| Non-inferiority Margin | 2.75 |
| Assay Sens. Endpoint | |
| Assay Sens. Finding | |
| <u>Power</u> | 90% power- "We determined the sample size on the basis of an expected rate of recurrent VTE of 2% in each group during 6 months,2,13,14 while requiring a power of 90% to exclude a hazard ratio of 2.75, an absolute risk increase of 3.6 percentage points for the primary outcome with dabigatran, and a 1-sided $\alpha$ level of 0.025" Schulman S, Kakkar AK, Goldhaber SZ, et al. Treatment of Acute Venous Thromboembolism With Dabigatran or Warfarin and Pooled Analysis. Circulation. 2014;129:764–772 |


| 180.253 | bilateral |
|---|---|
| 180.259 | Phlebitis and thrombophlebitis of unspecified calf muscular vein |
| 180.29 | Phlebitis and thrombophlebitis of other deep vessels of lower extremities |
| 180.291 | Phlebitis and thrombophlebitis of other deep vessels of right lower extremity |
| 180.292 | Phlebitis and thrombophlebitis of other deep vessels of left lower extremity |
| 180.293 | Phlebitis and thrombophlebitis of other deep vessels of lower extremity, bilate |
| 180.299 | Phlebitis and thrombophlebitis of other deep vessels of unspecified lower extre |
| 180.3 | Phlebitis and thrombophlebitis of lower extremities, unspecified |
| 182.4 | Acute embolism and thrombosis of deep veins of lower extremity |
| 182.40 | Acute embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.401 | Acute embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.402 | Acute embolism and thrombosis of unspecified deep veins of left lower extremity |
| 182.403 | bilateral |
| 182.409 | Acute embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| 182.41 | Acute embolism and thrombosis of femoral vein |
| 182.411 | Acute embolism and thrombosis of right femoral vein |
| 182.412 | Acute embolism and thrombosis of left femoral vein |
| 182.413 | bilateral |
| 182.419 | Acute embolism and thrombosis of unspecified femoral vein |
| 182.42 | Acute embolism and thrombosis of iliac vein |
| 182.421 | Acute embolism and thrombosis of right iliac vein |
| 182.422 | Acute embolism and thrombosis of left iliac vein |
| 182.423 | bilateral |
| 182.429 | Acute embolism and thrombosis of unspecified iliac vein |
| 182.43 | Acute embolism and thrombosis of popliteal vein |
| 182.431 | Acute embolism and thrombosis of right popliteal vein |
| 182.432 | Acute embolism and thrombosis of left popliteal vein |
| 182.433 | bilateral |
| 182.439 | Acute embolism and thrombosis of unspecified popliteal vein |
| 182.44 | Acute embolism and thrombosis of tibial vein |
| 182.441 | Acute embolism and thrombosis of right tibial vein |
| 182.442 | Acute embolism and thrombosis of left tibial vein |
| 182.443 | bilateral |

| 182.45 Acute embolism and thrombosis of peroneal vein | 182.449 | Acute embolism and thrombosis of unspecified tibial vein |
|---|---|---|
| 182.452 Acute embolism and thrombosis of left peroneal vein | 182.45 | Acute embolism and thrombosis of peroneal vein |
| 182.453 bilateral | 182.451 | Acute embolism and thrombosis of right peroneal vein |
| 182.459 Acute embolism and thrombosis of unspecified peroneal vein | 182.452 | Acute embolism and thrombosis of left peroneal vein |
| 182.46 Acute embolism and thrombosis of calf muscular vein 182.461 Acute embolism and thrombosis of right calf muscular vein 182.462 Acute embolism and thrombosis of left calf muscular vein 182.463 bilateral 182.469 Acute embolism and thrombosis of unspecified calf muscular vein 182.491 Acute embolism and thrombosis of other specified deep vein of lower extremity 182.492 Acute embolism and thrombosis of other specified deep vein of right lower extremity 182.493 Acute embolism and thrombosis of other specified deep vein of left lower extremity 182.499 Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity 182.491 Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity 182.492 Acute embolism and thrombosis of unspecified deep vein of unspecified lower extremity 182.493 Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity 182.474 Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity 182.475 Acute embolism and thrombosis of unspecified deep veins of listal lower extremity 182.476 Acute embolism and thrombosis of unspecified deep veins of distal lower extremity 182.477 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity 182.480 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity 182.470 Acute embolism and thrombosis of unspecified deep veins of lower extremity 182.481 Acute embolism and thrombosis of unspecified deep veins of lower extremity 182.492 Acute embolism and thrombosis of unspecified deep veins of lower extremity 182.503 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.504 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.505 Chronic embolism and thrombosis of unspecified deep veins of lower extremity | 182.453 | bilateral |
| 182.461 Acute embolism and thrombosis of right calf muscular vein 182.462 Acute embolism and thrombosis of left calf muscular vein 182.463 bilateral 182.469 Acute embolism and thrombosis of unspecified calf muscular vein 182.491 Acute embolism and thrombosis of other specified deep vein of lower extremity 182.492 Acute embolism and thrombosis of other specified deep vein of right lower extremity 182.493 bilateral 182.499 Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity 182.491 Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity 182.492 Acute embolism and thrombosis of unspecified deep vein of unspecified lower extremity 182.493 Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity 182.494 Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity 182.475 Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity 182.490 Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity 182.491 Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity 182.422 Acute embolism and thrombosis of unspecified deep veins of light distal lower extremity 182.423 bilateral 182.429 Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity 182.500 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.501 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.502 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.503 bilateral 182.509 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.509 Chronic embolism and thrombosis of unspecified deep veins of lower extremity | 182.459 | Acute embolism and thrombosis of unspecified peroneal vein |
| 182.462 Acute embolism and thrombosis of left calf muscular vein 182.463 bilateral 182.469 Acute embolism and thrombosis of unspecified calf muscular vein 182.491 Acute embolism and thrombosis of other specified deep vein of lower extremity 182.492 Acute embolism and thrombosis of other specified deep vein of right lower extremity 182.493 bilateral 182.499 Acute embolism and thrombosis of other specified deep vein of left lower extremity 182.491 Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity 182.492 Acute embolism and thrombosis of unspecified deep vein of unspecified lower extremity 182.493 Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity 182.494 Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity 182.495 Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity 182.496 Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity 182.497 Acute embolism and thrombosis of unspecified deep veins of listal lower extremity 182.421 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity 182.422 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity 182.423 bilateral 182.429 Acute embolism and thrombosis of unspecified deep veins of lower extremity 182.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.501 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.502 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.503 Chronic embolism and thrombosis of unspecified deep veins of lower extremity | 182.46 | Acute embolism and thrombosis of calf muscular vein |
| 182.463 | 182.461 | Acute embolism and thrombosis of right calf muscular vein |
| 182.469 Acute embolism and thrombosis of unspecified calf muscular vein 182.49 | 182.462 | Acute embolism and thrombosis of left calf muscular vein |
| Recute embolism and thrombosis of other specified deep vein of lower extremity | 182.463 | bilateral |
| Results | 182.469 | Acute embolism and thrombosis of unspecified calf muscular vein |
| Received the second content of the specified deep vein of left lower extremity | 182.49 | Acute embolism and thrombosis of other specified deep vein of lower extremity |
| 182.493 bilateral182.499Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity182.4YAcute embolism and thrombosis of unspecified deep veins of proximal lower extremity182.4Y1Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity182.4Y2Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity182.4Y3 bilateral182.4Y9Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity182.4ZAcute embolism and thrombosis of unspecified deep veins of distal lower extremity182.4Z1Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity182.4Z2Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity182.4Z3 bilateral182.4Z9Acute embolism and thrombosis of unspecified deep veins of lower extremity182.5Chronic embolism and thrombosis of unspecified deep veins of lower extremity182.50Chronic embolism and thrombosis of unspecified deep veins of lower extremity182.501Chronic embolism and thrombosis of unspecified deep veins of light lower extremity182.502Chronic embolism and thrombosis of unspecified deep veins of left lower extremity182.503 bilateral182.509Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.491 | Acute embolism and thrombosis of other specified deep vein of right lower extremity |
| Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremit Acute embolism and thrombosis of unspecified deep veins of distal lower extremity Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity Chronic embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity | 182.492 | Acute embolism and thrombosis of other specified deep vein of left lower extremity |
| Result R | 182.493 | bilateral |
| Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity | 182.499 | Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity |
| Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity bilateral Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremit Acute embolism and thrombosis of unspecified deep veins of distal lower extremity Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity Acute embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of right lower extremity Chronic embolism and thrombosis of unspecified deep veins of right lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity | 182.4Y | Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| 182.4Y3 | 182.4Y1 | Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity R2.4Z1 Acute embolism and thrombosis of unspecified deep veins of distal lower extremity R2.4Z1 Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity R2.4Z2 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity R2.4Z3 bilateral R2.4Z9 Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity R2.5 Chronic embolism and thrombosis of deep veins of lower extremity R2.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity R2.501 Chronic embolism and thrombosis of unspecified deep veins of right lower extremity R2.502 Chronic embolism and thrombosis of unspecified deep veins of left lower extremity R2.503 bilateral R2.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Y2 | Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| Acute embolism and thrombosis of unspecified deep veins of distal lower extremity 182.4Z1 Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity 182.4Z2 Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity 182.4Z3 bilateral 182.4Z9 Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity 182.5 Chronic embolism and thrombosis of deep veins of lower extremity 182.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.501 Chronic embolism and thrombosis of unspecified deep veins of right lower extremity 182.502 Chronic embolism and thrombosis of unspecified deep veins of left lower extremity 182.503 bilateral 182.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Y3 | bilateral |
| Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity I82.4Z3 bilateral I82.4Z9 Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity I82.5 Chronic embolism and thrombosis of deep veins of lower extremity I82.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity I82.501 Chronic embolism and thrombosis of unspecified deep veins of right lower extremity I82.502 Chronic embolism and thrombosis of unspecified deep veins of left lower extremity I82.503 bilateral I82.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Y9 | Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| 182.422Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity182.423 bilateral182.429Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity182.5Chronic embolism and thrombosis of deep veins of lower extremity182.50Chronic embolism and thrombosis of unspecified deep veins of lower extremity182.501Chronic embolism and thrombosis of unspecified deep veins of right lower extremity182.502Chronic embolism and thrombosis of unspecified deep veins of left lower extremity182.503 bilateral182.509Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Z | Acute embolism and thrombosis of unspecified deep veins of distal lower extremity |
| 182.423 bilateral182.429Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity182.5Chronic embolism and thrombosis of deep veins of lower extremity182.50Chronic embolism and thrombosis of unspecified deep veins of lower extremity182.501Chronic embolism and thrombosis of unspecified deep veins of right lower extremity182.502Chronic embolism and thrombosis of unspecified deep veins of left lower extremity182.503 bilateral182.509Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Z1 | Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity 182.5 Chronic embolism and thrombosis of deep veins of lower extremity 182.50 Chronic embolism and thrombosis of unspecified deep veins of lower extremity 182.501 Chronic embolism and thrombosis of unspecified deep veins of right lower extremity 182.502 Chronic embolism and thrombosis of unspecified deep veins of left lower extremity 182.503 bilateral 182.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.4Z2 | Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| Chronic embolism and thrombosis of deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of right lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity Expectation of the second of | 182.4Z3 | bilateral |
| Chronic embolism and thrombosis of unspecified deep veins of lower extremity Chronic embolism and thrombosis of unspecified deep veins of right lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity Expectation of the second of the secon | 182.4Z9 | Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |
| Chronic embolism and thrombosis of unspecified deep veins of right lower extremity Chronic embolism and thrombosis of unspecified deep veins of left lower extremity Lack Solution So | 182.5 | Chronic embolism and thrombosis of deep veins of lower extremity |
| 182.502Chronic embolism and thrombosis of unspecified deep veins of left lower extremity182.503 bilateral182.509Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.50 | Chronic embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.503 bilateral 182.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.501 | Chronic embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.509 Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity | 182.502 | Chronic embolism and thrombosis of unspecified deep veins of left lower extremity |
| | 182.503 | bilateral |
| 182.51 Chronic embolism and thrombosis of femoral vein | 182.509 | Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| | 182.51 | Chronic embolism and thrombosis of femoral vein |

| 182.511 | Chronic embolism and thrombosis of right femoral vein |
|---|---|
| 182.512 | Chronic embolism and thrombosis of left femoral vein |
| 182.513 | bilateral |
| 182.519 | Chronic embolism and thrombosis of unspecified femoral vein |
| 182.52 | Chronic embolism and thrombosis of iliac vein |
| 182.521 | Chronic embolism and thrombosis of right iliac vein |
| 182.522 | Chronic embolism and thrombosis of left iliac vein |
| 182.523 | bilateral |
| 182.529 | Chronic embolism and thrombosis of unspecified iliac vein |
| 182.53 | Chronic embolism and thrombosis of popliteal vein |
| 182.531 | Chronic embolism and thrombosis of right popliteal vein |
| 182.532 | Chronic embolism and thrombosis of left popliteal vein |
| 182.533 | bilateral |
| 182.539 | Chronic embolism and thrombosis of unspecified popliteal vein |
| 182.54 | Chronic embolism and thrombosis of tibial vein |
| 182.541 | Chronic embolism and thrombosis of right tibial vein |
| 182.542 | Chronic embolism and thrombosis of left tibial vein |
| 182.543 | bilateral |
| 182.549 | Chronic embolism and thrombosis of unspecified tibial vein |
| 182.55 | Chronic embolism and thrombosis of peroneal vein |
| 182.551 | Chronic embolism and thrombosis of right peroneal vein |
| 182.552 | Chronic embolism and thrombosis of left peroneal vein |
| 182.553 | bilateral |
| 182.559 | Chronic embolism and thrombosis of unspecified peroneal vein |
| 182.56 | Chronic embolism and thrombosis of calf muscular vein |
| 182.561 | Chronic embolism and thrombosis of right calf muscular vein |
| 182.562 | Chronic embolism and thrombosis of left calf muscular vein |
| 182.563 | bilateral |
| 182.569 | Chronic embolism and thrombosis of unspecified calf muscular vein |
| 182.59 | Chronic embolism and thrombosis of other specified deep vein of lower extremity |
| 182.591 | Chronic embolism and thrombosis of other specified deep vein of right lower extremity |
| 182.592 | Chronic embolism and thrombosis of other specified deep vein of left lower extremity |
| 182.593 | bilateral |

| 182.599 | Chronic embolism and thrombosis of other specified deep vein of unspecified lower extremity |
|---|---|
| 182.5Y | Chronic embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| 182.5Y1 | Chronic embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| 182.5Y2 | Chronic embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| 182.5Y3 | bilateral |
| 182.5Y9 | Chronic embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| 182.5Z | Chronic embolism and thrombosis of unspecified deep veins of distal lower extremity |
| I82.5Z1 | Chronic embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| 182.5Z2 | Chronic embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| 182.5Z3 | bilateral |
| 182.5Z9 | Chronic embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |


#### **Dialysis**

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

-ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

-ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

CPT/Lcodes

#### **Pregnancy** Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION
#### Appendix A

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

#### Appendix A

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS



| | | | | | Unmatched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optu | m | | Markets | Scan | | Medicare | | | Poforone | POOLED Dahigatran | |
| ariable | WARFARIN Copy | Dabigatran 150mg Copy | St. Diff. Refe | rence - warfarin Copy ! - | Dabigatran 150mg Copy | St. Diff. Refe | rence - warfarin Copy at | ran 150mg Copy | St. Diff. | Reference - warfarin<br>Copy | Exposure - Dabigatran<br>150mg Copy | St |
| umber of patients | 12,559 | 400 | | 18,874 | 727 | | 65,437 | 1.592 | | 96,870 | 2,719 | - |
| ge | , | | | , | | | , | -, | | , | -, | |
| mean (sd) | 65.83 (14.67) | 60.86 (15.91) | 0.32 | 57.54 (15.42) | 55.10 (15.33) | 0.16 | 76.75 (8.13) | 75.79 (7.70) | 0.12 | 71.59 (10.90) | 68.06 (11.61) | |
| ge categories without zero category | , | | | , | | | | | | , | | |
| 18 - 54; n (%) | 2,744 (21.8%) | 135 (33.8%) | -0.27 | 7,725 (40.9%) | 356 (49.0%) | -0.16 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 10,469 (10.8%) | 491 (18.1%) | |
| 55 - 64; n (%) | 2,310 (18.4%) | 77 (19.2%) | -0.02 | 6,043 (32.0%) | 206 (28.3%) | 0.08 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 8,353 (8.6%) | 283 (10.4%) | |
| .65 - 74; n (%) | 3,544 (28.2%) | 107 (26.8%) | 0.03 | 2,298 (12.2%) | 80 (11.0%) | 0.04 | 29,940 (45.8%) | 796 (50.0%) | -0.08 | 35,782 (36.9%) | 983 (36.2%) | |
| .>= 75; n (%) | 3,961 (31.5%) | 81 (20.2%) | 0.26 | 2,808 (14.9%) | 85 (11.7%) | 0.09 | 35,497 (54.2%) | 796 (50.0%) | 0.08 | 42,266 (43.6%) | 962 (35.4%) | |
| ender without zero category- United | .,, | | | , , | | | , , | , | | ,, | | |
| Males: n (%) | 5,947 (47.4%) | 194 (48.5%) | -0.02 | 9,614 (50.9%) | 383 (52.7%) | -0.04 | 25.561 (39.1%) | 640 (40.2%) | -0.02 | 41.122 (42.5%) | 1.217 (44.8%) | |
| Females: n (%) | 6,612 (52.6%) | 206 (51.5%) | 0.02 | 9,260 (49.1%) | 344 (47.3%) | 0.04 | 39,876 (60.9%) | 952 (59.8%) | 0.02 | 55,748 (57.5%) | 1,502 (55.2%) | |
| ace | .,. (, | , | | .,, | , | | ,. | | | | , , , | |
| White; n (%) | | | | | | | 58,175 (88.9%) | 1,414 (88.8%) | | 58,175 (88.9%) | 1,414 (88.8%) | |
| Black; n (%) | | | | | | | 4,876 (7.5%) | 106 (6.7%) | | 4,876 (7.5%) | 106 (6.7%) | |
| Asian; n (%) | | | | | | | 343 (0.5%) | 9 (0.6%) | | 343 (0.5%) | 9 (0.6%) | |
| Hispanic; n (%) | | | | | | | 786 (1.2%) | 22 (1.4%) | | 786 (1.2%) | 22 (1.4%) | |
| North American Native: n (%) | | | | | | | 218 (0.3%) | 3 (0.2%) | | 218 (0.3%) | 3 (0.2%) | |
| Other/Unknown; n (%) egion without zero category- United v3 (lumping | | | | | | | 1,039 (1.6%) | 38 (2.4%) | | 1,039 (1.6%) | 38 (2.4%) | |
| sing&other category with West) | | | | | | | | | | | | |
| Northeast; n (%) | 1,387 (11.0%) | 44 (11.0%) | 0.00 | 3,508 (18.6%) | 169 (23.2%) | -0.11 | 13,285 (20.3%) | 383 (24.1%) | -0.09 | 18,180 (18.8%) | 596 (21.9%) | |
| South; n (%) | 3,736 (29.7%) | 167 (41.8%) | -0.25 | 5,758 (30.5%) | 125 (17.2%) | 0.32 | 20,262 (31.0%) | 558 (35.1%) | -0.09 | 29,756 (30.7%) | 850 (31.3%) | |
| Midwest; n (%) | 3,599 (28.7%) | 88 (22.0%) | 0.15 | 5,483 (29.1%) | 230 (31.6%) | -0.05 | 18,819 (28.8%) | 317 (19.9%) | 0.21 | 27,901 (28.8%) | 635 (23.4%) | |
| Vest; n (%) | 3,837 (30.6%) | 101 (25.2%) | 0.12 | 3,922 (20.8%) | 200 (27.5%) | -0.16 | 12,972 (19.8%) | 330 (20.7%) | -0.02 | 20,731 (21.4%) | 631 (23.2%) | |
| Inknown+missing; n (%) | N/A | N/A | #VALUE! | 203 (1.1%) | 3 (0.4%) | 0.08 | N/A | N/A | #VALUE! | 203 (1.1%) | 3 (0.4%) | |
| Covariates | | | | | | | | | | | | |
| hemic heart disease; n (%) | 1,832 (14.6%) | 43 (10.8%) | 0.11 | 1,777 (9.4%) | 71 (9.8%) | -0.01 | 12,693 (19.4%) | 322 (20.2%) | -0.02 | 16,302 (16.8%) | 436 (16.0%) | |
| ute MI; n (%) | 77 (0.6%) | 1 (0.2%) | 0.06 | 77 (0.4%) | 4 (0.6%) | -0.03 | 495 (0.8%) | 12 (0.8%) | 0.00 | 649 (0.7%) | 17 (0.6%) | |
| S/unstable angina; n (%) | 71 (0.6%) | 4 (1.0%) | -0.04 | 66 (0.3%) | 4 (0.6%) | -0.04 | 473 (0.7%) | 11 (0.7%) | 0.00 | 610 (0.6%) | 19 (0.7%) | |
| d MI; n (%) | 332 (2.6%) | 8 (2.0%) | 0.04 | 237 (1.3%) | 15 (2.1%) | -0.06 | 2,550 (3.9%) | 65 (4.1%) | -0.01 | 3119 (3.2%) | 88 (3.2%) | |
| ble angina; n (%) | 170 (1.4%) | 3 (0.8%) | 0.06 | 131 (0.7%) | 10 (1.4%) | -0.07 | 871 (1.3%) | 34 (2.1%) | -0.06 | 1,172 (1.2%) | 047 (1.7%) | |
| ronary atherosclerosis and other forms of chronic | | | | | | | | | | | | |
| hemic heart disease; n (%) | 1,675 (13.3%) | 42 (10.5%) | 0.09 | 1,643 (8.7%) | 61 (8.4%) | 0.01 | 11,779 (18.0%) | 298 (18.7%) | -0.02 | 15,097 (15.6%) | 401 (14.7%) | |
| her atherosclerosis with ICD10 v2 Copy; n (%) | 101 (0.8%) | 2 (0.5%) | 0.04 | 124 (0.7%) | 6 (0.8%) | -0.01 | 843 (1.3%) | 14 (0.9%) | 0.04 | 1068 (1.1%) | 22 (0.8%) | |
| evious cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | | | | |
| ; n (%) | 34 (0.3%) | 2 (0.5%) | -0.03 | 36 (0.2%) | 2 (0.3%) | -0.02 | 181 (0.3%) | 8 (0.5%) | -0.03 | 251 (0.3%) | 12 (0.4%) | |
| story of CABG or PTCA; n (%) | 440 (3.5%) | 9 (2.2%) | 0.08 | 226 (1.2%) | 10 (1.4%) | -0.02 | 3,774 (5.8%) | 122 (7.7%) | -0.08 | 4,440 (4.6%) | 141 (5.2%) | |
| y stroke; n (%) | 451 (3.6%) | 14 (3.5%) | 0.01 | 526 (2.8%) | 13 (1.8%) | 0.07 | 3,441 (5.3%) | 76 (4.8%) | 0.02 | 4,418 (4.6%) | 103 (3.8%) | |
| hemic stroke (w and w/o mention of cerebral | | | | | | | | | | | | |
| arction); n (%) | 451 (3.6%) | 14 (3.5%) | 0.01 | 526 (2.8%) | 13 (1.8%) | 0.07 | 3,441 (5.3%) | 76 (4.8%) | 0.02 | 4,418 (4.6%) | 103 (3.8%) | |
| morrhagic stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 0 (0.0%) | |
| ; n (%) | 100 (0.8%) | 1 (0.2%) | 0.09 | 101 (0.5%) | 5 (0.7%) | -0.03 | 704 (1.1%) | 26 (1.6%) | -0.04 | 905 (0.9%) | 32 (1.2%) | |
| her cerebrovascular disease; n (%) | 200 (1.6%) | 7 (1.8%) | -0.02 | 216 (1.1%) | 10 (1.4%) | -0.03 | 1,482 (2.3%) | 31 (1.9%) | 0.03 | 1898 (2.0%) | 48 (1.8%) | |
| rebrovascular procedure; n (%) | 2 (0.0%) | 0 (0.0%) | #DIV/0! | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 34 (0.1%) | 2 (0.1%) | 0.00 | 039 (0.0%) | 2 (0.1%) | |
| art failure (CHF); n (%) | 1,245 (9.9%) | 28 (7.0%) | 0.10 | 993 (5.3%) | 40 (5.5%) | -0.01 | 7,488 (11.4%) | 191 (12.0%) | -0.02 | 9,726 (10.0%) | 259 (9.5%) | |
| ripheral Vascular Disease (PVD) or PVD Surgery v2; | | | | | | | | | | | | |
| %) | 1,037 (8.3%) | 35 (8.8%) | -0.02 | 944 (5.0%) | 33 (4.5%) | 0.02 | 6,344 (9.7%) | 155 (9.7%) | 0.00 | 8,325 (8.6%) | 223 (8.2%) | |
| rial fibrillation; n (%) | 1,476 (11.8%) | 51 (12.8%) | -0.03 | 1,184 (6.3%) | 65 (8.9%) | -0.10 | 9,318 (14.2%) | 238 (14.9%) | -0.02 | 11,978 (12.4%) | 354 (13.0%) | |
| her cardiac dysrhythmia; n (%) | 2,089 (16.6%) | 74 (18.5%) | -0.05 | 2,071 (11.0%) | 105 (14.4%) | -0.10 | 11,009 (16.8%) | 313 (19.7%) | -0.08 | 15,169 (15.7%) | 492 (18.1%) | |
| rdiac conduction disorders; n (%) | 613 (4.9%) | 21 (5.2%) | -0.01 | 552 (2.9%) | 16 (2.2%) | 0.04 | 3,328 (5.1%) | 94 (5.9%) | -0.04 | 4493 (4.6%) | 131 (4.8%) | |
| her CVD; n (%) | 2,404 (19.1%) | 75 (18.8%) | 0.01 | 2,244 (11.9%) | 94 (12.9%) | -0.03 | 10,471 (16.0%) | 306 (19.2%) | -0.08 | 15,119 (15.6%) | 475 (17.5%) | |
| betes-related complications | | | | | | | | | | | | |
| currence of Diabetic Neuropathy v2 Copy; n (%)<br>currence of diabetic nephropathy V3 with ICD10 | 488 (3.9%) | 15 (3.8%) | 0.01 | 413 (2.2%) | 11 (1.5%) | 0.05 | 2,446 (3.7%) | 59 (3.7%) | 0.00 | 3347 (3.5%) | 85 (3.1%) | |
| oy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 294 (0.4%) | 17 (1.1%) | -0.08 | 294 (0.3%) | 017 (0.6%) | |
| poglycemia v2; n (%) | 75 (0.6%) | 1 (0.2%) | 0.06 | 109 (0.6%) | 2 (0.3%) | 0.04 | 1,065 (1.6%) | 25 (1.6%) | 0.00 | 1249 (1.3%) | 28 (1.0%) | |
| perglycemia; n (%) | 727 (5.8%) | 17 (4.2%) | 0.07 | 641 (3.4%) | 24 (3.3%) | 0.01 | 4,147 (6.3%) | 140 (8.8%) | -0.09 | 5515 (5.7%) | 181 (6.7%) | |
| betic ketoacidosis; n (%) | 14 (0.1%) | 0 (0.0%) | 0.04 | 22 (0.1%) | 0 (0.0%) | 0.04 | 78 (0.1%) | 2 (0.1%) | 0.00 | 114 (0.1%) | 02 (0.1%) | |
| pertension: 1 inpatient or 2 outpatient claims | | | | | | | | | | | | |
| hin 365 days; n (%) | 7,347 (58.5%) | 217 (54.2%) | 0.09 | 8,418 (44.6%) | 264 (36.3%) | 0.17 | 49,234 (75.2%) | 1,197 (75.2%) | 0.00 | 64,999 (67.1%) | 1,678 (61.7%) | |
| erlipidemia v2; n (%) | 5,245 (41.8%) | 159 (39.8%) | 0.04 | 6,037 (32.0%) | 196 (27.0%) | 0.11 | 29,994 (45.8%) | 775 (48.7%) | -0.06 | 41,276 (42.6%) | 1,130 (41.6%) | |
| ma; n (%) | 2,533 (20.2%) | 92 (23.0%) | -0.07 | 3,140 (16.6%) | 129 (17.7%) | -0.03 | 12,415 (19.0%) | 358 (22.5%) | -0.09 | 18088 (18.7%) | 579 (21.3%) | |
| al Dysfunction (non-diabetic) v2; n (%) | 15 (0.1%) | 0 (0.0%) | 0.04 | 19 (0.1%) | 2 (0.3%) | -0.04 | 72 (0.1%) | 3 (0.2%) | -0.03 | 106 (0.1%) | 005 (0.2%) | |
| urrence of acute renal disease v2; n (%) | 7 (0.1%) | 0 (0.0%) | 0.04 | 12 (0.1%) | 1 (0.1%) | 0.00 | 58 (0.1%) | 2 (0.1%) | 0.00 | 77 (0.1%) | 3 (0.1%) | |
| currence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | |
| onic kidney disease v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | |
| Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | |
| currence of hypertensive nephropathy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | |
| currence of miscellaneous renal insufficiency v2; n | | • | | • | | | • | | | • | • | |
| | 8 (0.1%) | 0 (0.0%) | 0.04 | 7 (0.0%) | 1 (0.1%) | -0.04 | 13 (0.0%) | 1 (0.1%) | -0.04 | 28 (0.0%) | 002 (0.1%) | |
| ner Covariates | | . , | | . , | . , | | | | | | | |
| er disease; n (%) | 58 (0.5%) | 1 (0.2%) | 0.05 | 73 (0.4%) | 3 (0.4%) | 0.00 | 325 (0.5%) | 7 (0.4%) | 0.01 | 456 (0.5%) | 11 (0.4%) | |
| | | | | 3,577 (19.0%) | 126 (17.3%) | | | 507 (31.8%) | | | · | |

| Other arthritis. arthropathies and musculoskeletal | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pain; n (%) | 7,837 (62.4%) | 291 (72.8%) | -0.22 | 12,397 (65.7%) | 492 (67.7%) | -0.04 | 39,418 (60.2%) | 1,054 (66.2%) | -0.12 | 59652 (61.6%) | 1837 (67.6%) | -0.13 |
| Dorsopathies; n (%) | 3,526 (28.1%) | 123 (30.8%) | -0.06 | 4,793 (25.4%) | 180 (24.8%) | 0.01 | 17,513 (26.8%) | 455 (28.6%) | -0.04 | 25832 (26.7%) | 758 (27.9%) | -0.03 |
| Fractures; n (%) | 1,004 (8.0%) | 37 (9.2%) | -0.04 | 1,348 (7.1%) | 53 (7.3%) | -0.01 | 5,946 (9.1%) | 144 (9.0%) | 0.00 | 8298 (8.6%) | 234 (8.6%) | 0.00 |
| Falls v2; n (%) | 1,037 (8.3%) | 34 (8.5%) | -0.01 | 683 (3.6%) | 30 (4.1%) | -0.03 | 2,858 (4.4%) | 73 (4.6%) | -0.01 | 4578 (4.7%) | 137 (5.0%) | -0.01 |
| Osteoporosis; n (%) | 942 (7.5%) | 19 (4.8%) | 0.11 | 712 (3.8%) | 19 (2.6%) | 0.07 | 7,465 (11.4%) | 161 (10.1%) | 0.04 | 9119 (9.4%) | 199 (7.3%) | 0.08 |
| Depression; n (%) | 1,755 (14.0%) | 53 (13.2%) | 0.02 | 2,091 (11.1%) | 66 (9.1%) | 0.07 | 8,730 (13.3%) | 214 (13.4%) | 0.00 | 12576 (13.0%) | 333 (12.2%) | 0.02 |
| Anxiety; n (%) | 1,714 (13.6%) | 64 (16.0%) | -0.07 | 1,977 (10.5%) | 79 (10.9%) | -0.01 | 7,201 (11.0%) | 208 (13.1%) | -0.06 | 10892 (11.2%) | 351 (12.9%) | -0.05 |
| Sleep_Disorder; n (%) | 1,002 (8.0%) | 11 (2.8%) | 0.23 | 1,800 (9.5%) | 28 (3.9%) | 0.23 | 4,455 (6.8%) | 57 (3.6%) | 0.14 | 7257 (7.5%) | 96 (3.5%) | 0.18 |
| Dementia; n (%) | 988 (7.9%) | 22 (5.5%) | 0.10 | 717 (3.8%) | 31 (4.3%) | -0.03 | 9,297 (14.2%) | 196 (12.3%) | 0.06 | 11002 (11.4%) | 249 (9.2%) | 0.07 |
| Delirium; n (%) | 319 (2.5%) | 7 (1.8%) | 0.05 | 294 (1.6%) | 13 (1.8%) | -0.02 | 2,379 (3.6%) | 60 (3.8%) | -0.01 | 2992 (3.1%) | 80 (2.9%) | 0.01 |
| Psychosis; n (%) | 275 (2.2%) | 8 (2.0%) | 0.01<br>0.01 | 195 (1.0%) | 3 (0.4%) | 0.07<br>-0.02 | 1,851 (2.8%) | 33 (2.1%) | 0.05<br>-0.03 | 2321 (2.4%) | 44 (1.6%) | 0.06<br>-0.03 |
| Obesity; n (%) Overweight; n (%) | 2,754 (21.9%)<br>538 (4.3%) | 86 (21.5%)<br>23 (5.8%) | -0.07 | 3,425 (18.1%)<br>459 (2.4%) | 137 (18.8%)<br>24 (3.3%) | -0.02 | 9,371 (14.3%)<br>2.161 (3.3%) | 242 (15.2%)<br>59 (3.7%) | -0.03 | 15550 (16.1%)<br>3158 (3.3%) | 465 (17.1%)<br>106 (3.9%) | -0.03 |
| Smoking: n (%) | 2,612 (20.8%) | 94 (23.5%) | -0.07 | 2,264 (12.0%) | 24 (3.3%)<br>86 (11.8%) | 0.05 | 14,702 (22.5%) | 446 (28.0%) | -0.02 | 19578 (20.2%) | 626 (23.0%) | -0.03 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13 (0.0%) | 1 (0.1%) | -0.13 | 13 (0.0%) | 1 (0.0%) | #DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| COPD; n (%) | 1,828 (14.6%) | 49 (12.2%) | 0.07 | 1,476 (7.8%) | 44 (6.1%) | 0.07 | 10,257 (15.7%) | 281 (17.7%) | -0.05 | 13561 (14.0%) | 374 (13.8%) | 0.01 |
| Asthma; n (%) | 1,147 (9.1%) | 44 (11.0%) | -0.06 | 1,506 (8.0%) | 47 (6.5%) | 0.06 | 4,978 (7.6%) | 135 (8.5%) | -0.03 | 7631 (7.9%) | 226 (8.3%) | -0.01 |
| Obstructive sleep apnea; n (%) | 1,369 (10.9%) | 45 (11.2%) | -0.01 | 1,836 (9.7%) | 57 (7.8%) | 0.07 | 4,452 (6.8%) | 120 (7.5%) | -0.03 | 7657 (7.9%) | 222 (8.2%) | -0.01 |
| Pneumonia; n (%) | 1,066 (8.5%) | 37 (9.2%) | -0.02 | 1,329 (7.0%) | 58 (8.0%) | -0.04 | 5,876 (9.0%) | 142 (8.9%) | 0.00 | 8271 (8.5%) | 237 (8.7%) | -0.01 |
| Other Medications | | | | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 2,869 (22.8%) | 77 (19.2%) | 0.09 | 3,586 (19.0%) | 100 (13.8%) | 0.14 | 17,313 (26.5%) | 400 (25.1%) | 0.03 | 23768 (24.5%) | 577 (21.2%) | 0.08 |
| Use of ARBs; n (%) | 1,610 (12.8%) | 44 (11.0%) | 0.06 | 2,144 (11.4%) | 71 (9.8%) | 0.05 | 10,615 (16.2%) | 307 (19.3%) | -0.08 | 14369 (14.8%) | 422 (15.5%) | -0.02 |
| Use of Loop Diuretics - United; n (%) | 1,703 (13.6%) | 38 (9.5%) | 0.13 | 1,707 (9.0%) | 50 (6.9%) | 0.08 | 12,745 (19.5%) | 295 (18.5%) | 0.03 | 16155 (16.7%) | 383 (14.1%) | 0.07 |
| Use of other diuretics- United; n (%) | 276 (2.2%) | 9 (2.2%) | 0.00 | 366 (1.9%) | 9 (1.2%) | 0.06 | 1,909 (2.9%) | 55 (3.5%) | -0.03 | 2551 (2.6%) | 73 (2.7%) | -0.01 |
| Use of nitrates-United; n (%) | 342 (2.7%) | 3 (0.8%) | 0.15 | 365 (1.9%) | 10 (1.4%) | 0.04 | 3,101 (4.7%) | 80 (5.0%) | -0.01 | 3808 (3.9%) | 93 (3.4%) | 0.03 |
| Use of other hypertension drugs; n (%) | 520 (4.1%) | 16 (4.0%) | 0.01 | 444 (2.4%) | 13 (1.8%) | 0.04 | 3,247 (5.0%) | 80 (5.0%) | 0.00 | 4211 (4.3%) | 109 (4.0%) | 0.02 |
| Use of Anti-arrhythmics; n (%) | 176 (1.4%) | 6 (1.5%) | -0.01 | 211 (1.1%) | 16 (2.2%) | -0.09 | 1,375 (2.1%) | 42 (2.6%) | -0.03 | 1762 (1.8%) | 64 (2.4%) | -0.04 |
| Use of COPD/asthma meds- United; n (%) | 2,066 (16.5%) | 60 (15.0%) | 0.04 | 2,940 (15.6%) | 110 (15.1%) | 0.01 | 12,191 (18.6%) | 332 (20.9%) | -0.06 | 17197 (17.8%) | 502 (18.5%) | -0.02 |
| Use of statins; n (%) | 4,290 (34.2%) | 120 (30.0%) | 0.09 | 5,037 (26.7%) | 153 (21.0%) | 0.13 | 27,479 (42.0%) | 643 (40.4%) | 0.03 | 36806 (38.0%) | 916 (33.7%) | 0.09 |
| Use of other lipid-lowering drugs; n (%) | 552 (4.4%) | 21 (5.2%) | -0.04 | 857 (4.5%) | 19 (2.6%) | 0.10 | 3,697 (5.6%) | 88 (5.5%) | 0.00 | 5106 (5.3%) | 128 (4.7%) | 0.03 |
| Use of antiplatelet agents; n (%) | 574 (4.6%) | 21 (5.2%) | -0.03 | 859 (4.6%) | 42 (5.8%) | -0.05 | 4,480 (6.8%) | 139 (8.7%) | -0.07 | 5913 (6.1%) | 202 (7.4%) | -0.05 |
| Use of heparin and other low-molecular weight<br>heparins: n (%) | 4.744 (37.8%) | 93 (23.2%) | 0.32 | 22 (0.1%) | 0 (0.0%) | 0.04 | 24.694 (37.7%) | 299 (18.8%) | 0.43 | 29460 (30.4%) | 392 (14.4%) | 0.39 |
| Use of NSAIDs: n (%) | 1,843 (14.7%) | 81 (20.2%) | -0.15 | 3,344 (17.7%) | 161 (22.1%) | -0.11 | 8,958 (13.7%) | 279 (17.5%) | -0.10 | 14145 (14.6%) | 521 (19.2%) | -0.12 |
| Use of oral corticosteroids; n (%) | 2,853 (22.7%) | 97 (24.2%) | -0.04 | 4,300 (22.8%) | 179 (24.6%) | -0.04 | 16,673 (25.5%) | 458 (28.8%) | -0.10 | 23826 (24.6%) | 734 (27.0%) | -0.05 |
| Use of bisphosphonate (United); n (%) | 363 (2.9%) | 8 (2.0%) | 0.06 | 291 (1.5%) | 9 (1.2%) | 0.03 | 2,676 (4.1%) | 54 (3.4%) | 0.04 | 3330 (3.4%) | 71 (2.6%) | 0.05 |
| Use of opioids- United; n (%) | 4,758 (37.9%) | 159 (39.8%) | -0.04 | 8,083 (42.8%) | 301 (41.4%) | 0.03 | 23,923 (36.6%) | 635 (39.9%) | -0.07 | 36764 (38.0%) | 1095 (40.3%) | -0.05 |
| Use of antidepressants; n (%) | 3,087 (24.6%) | 94 (23.5%) | 0.03 | 4,318 (22.9%) | 149 (20.5%) | 0.06 | 19,013 (29.1%) | 466 (29.3%) | 0.00 | 26418 (27.3%) | 709 (26.1%) | 0.03 |
| Use of antipsychotics; n (%) | 487 (3.9%) | 16 (4.0%) | -0.01 | 500 (2.6%) | 15 (2.1%) | 0.03 | 3,676 (5.6%) | 77 (4.8%) | 0.04 | 4663 (4.8%) | 108 (4.0%) | 0.04 |
| Labs | , | ., ., | | , | | | -,,- | | | 31,433 | 1,127 | |
| Lab values- HbA1c (%) v3; n (%) | 1,354 (10.8%) | 41 (10.2%) | 0.02 | 142 (0.8%) | 3 (0.4%) | 0.05 | N/A | N/A | #VALUE! | 1,496 (4.8%) | 044 (3.9%) | 0.04 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 844 (6.7%) | 27 (6.8%) | 0.00 | 95 (0.5%) | 1 (0.1%) | 0.07 | N/A | N/A | #VALUE! | 939 (3.0%) | 028 (2.5%) | 0.03 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 1,354 (10.8%) | 41 (10.2%) | 0.02 | 142 (0.8%) | 3 (0.4%) | 0.05 | N/A | N/A | #VALUE! | 1,496 (4.8%) | 044 (3.9%) | 0.04 |
| Lab values- BNP; n (%) | 123 (1.0%) | 8 (2.0%) | -0.08 | 15 (0.1%) | 2 (0.3%) | -0.04 | N/A | N/A | #VALUE! | 138 (0.4%) | 010 (0.9%) | -0.06 |
| Lab values- BNP (within 3 months); n (%) | 100 (0.8%) | 4 (1.0%) | -0.02 | 11 (0.1%) | 1 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 111 (0.4%) | 005 (0.4%) | 0.00 |
| Lab values- BNP (within 6 months); n (%) | 123 (1.0%) | 8 (2.0%) | -0.08 | 15 (0.1%) | 2 (0.3%) | -0.04 | N/A | N/A | #VALUE! | 138 (0.4%) | 010 (0.9%) | -0.06 |
| Lab values- BUN (mg/dl); n (%) | 2,913 (23.2%) | 123 (30.8%) | -0.17 | 194 (1.0%) | 6 (0.8%) | 0.02 | N/A | N/A | #VALUE! | 3,107 (9.9%) | 129 (11.4%) | -0.05 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 2,019 (16.1%) | 87 (21.8%) | -0.15 | 142 (0.8%) | 4 (0.6%) | 0.02 | N/A | N/A | #VALUE! | 2,161 (6.9%) | 091 (8.1%) | -0.05 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 2,913 (23.2%) | 123 (30.8%) | -0.17 | 194 (1.0%) | 6 (0.8%) | 0.02 | N/A | N/A | #VALUE! | 3,107 (9.9%) | 129 (11.4%) | -0.05 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 2,983 (23.8%) | 128 (32.0%) | -0.18 | 199 (1.1%) | 6 (0.8%) | 0.03 | N/A | N/A | #VALUE! | 3,182 (10.1%) | 134 (11.9%) | -0.06 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2;<br>n (%) | 2,070 (16.5%) | 93 (23.2%) | -0.17 | 145 (0.8%) | 4 (0.6%) | 0.02 | N/A | N/A | #VALUE! | 2,215 (7.0%) | 097 (8.6%) | -0.06 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | 2,0.0 (10.3/0) | 33 (23.2/0) | 0.17 | 1-3 (0.070) | 4 (0.070) | 3.02 | IV/A | 19/0 | EOE: | 2,223 (7.070) | 557 (0.070) | -0.00 |
| n (%) | 2,983 (23.8%) | 128 (32.0%) | -0.18 | 199 (1.1%) | 6 (0.8%) | 0.03 | N/A | N/A | #VALUE! | 3,182 (10.1%) | 134 (11.9%) | -0.06 |
| Lab values- HDL level (mg/dl); n (%) | 1,798 (14.3%) | 75 (18.8%) | -0.12 | 110 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,908 (6.1%) | 078 (6.9%) | -0.03 |
| | , , | | | | | | | | | | | |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 1,041 (8.3%) | 46 (11.5%) | -0.11 | 67 (0.4%) | 1 (0.1%) | 0.06 | N/A | N/A | #VALUE! | 1,108 (3.5%) | 047 (4.2%) | -0.04 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 1,798 (14.3%) | 75 (18.8%) | -0.12 | 110 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,908 (6.1%) | 078 (6.9%) | -0.03 |
| Lab values- LDL level (mg/dl) v2; n (%) | 1,798 (14.3%) | 78 (19.5%) | -0.12 | 128 (0.7%) | 3 (0.4%) | 0.03 | N/A | N/A<br>N/A | #VALUE! | 2,035 (6.5%) | 081 (7.2%) | -0.03 |
| Lab values-LDL level (mg/dl) (within 3 months) v2; n | 1,507 (13.270) | 70 (15.370) | -0.11 | 120 (0.770) | 3 (0.4%) | 0.04 | N/A | N/A | #VALUE: | 2,033 (0.370) | 001 (7.270) | *0.03 |
| (%) | 1,101 (8.8%) | 50 (12.5%) | -0.12 | 77 (0.4%) | 1 (0.1%) | 0.06 | N/A | N/A | #VALUE! | 1,178 (3.7%) | 051 (4.5%) | -0.04 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n | 1,101 (0.070) | 30 (12.370) | 0.11 | ,, (0.470) | 1 (0.170) | 0.00 | 14/0 | | | 1,1,0 (3.7,0) | 032 (4.370) | 3.54 |
| (%) | 1,907 (15.2%) | 78 (19.5%) | -0.11 | 128 (0.7%) | 3 (0.4%) | 0.04 | N/A | N/A | #VALUE! | 2,035 (6.5%) | 081 (7.2%) | -0.03 |
| Lab values- NT-proBNP; n (%) | 27 (0.2%) | 0 (0.0%) | 0.06 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 28 (0.1%) | 0 (0.0%) | 0.04 |
| Lab values- NT-proBNP (within 3 months); n (%) | 22 (0.2%) | 0 (0.0%) | 0.06 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 22 (0.1%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 27 (0.2%) | 0 (0.0%) | 0.06 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 28 (0.1%) | 0 (0.0%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 1,844 (14.7%) | 78 (19.5%) | -0.13 | 107 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,951 (6.2%) | 081 (7.2%) | -0.04 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | | | | |
| months) v2; n (%) | 1,072 (8.5%) | 50 (12.5%) | -0.13 | 65 (0.3%) | 1 (0.1%) | 0.04 | N/A | N/A | #VALUE! | 1,137 (3.6%) | 051 (4.5%) | -0.05 |
| Lab values-Total cholesterol (mg/dl) (within 6 | 4 044 ***** | 70 / | | 40-7 | | | | | | 4.05 - / // | | |
| months) v2; n (%) | 1,844 (14.7%) | 78 (19.5%) | -0.13 | 107 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,951 (6.2%) | 081 (7.2%) | -0.04 |
| Lab values-Triglyceride level (mg/dl); n (%) | 1,803 (14.4%) | 78 (19.5%) | -0.14 | 106 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,909 (6.1%) | 081 (7.2%) | -0.04 |
| Lab values-Triglyceride level (mg/dl) (within 3 | 1,048 (8.3%) | 50 (12.5%) | -0.14 | 63 (0.3%) | 1 (0.1%) | 0.04 | N/A | N/A | #VALUE! | 1,111 (3.5%) | 051 (4.5%) | -0.05 |
| months); n (%) | 1,048 (8.3%) | JU (12.3%) | -0.14 | U3 (U.3%) | 1 (U.176) | 0.04 | IN/A | N/A | #VALUE! | 1,111 (3.3%) | 031 (4.3%) | -0.05 |

| lah valuas Taialussaida laval (asa (dl) (viibbia C | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lab values-Triglyceride level (mg/dl) (within 6 months): n (%) | 1,803 (14.4%) | 78 (19.5%) | -0.14 | 106 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 1,909 (6.1%) | 081 (7.2%) | -0.04 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | _,===(=, | (====, | | | - ( | | | .4 | | _,=== (====, | ( | |
| included) v4 | 1,343 | 41 | | 140 | 3 | | N/A | N/A | | 1,483 | 44 | |
| mean (sd) | 6.41 (1.25) | 6.18 (0.73) | 0.22 | 7.02 (1.62) | 5.93 (0.40) | 0.92 | N/A | N/A | #VALUE! | 6.47 (1.29) | 6.16 (0.73) | 0.30 |
| Missing; n (%) | 11,216 (89.3%) | 359 (89.8%) | -0.02 | 18,734 (99.3%) | 724 (99.6%) | -0.04 | N/A | N/A | #VALUE! | 29,950 (95.3%) | 1,083 (96.1%) | -0.04 |
| Lab result number- BNP mean v2 | 123 | 8 | 0.20 | 15 | 2 | 0.54 | N/A | N/A | #VALUE! | 138 | 10 | 0.20 |
| mean (sd) | 192.47 (369.22)<br>12,436 (99.0%) | 134.34 (166.13)<br>392 (98.0%) | 0.20 | 169.87 (442.05)<br>18,859 (99.9%) | 0.00 (0.00)<br>725 (99.7%) | 0.54 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 190.01 (378.76)<br>31,295 (99.6%) | 107.47 (166.13)<br>1,117 (99.1%) | 0.28 |
| Missing; n (%)<br>Lab result number- BUN (mg/dl) mean v2 | 2,436 (99.0%) | 392 (98.0%)<br>123 | 0.08 | 18,859 (99.9%) | 725 (99.7%) | 0.04 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 31,295 (99.6%) | 1,117 (99.1%) | 0.06 |
| mean (sd) | 16.64 (5.97) | 15.98 (5.29) | 0.12 | 17.10 (7.20) | 13.88 (2.72) | 0.59 | N/A | N/A | #VALUE! | 16.67 (6.05) | 15.88 (5.23) | 0.14 |
| Missing; n (%) | 9,646 (76.8%) | 277 (69.2%) | 0.17 | 18,680 (99.0%) | 721 (99.2%) | -0.02 | N/A | N/A | #VALUE! | 28,326 (90.1%) | 998 (88.6%) | 0.05 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | .,, | | | .,, | , | | | | | .,, | , | |
| to 15 included) v3 | 2,949 | 128 | | 198 | 6 | | N/A | N/A | | 3,147 | 134 | |
| mean (sd) | 0.92 (0.23) | 0.92 (0.18) | 0.00 | 0.93 (0.25) | 0.87 (0.14) | 0.30 | N/A | N/A | #VALUE! | 0.92 (0.23) | 0.92 (0.18) | 0.00 |
| Missing; n (%) | 9,610 (76.5%) | 272 (68.0%) | 0.19 | 18,676 (99.0%) | 721 (99.2%) | -0.02 | N/A | N/A | #VALUE! | 28,286 (90.0%) | 993 (88.1%) | 0.06 |
| Lab result number- HDL level (mg/dl) mean (only<br>=<5000 included) v2 | 1,798 | 75 | | 110 | 3 | | N/A | N/A | | 1,908 | 78 | |
| mean (sd) | 53.28 (17.20) | 54.91 (14.00) | -0.10 | 47.03 (15.15) | 53.67 (10.26) | -0.51 | N/A | N/A | #VALUE! | 52.92 (17.09) | 54.86 (14.01) | -0.12 |
| Missing; n (%) | 10,761 (85.7%) | 325 (81.2%) | 0.12 | 18,764 (99.4%) | 724 (99.6%) | -0.03 | N/A | N/A | #VALUE! | 29,525 (93.9%) | 1,049 (93.1%) | 0.03 |
| Lab result number-LDL level (mg/dl) mean (only | , () | (, | | , () | ( , | | .4 | .4 | | , (, | _,(, | |
| =<5000 included) v2 | 1,851 | 76 | | 103 | 3 | | N/A | N/A | | 1,954 | 79 | |
| mean (sd) | 100.71 (36.46) | 103.41 (36.79) | -0.07 | 98.61 (40.99) | 104.33 (41.40) | -0.14 | N/A | N/A | #VALUE! | 100.60 (36.72) | 103.44 (37.16) | -0.08 |
| Missing; n (%) | 10,708 (85.3%) | 324 (81.0%) | 0.12 | 18,771 (99.5%) | 724 (99.6%) | -0.01 | N/A | N/A | #VALUE! | 29,479 (93.8%) | 1,048 (93.0%) | 0.03 |
| Lab result number-Total cholesterol (mg/dl) mean | 4.044 | 70 | | 107 | | | *** | | | 4.040 | | |
| (only =<5000 included) v2<br>mean (sd) | 1,841<br>182.43 (42.98) | 78<br>187.48 (39.96) | -0.12 | 107<br>180.30 (59.20) | 187.67 (27.61) | -0.16 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 1,948<br>182.31 (44.03) | 187.49 (39.95) | -0.12 |
| mean (sq)Missing; n (%) | 10.718 (85.3%) | 322 (80.5%) | 0.12 | 18.767 (99.4%) | 724 (99.6%) | -0.16 | N/A<br>N/A | N/A | #VALUE! | 29.485 (93.8%) | 1,046 (92.8%) | 0.12 |
| Lab result number-Triglyceride level (mg/dl) mean | 10,710 (03.370) | 322 (80.3%) | 0.13 | 18,707 (33.476) | 724 (33.0%) | -0.03 | N/A | N/A | #VALUE: | 25,463 (55.676) | 1,040 (52.6%) | 0.04 |
| (only =<5000 included) v2 | 1,803 | 78 | | 106 | 3 | | N/A | N/A | | 1,909 | 81 | |
| mean (sd) | 137.59 (83.23) | 145.68 (93.13) | -0.09 | 154.79 (111.79) | 147.00 (50.86) | 0.09 | N/A | N/A | #VALUE! | 138.55 (85.07) | 145.73 (92.89) | -0.08 |
| Missing; n (%) | 10,756 (85.6%) | 322 (80.5%) | 0.14 | 18,768 (99.4%) | 724 (99.6%) | -0.03 | N/A | N/A | #VALUE! | 29,524 (93.9%) | 1,046 (92.8%) | 0.04 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | | | | |
| included) | 2,383 | 106 | | 163 | 6 | | N/A | N/A | | 2,546 | 112 | |
| mean (sd) | 13.65 (1.74) | 13.90 (1.70) | -0.15<br>0.18 | 13.38 (1.68) | 13.42 (1.17) | -0.03<br>-0.01 | N/A | N/A | #VALUE!<br>#VALUE! | 13.63 (1.74) | 13.87 (1.69) | -0.14<br>0.06 |
| Missing; n (%)<br>Lab result number-Serum sodium mean (only > 90 | 10,176 (81.0%) | 294 (73.5%) | 0.18 | 18,711 (99.1%) | 721 (99.2%) | -0.01 | N/A | N/A | #VALUE! | 28,887 (91.9%) | 1,015 (90.1%) | 0.06 |
| and < 190 included) | 2.809 | 122 | | 190 | 6 | | N/A | N/A | | 2,999 | 128 | |
| mean (sd) | 140.39 (2.82) | 140.62 (2.21) | -0.09 | 139.45 (2.80) | 139.19 (2.10) | 0.11 | N/A | N/A | #VALUE! | 140.33 (2.82) | 140.55 (2.21) | -0.09 |
| Missing; n (%) | 9,750 (77.6%) | 278 (69.5%) | 0.18 | 18,684 (99.0%) | 721 (99.2%) | -0.02 | N/A | N/A | #VALUE! | 28,434 (90.5%) | 999 (88.6%) | 0.06 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | | | | |
| included) | 2,555 | 122 | | 149 | 3 | | N/A | N/A | | 2,704 | 125 | |
| mean (sd) | 4.10 (0.38) | 4.21 (0.37) | -0.29 | 3.98 (0.55) | 3.90 (0.35) | 0.17 | N/A | N/A | #VALUE! | 4.09 (0.39) | 4.20 (0.37) | -0.29 |
| Missing; n (%) | 10,004 (79.7%) | 278 (69.5%) | 0.24 | 18,725 (99.2%) | 724 (99.6%) | -0.05 | N/A | N/A | #VALUE! | 28,729 (91.4%) | 1,002 (88.9%) | 0.08 |
| Lab result number-Glucose (fasting or random) mean<br>(only 10-1000 included) | 2.793 | 122 | | 194 | 7 | | N/A | N/A | | 2,987 | 129 | |
| mean (sd) | 108.41 (36.03) | 102.95 (22.39) | 0.18 | 129.30 (53.76) | 116.12 (16.32) | 0.33 | N/A | N/A | #VALUE! | 109.77 (37.44) | 103.66 (22.23) | 0.20 |
| Missing; n (%) | 9,766 (77.8%) | 278 (69.5%) | 0.19 | 18,680 (99.0%) | 720 (99.0%) | 0.00 | N/A | N/A | #VALUE! | 28,446 (90.5%) | 998 (88.6%) | 0.06 |
| Lab result number-Potassium mean (only 1-7 | | | | | | | | | | | | |
| included) | 2,957 | 129 | | 189 | 6 | | N/A | N/A | | 3,146 | 135 | |
| mean (sd) | 4.33 (0.41) | 4.35 (0.43) | -0.05 | 4.29 (0.41) | 4.30 (0.28) | -0.03 | N/A | N/A | #VALUE! | 4.33 (0.41) | 4.35 (0.43) | -0.05 |
| Missing; n (%) | 9,602 (76.5%) | 271 (67.8%) | 0.20 | 18,685 (99.0%) | 721 (99.2%) | -0.02 | N/A | N/A | #VALUE! | 28,287 (90.0%) | 992 (88.0%) | 0.06 |
| Comorbidity Scores Combined comorbidity score, 365 days Copy | | | | | | | | | | | | |
| mean (sd) | 1.79 (2.15) | 1.83 (2.15) | -0.02 | 1.14 (1.88) | 1.40 (1.87) | -0.14 | 255.04 (382.17) | 243.82 (378.73) | 0.03 | 172.74 (314.11) | 143.40 (289.87) | 0.10 |
| Non-Frailty; n (%) | 6,140 (48.9%) | 194 (48.5%) | 0.01 | 8,179 (43.3%) | 292 (40.2%) | 0.06 | 1,696 (2.6%) | 33 (2.1%) | 0.03 | 16,015 (16.5%) | 519 (19.1%) | -0.07 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | | | | | | |
| mean (sd) | 0.18 (0.07) | 0.17 (0.07) | 0.14 | 0.16 (0.06) | 0.15 (0.05) | 0.18 | 0.09 (0.07) | 0.08 (0.07) | 0.14 | 0.12 (0.07) | 0.11 (0.07) | 0.14 |
| Healthcare Utilization | | | | | | | | | | | _ | |
| Any hospitalization; n (%) | 5,166 (41.1%) | 201 (50.2%) | -0.18 | 7,772 (41.2%) | 313 (43.1%) | -0.04 | 28,960 (44.3%) | 828 (52.0%) | -0.15 | 41,898 (43.3%) | 1,342 (49.4%) | -0.12 |
| Any hospitalization within prior 30 days; n (%) | 4,405 (35.1%) | 170 (42.5%) | -0.15 | 6,695 (35.5%) | 267 (36.7%) | -0.02 | 22,606 (34.5%) | 637 (40.0%) | -0.11 | 33706 (34.8%) | 1074 (39.5%) | -0.10 |
| Any hospitalization during prior 31-180 days; n (%) Internal medicine/family medicine visits; n (%) | 1,178 (9.4%)<br>10,558 (84.1%) | 41 (10.2%)<br>334 (83.5%) | -0.03<br>0.02 | 1,506 (8.0%)<br>15,210 (80.6%) | 66 (9.1%)<br>528 (72.6%) | -0.04<br>0.19 | 9,511 (14.5%)<br>57,081 (87.2%) | 272 (17.1%)<br>1,424 (89.4%) | -0.07<br>-0.07 | 12195 (12.6%)<br>82849 (85.5%) | 379 (13.9%)<br>2286 (84.1%) | -0.04<br>0.04 |
| Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits (30 days | 10,558 (84.1%) | 334 (83.3%) | 0.02 | 15,210 (80.0%) | 528 (72.0%) | 0.19 | 57,081 (87.2%) | 1,424 (89.4%) | -0.07 | 82849 (83.3%) | 2280 (84.1%) | 0.04 |
| prior) v2; n (%) | 8,811 (70.2%) | 287 (71.8%) | -0.04 | 11,692 (61.9%) | 417 (57.4%) | 0.09 | 45,741 (69.9%) | 1,222 (76.8%) | -0.16 | 66244 (68.4%) | 1926 (70.8%) | -0.05 |
| Internal medicine/family medicine visits (31 to 180 | | | | , | | | , | , , , , , , , | | , , | , | |
| days prior) v2; n (%) | 8,508 (67.7%) | 246 (61.5%) | 0.13 | 12,135 (64.3%) | 405 (55.7%) | 0.18 | 47,557 (72.7%) | 1,155 (72.6%) | 0.00 | 68200 (70.4%) | 1806 (66.4%) | 0.09 |
| Cardiologist visit; n (%) | 5,451 (43.4%) | 198 (49.5%) | -0.12 | 4,402 (23.3%) | 170 (23.4%) | 0.00 | 29,552 (45.2%) | 852 (53.5%) | -0.17 | 39405 (40.7%) | 1220 (44.9%) | -0.08 |
| Number of Cardiologist visits (30 days prior); n (%) | 3,913 (31.2%) | 160 (40.0%) | -0.18 | 2,711 (14.4%) | 118 (16.2%) | -0.05 | 18,575 (28.4%) | 621 (39.0%) | -0.23 | 25199 (26.0%) | 899 (33.1%) | -0.16 |
| Number of Cardiologist visits (31 to 180 days prior); | 2.740 (24.50) | 00 (20 00) | | 2.470.42.40() | 00 (4.2. 20%) | 0.00 | 10 201 (27 51) | 470 (20 40) | 2.25 | 22404 (24.20) | C40 (22 00) | |
| n (%) | 2,718 (21.6%)<br>6.421 (51.1%) | 80 (20.0%)<br>226 (56.5%) | 0.04<br>-0.11 | 2,479 (13.1%)<br>6.680 (35.4%) | 89 (12.2%)<br>284 (39.1%) | 0.03<br>-0.08 | 18,204 (27.8%)<br>34.182 (52.2%) | 479 (30.1%)<br>1.001 (62.9%) | -0.05<br>-0.22 | 23401 (24.2%)<br>47283 (48.8%) | 648 (23.8%)<br>1511 (55.6%) | 0.01<br>-0.14 |
| Electrocardiogram v2; n (%) Use of glucose test strips; n (%) | 107 (0.9%) | 5 (1.2%) | -0.11<br>-0.03 | 126 (0.7%) | 284 (39.1%) 2 (0.3%) | 0.08 | 34,182 (52.2%)<br>719 (1.1%) | 20 (1.3%) | -0.22<br>-0.02 | 47283 (48.8%)<br>952 (1.0%) | 27 (1.0%) | 0.00 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! |
| number of different/distinct medication | | | | | / | , | · //-/ | | *** | | / | • • • • |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 7.97 (4.88) | 7.75 (5.15) | 0.04 | 7.81 (4.94) | 7.34 (4.82) | 0.10 | 8.96 (4.95) | 9.31 (4.99) | -0.07 | 8.61 (4.94) | 8.55 (4.97) | 0.00 |
| Number of Hospitalizations | 0 () | 0 / | | 0 (= :) | 0 // | | | 0.6=1=== | | 0 | | |
| mean (sd) | 0.49 (0.68) | 0.59 (0.67) | -0.15 | 0.47 (0.63) | 0.50 (0.64) | -0.05 | 0.57 (0.76) | 0.67 (0.82) | -0.13 | 0.54 (0.73) | 0.61 (0.75) | 0.00 |

| Number of hospital days | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 2.38 (4.28) | 2.28 (3.48) | 0.03 | 2.28 (4.36) | 1.95 (4.02) | 0.08 | 2.73 (4.90) | 2.74 (4.25) | 0.00 | 2.60 (4.72) | 2.46 (4.08) | 0.00 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | | | | |
| mean (sd) | 1.21 (1.75) | 1.50 (2.07) | -0.15 | 1.08 (3.19) | 1.14 (2.87) | -0.02 | 1.31 (1.90) | 1.61 (2.03) | -0.15 | 1.25 (2.20) | 1.47 (2.29) | 0.00 |
| Number of Office visits | 5 44 (4 50) | 5 47 (4 50) | 0.07 | 5.05 (4.52) | 4.74 (4.20) | 0.07 | 44.04.(43.03) | 42.22 (45.07) | -0.09 | 0.70 (44.55) | 0.07(43.40) | 0.00 |
| mean (sd) Number of internal medicine/family medicine visits | 5.14 (4.58) | 5.47 (4.68) | -0.07 | 5.05 (4.52) | 4.74 (4.30) | 0.07 | 11.91 (13.83) | 13.32 (15.87) | -0.09 | 9.70 (11.66) | 9.87 (12.48) | 0.00 |
| mean (sd) | 10.15 (13.39) | 8.50 (12.76) | 0.13 | 6.81 (11.07) | 5.46 (9.47) | 0.13 | 9.72 (11.37) | 9.24 (10.36) | 0.04 | 9.21 (11.60) | 8.12 (10.52) | 0.00 |
| Number of Cardiologist visits | 10:15 (15:55) | 0.30 (12.70) | 0.13 | 0.01(11.07) | 3.40 (3.47) | 0.13 | 3.72 (11.57) | 3.24 (20.30) | 0.04 | 3.22 (22.00) | 0.12 (10.52) | 0.00 |
| mean (sd) | 1.69 (3.88) | 1.82 (3.21) | -0.04 | 0.74 (2.40) | 0.81 (2.34) | -0.03 | 1.95 (4.28) | 2.51 (4.62) | -0.13 | 1.68 (3.93) | 1.95 (3.93) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | | | | |
| mean (sd) | 1.14 (1.80) | 1.36 (1.80) | -0.12 | 0.67 (1.22) | 0.76 (1.18) | -0.07 | 1.17 (1.67) | 1.51 (1.86) | -0.19 | 1.07 (1.61) | 1.29 (1.70) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.29 (0.60) | 0.29 (0.62) | 0.00 | 0.19 (0.49) | 0.18 (0.46) | 0.02 | 0.34 (0.66) | 0.38 (0.69) | -0.06 | 0.30 (0.62) | 0.31 (0.63) | 0.00 |
| Number of glucose tests ordered | 0.40 (2.50) | 0.40(4.04) | 0.00 | 0.40 (0.55) | 0.40 (0.45) | -0.04 | 0.43 (0.55) | 0.45 (0.54) | 2.25 | 0.42 (4.20) | 0.45 (0.55) | 0.00 |
| mean (sd)<br>Number of lipid tests ordered | 0.19 (3.50) | 0.18 (1.01) | 0.00 | 0.10 (0.55) | 0.12 (0.46) | -0.04 | 0.13 (0.65) | 0.16 (0.61) | -0.05 | 0.13 (1.39) | 0.15 (0.65) | 0.00 |
| mean (sd) | 0.45 (0.70) | 0.48 (0.69) | -0.04 | 0.33 (0.68) | 0.30 (0.61) | 0.05 | 0.49 (0.67) | 0.54 (0.72) | -0.07 | 0.45 (0.68) | 0.47 (0.69) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | , | | , | , | | , | , ,, | |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 7.58 (9.90) | 10.04 (11.37) | -0.23 | 4.03 (7.13) | 5.51 (8.06) | -0.19 | 9.32 (11.36) | 12.72 (12.88) | -0.28 | 8.06 (10.48) | 10.40 (11.56) | 0.00 |
| For PS | | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | 202 (4.50() | 7 (4 00/) | 0.00 | 247 (4 40() | 40 (4 40() | | 4 500 (2 20() | 22 (2 40() | 2.24 | 4020 (2.00() | 50 (4.00() | |
| disease+Cerebrovascular procedure (for PS); n (%) immobilization; n (%) | 202 (1.6%)<br>863 (6.9%) | 7 (1.8%)<br>29 (7.2%) | -0.02<br>-0.01 | 217 (1.1%)<br>1,257 (6.7%) | 10 (1.4%)<br>52 (7.2%) | -0.03<br>-0.02 | 1,509 (2.3%)<br>4,469 (6.8%) | 33 (2.1%)<br>110 (6.9%) | 0.01<br>0.00 | 1928 (2.0%)<br>1,257 (6.7%) | 50 (1.8%)<br>52 (7.2%) | 0.01<br>-0.02 |
| immobilization; n (%) | 803 (0.9%) | 29 (7.2%) | -0.01 | 1,257 (0.7%) | 52 (7.2%) | -0.02 | 4,409 (0.8%) | 110 (6.9%) | 0.00 | 1,257 (0.7%) | 52 (7.2%) | -0.02 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 798 (6.4%) | 33 (8.2%) | -0.07 | 1,158 (6.1%) | 94 (12.9%) | -0.23 | 5.855 (8.9%) | 169 (10.6%) | -0.06 | 7811 (8.1%) | 296 (10.9%) | -0.10 |
| Occurrence of BUN tests ordered (for PS); n (%) | 345 (2.7%) | 14 (3.5%) | -0.05 | 543 (2.9%) | 40 (5.5%) | -0.13 | 2,956 (4.5%) | 87 (5.5%) | -0.05 | 3844 (4.0%) | 141 (5.2%) | -0.06 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | | | | | | | | | |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Acute kidney injury; n (%) Bladder stones+Kidney stones (for PS); n (%) | 14 (0.1%)<br>224 (1.8%) | 0 (0.0%)<br>12 (3.0%) | 0.04<br>-0.08 | 13 (0.1%)<br>292 (1.5%) | 1 (0.1%)<br>11 (1.5%) | 0.00 | 94 (0.1%)<br>1,199 (1.8%) | 3 (0.2%)<br>37 (2.3%) | -0.03<br>-0.04 | 13 (0.1%)<br>1715 (1.8%) | 1 (0.1%)<br>60 (2.2%) | 0.00<br>-0.03 |
| Alcohol abuse or dependence+Drug abuse or | 224 (1.8%) | 12 (3.0%) | -0.08 | 292 (1.5%) | 11 (1.5%) | 0.00 | 1,199 (1.8%) | 37 (2.3%) | -0.04 | 1/15 (1.8%) | 00 (2.2%) | -0.03 |
| dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13 (0.0%) | 1 (0.1%) | -0.04 | 13 (0.0%) | 1 (0.0%) | #DIV/0! |
| Other atherosclerosis+Cardiac conduction | | | | | | | | | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 2,812 (22.4%) | 93 (23.2%) | -0.02 | 2,706 (14.3%) | 109 (15.0%) | -0.02 | 13,267 (20.3%) | 377 (23.7%) | -0.08 | 18785 (19.4%) | 579 (21.3%) | -0.05 |
| Previous cardiac procedure (CABG or PTCA or Stent) + | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 452 (3.6%) | 10 (2.5%) | 0.06 | 235 (1.2%) | 11 (1.5%) | -0.03 | 3,807 (5.8%) | 123 (7.7%) | -0.08 | 4494 (4.6%) | 144 (5.3%) | -0.03 |
| Diabetes with complication; n (%) | 761 (6.1%)<br>536 (4.3%) | 19 (4.8%)<br>14 (3.5%) | 0.06<br>0.04 | 715 (3.8%)<br>448 (2.4%) | 15 (2.1%)<br>16 (2.2%) | 0.10<br>0.01 | 4,915 (7.5%)<br>3,785 (5.8%) | 123 (7.7%)<br>82 (5.2%) | -0.01<br>0.03 | 715 (3.8%)<br>4769 (4.9%) | 15 (2.1%)<br>112 (4.1%) | 0.10 |
| Delirium + Psychosis (for PS); n (%)<br>Any use of Meglitinides (for PS); n (%) | 9 (0.1%) | 0 (0.0%) | 0.04 | 16 (0.1%) | 0 (0.0%) | 0.01 | 130 (0.2%) | 2 (0.1%) | 0.03 | 155 (0.2%) | 2 (0.1%) | 0.04 |
| Any use of AGIs (for PS); n (%) | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 5 (0.0%) | 0 (0.0%) | #DIV/0! | 30 (0.0%) | 0 (0.0%) | #DIV/0! | 39 (0.0%) | 0 (0.0%) | #DIV/0! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of thiazide- United; n (%) | 1,075 (8.6%) | 38 (9.5%) | -0.03 | 1,344 (7.1%) | 35 (4.8%) | 0.10 | 6,824 (10.4%) | 166 (10.4%) | 0.00 | 9243 (9.5%) | 239 (8.8%) | 0.02 |
| Use of beta blockers; n (%) | 3,364 (26.8%) | 89 (22.2%) | 0.11 | 3,825 (20.3%) | 135 (18.6%) | 0.04 | 23,544 (36.0%) | 582 (36.6%) | -0.01 | 30733 (31.7%) | 806 (29.6%) | 0.05 |
| Use of calcium channel blockers; n (%) | 2,231 (17.8%) | 68 (17.0%) | 0.02 | 2,626 (13.9%) | 91 (12.5%) | 0.04 | 15,179 (23.2%) | 365 (22.9%) | 0.01 | 20036 (20.7%) | 524 (19.3%) | 0.04 |
| All antidiabetic medications except Insulin; n (%) | 1,512 (12.0%) | 27 (6.8%) | 0.18 | 1,900 (10.1%) | 59 (8.1%) | 0.07 | 9,285 (14.2%) | 229 (14.4%) | -0.01 | 12697 (13.1%) | 315 (11.6%) | 0.05 |
| DM Medications - Insulin Copy; n (%) | 425 (3.4%)<br>2,730 (21.7%) | 9 (2.2%)<br>70 (17.5%) | 0.07 | 581 (3.1%)<br>3,029 (16.0%) | 12 (1.7%)<br>82 (11.3%) | 0.09 | 2,442 (3.7%)<br>18.159 (27.8%) | 52 (3.3%)<br>393 (24.7%) | 0.02 | 3448 (3.6%)<br>23918 (24.7%) | 73 (2.7%)<br>545 (20.0%) | 0.05<br>0.11 |
| Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) | 1,618 (12.9%) | 70 (17.5%)<br>50 (12.5%) | 0.11 | 2,005 (10.6%) | 72 (9.9%) | 0.14 | 9,675 (14.8%) | 262 (16.5%) | -0.05 | 13298 (13.7%) | 384 (14.1%) | -0.01 |
| Malignant hypertension; n (%) | 468 (3.7%) | 4 (1.0%) | 0.18 | 5,024 (26.6%) | 64 (8.8%) | 0.48 | 13,050 (19.9%) | 171 (10.7%) | 0.26 | 18542 (19.1%) | 239 (8.8%) | 0.30 |
| Cardiovascular stress test; n (%) | 81 (0.6%) | 2 (0.5%) | 0.01 | 100 (0.5%) | 3 (0.4%) | 0.01 | 570 (0.9%) | 15 (0.9%) | 0.00 | 751 (0.8%) | 20 (0.7%) | 0.01 |
| Echocardiogram; n (%) | 3,355 (26.7%) | 131 (32.8%) | -0.13 | 4,243 (22.5%) | 171 (23.5%) | -0.02 | 16,457 (25.1%) | 542 (34.0%) | -0.20 | 24055 (24.8%) | 844 (31.0%) | -0.14 |
| Number of BNP tests | | | | | | | | | | | | |
| mean (sd) | 0.10 (0.38) | 0.11 (0.37) | -0.03 | 0.06 (0.34) | 0.09 (0.31) | -0.09 | 0.12 (0.43) | 0.15 (0.50) | -0.06 | 0.11 (0.41) | 0.13 (0.44) | -0.05 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, N<br>mean (sd) | lyoglobin, CPK)<br>0.32 (1.08) | 0.44 (1.63) | -0.09 | 0.25 (0.89) | 0.24 (0.74) | 0.01 | 0.22 (0.55) | 0.26 (0.59) | -0.07 | 0.24 (0.71) | 0.28 (0.86) | 0.00 |
| mean (su) | 0.32 (1.08) | 0.44 (1.03) | -0.09 | 0.25 (0.89) | 0.24 (0.74) | 0.01 | 0.22 (0.55) | 0.26 (0.59) | -0.07 | 0.24 (0.71) | 0.28 (0.86) | 0.00 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.05) | 0.00 (0.05) | 0.00 | 0.00 (0.04) | 0.00 (0.05) | 0.00 | 0.00 (0.03) | 0.00 (0.00) | 0.00 | 0.00 (0.04) | 0.00 (0.03) | 0.00 |
| N of days on antihypertensive medications during baseli | | | | | | | 0 | 0 | | | | |
| mean (sd) | 79.82 (80.23) | 71.81 (80.61) | 0.10 | 64.28 (78.46) | 52.59 (73.78) | 0.15 | 102.06 (78.84) | 104.42 (78.60) | -0.03 | 91.82 (78.95) | 85.76 (77.64) | 0.00 |
| N of days in database anytime prior | 4 700 74 (4 255 20) | 4 070 54 (4 402 74) | 0.05 | 2 4 4 2 4 5 (4 4 4 5 6 7) | 2 077 55 (4 420 00) | | 0 | 0 | 0.00 | 4455 24 (222 42) | 4277 24 (4044 05) | 0.00 |
| mean (sd) | 1,790.71 (1,365.39) | 1,879.61 (1,483.74) | -0.06 | 2,142.15 (1,446.67) | 2,077.56 (1,420.98) | 0.05 | 748.63 (585.17) | /00.54 (524.10) | -0.02 | 1155.24 (938.49) | 1277.31 (1011.96) | 0.00 |
| Mean Copay for per prescription cost (charges in U.S. \$) | 180-1 day prior) | | | | | | 0 | 0 | | | | |
| mean (sd) | 25.10 (43.30) | 29.60 (62.15) | -0.08 | 12.89 (19.50) | 14.46 (21.55) | -0.08 | 110.01 (139.60) | - | 0.03 | 80.08 (116.11) | 70.14 (84.35) | 0.00 |
| Missing; n (%) | 1,152 (9.2%) | 33 (8.2%) | 0.04 | 1,835 (9.7%) | 72 (9.9%) | -0.01 | 4,098 (6.3%) | 65 (4.1%) | 0.10 | 7085 (7.3%) | 170 (6.3%) | 0.04 |
| Colonoscopy; n (%) | 379 (3.0%) | 15 (3.8%) | -0.04 | 650 (3.4%) | 21 (2.9%) | 0.03 | 2,246 (3.4%) | 52 (3.3%) | 0.01 | 3275 (3.4%) | 88 (3.2%) | 0.01 |
| Fecal occult blood (FOB) test; n (%) | 351 (2.8%) | 12 (3.0%) | -0.01 | 468 (2.5%) | 26 (3.6%) | -0.06 | 1,324 (2.0%) | 44 (2.8%) | -0.05 | 2143 (2.2%) | 82 (3.0%) | -0.05 |
| Flu vaccine; n (%) | 1,949 (15.5%) | 76 (19.0%) | -0.09 | 1.922 (10.2%) | 59 (8.1%) | 0.07 | 18,232 (27.9%) | 459 (28.8%) | -0.02 | 22103 (22.8%) | 594 (21.8%) | 0.02 |
| Mammogram: n (%) | | | | | | | | | | | | |
| | 1,257 (10.0%) | 32 (8.0%) | 0.07 | 1,747 (9.3%) | 66 (9.1%) | 0.01 | 6,822 (10.4%) | 174 (10.9%) | -0.02 | 9826 (10.1%) | 272 (10.0%) | 0.00 |
| Pap smear; n (%) Pneumonia vaccine; n (%) | | | 0.07<br>-0.13<br>-0.15 | 1,747 (9.3%)<br>1,059 (5.6%)<br>1,392 (7.4%) | 66 (9.1%)<br>43 (5.9%)<br>84 (11.6%) | 0.01<br>-0.01<br>-0.14 | | | -0.02<br>-0.05<br>-0.15 | | | 0.00<br>-0.06<br>-0.12 |

| PSA test or Prostate exam for DRE; n (%) | 1,248 (9.9%) | 45 (11.2%) | -0.04 | 1,603 (8.5%) | 52 (7.2%) | 0.05 | 6,723 (10.3%) | 213 (13.4%) | -0.10 | 9574 (9.9%) | 310 (11.4%) | -0.05 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Bone mineral density; n (%) | 424 (3.4%) | 11 (2.8%) | 0.03 | 301 (1.6%) | 7 (1.0%) | 0.05 | 2,616 (4.0%) | 75 (4.7%) | -0.03 | 3341 (3.4%) | 93 (3.4%) | 0.00 |
| Use of CNS stimulants; n (%) | 76 (0.6%) | 6 (1.5%) | -0.09 | 184 (1.0%) | 9 (1.2%) | -0.02 | 254 (0.4%) | 6 (0.4%) | 0.00 | 514 (0.5%) | 21 (0.8%) | -0.04 |
| Use of estrogens, progestins, androgens; n (%) | 610 (4.9%) | 29 (7.2%) | -0.10 | 1,772 (9.4%) | 93 (12.8%) | -0.11 | 1,683 (2.6%) | 63 (4.0%) | -0.08 | 4065 (4.2%) | 185 (6.8%) | -0.11 |
| Use of Angiogenesis inhibitors; n (%) | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 10 (0.1%) | 0 (0.0%) | 0.04 | 32 (0.0%) | 0 (0.0%) | #DIV/0! | 45 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Oral Immunosuppressants; n (%) | 15 (0.1%) | 1 (0.2%) | -0.03 | 52 (0.3%) | 2 (0.3%) | 0.00 | 42 (0.1%) | 2 (0.1%) | 0.00 | 109 (0.1%) | 5 (0.2%) | -0.03 |
| Use of fondaparinux or Bivalirudin; n (%) | 43 (0.3%) | 5 (1.2%) | -0.10 | 134 (0.7%) | 7 (1.0%) | -0.03 | 196 (0.3%) | 6 (0.4%) | -0.02 | 373 (0.4%) | 18 (0.7%) | -0.04 |
| Use of other direct thrombin inhibitors (lepirudin, | | | | | | | | | | | | |
| desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 7 (0.1%) | 1 (0.2%) | -0.03 | 8 (0.0%) | 2 (0.3%) | -0.08 | 3 (0.0%) | 1 (0.1%) | -0.04 | 18 (0.0%) | 4 (0.1%) | -0.04 |
| Use of Ticagrelor; n (%) | 14 (0.1%) | 1 (0.2%) | -0.03 | 15 (0.1%) | 4 (0.6%) | -0.08 | 63 (0.1%) | 5 (0.3%) | -0.04 | 92 (0.1%) | 10 (0.4%) | -0.06 |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.10 (0.35) | 0.24 (0.63) | -0.27 | 0.11 (0.38) | 0.14 (0.40) | -0.08 | 0.10 (0.33) | 0.15 (0.49) | -0.12 | 0.10 (0.34) | 0.16 (0.49) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | | |
| mean (sd) | 0.11 (0.52) | 0.10 (0.38) | 0.02 | 0.08 (0.41) | 0.08 (0.34) | 0.00 | 0.12 (0.55) | 0.13 (0.50) | -0.02 | 0.11 (0.52) | 0.11 (0.45) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | | | | | | |
| mean (sd) | 2.89 (4.03) | 0.83 (1.59) | 0.67 | 1.91 (3.27) | 0.56 (1.18) | 0.55 | 2.50 (4.13) | 0.52 (1.22) | 0.65 | 2.44 (3.96) | 0.58 (1.27) | 0.01 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.01) | 0.00 (0.00) | 0.00 | 0.00 (0.01) | 0.00 (0.00) | 0.00 | 0.00 (0.01) | 0.00 (0.00) | 0.00 | 0.00 (0.01) | 0.00 (0.00) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| mean (sd) | 2.61 (1.02) | 2.53 (1.04) | 0.08 | 2.15 (1.00) | 2.09 (1.01) | 0.06 | 3.22 (0.76) | 3.29 (0.81) | -0.09 | 2.93 (0.85) | 2.86 (0.90) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | | |
| mean (sd) | 16.82 (17.46) | 14.16 (17.42) | 0.15 | 12.61 (11.66) | 10.41 (11.48) | 0.19 | 17.66 (16.27) | 17.15 (15.14) | 0.03 | 16.57 (15.65) | 14.91 (14.63) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 2.26 (4.40) | 3.61 (5.24) | -0.28 | 2.19 (3.42) | 3.14 (3.34) | -0.28 | 2.54 (4.39) | 3.76 (4.92) | -0.26 | 2.44 (4.22) | 3.57 (4.60) | 0.00 |
| Use of clopidogrel ; n (%) | 378 (3.0%) | 12 (3.0%) | 0.00 | 446 (2.4%) | 14 (1.9%) | 0.03 | 3,206 (4.9%) | 103 (6.5%) | -0.07 | 4030 (4.2%) | 129 (4.7%) | -0.02 |
| Systemic embolism; n (%) | 301 (2.4%) | 4 (1.0%) | 0.11 | 364 (1.9%) | 17 (2.3%) | -0.03 | 1,097 (1.7%) | 24 (1.5%) | 0.02 | 1762 (1.8%) | 45 (1.7%) | 0.01 |
| DVT; n (%) | 9,006 (71.7%) | 284 (71.0%) | 0.02 | 14,258 (75.5%) | 531 (73.0%) | 0.06 | 48,425 (74.0%) | 1,249 (78.5%) | -0.11 | 71689 (74.0%) | 2064 (75.9%) | -0.04 |
| Post-thrombotic syndrome; n (%) | 68 (0.5%) | 4 (1.0%) | -0.06 | 66 (0.3%) | 4 (0.6%) | -0.04 | 164 (0.3%) | 7 (0.4%) | -0.02 | 66 (0.3%) | 4 (0.6%) | -0.04 |
| PE; n (%) | 6,185 (49.2%) | 189 (47.2%) | 0.04 | 8,051 (42.7%) | 336 (46.2%) | -0.07 | 27,050 (41.3%) | 615 (38.6%) | 0.06 | 41286 (42.6%) | 1140 (41.9%) | 0.01 |
| Coagulation defects; n (%) | 464 (3.7%) | 17 (4.2%) | -0.03 | 686 (3.6%) | 21 (2.9%) | 0.04 | 1,656 (2.5%) | 32 (2.0%) | 0.03 | 686 (3.6%) | 21 (2.9%) | 0.04 |
| Diabetes: 1 inpatient or 2 outpatient claims within | | | | | | | | | | | | |
| 183 days; n (%) | 2,289 (18.2%) | 48 (12.0%) | 0.17 | 2,570 (13.6%) | 69 (9.5%) | 0.13 | 15,045 (23.0%) | 354 (22.2%) | 0.02 | 19904 (20.5%) | 471 (17.3%) | 0.08 |
| Intracranial or retroperitoneal hemorrhage: 1 | | | | | | | | | | | | |
| inpatient or 2 outpatient claims within 183 days; n | | | | | | | | | | | | |
| (%) | 22 (0.2%) | 1 (0.2%) | 0.00 | 19 (0.1%) | 1 (0.1%) | 0.00 | 112 (0.2%) | 2 (0.1%) | 0.03 | 153 (0.2%) | 4 (0.1%) | 0.03 |
| Peptic Ulcer Disease; n (%) | 2,465 (19.6%) | 68 (17.0%) | 0.07 | 2,736 (14.5%) | 97 (13.3%) | 0.03 | 13,623 (20.8%) | 334 (21.0%) | 0.00 | 18824 (19.4%) | 499 (18.4%) | 0.03 |
| Upper GI bleed; n (%) | 9 (0.1%) | 0 (0.0%) | 0.04 | 14 (0.1%) | 0 (0.0%) | 0.04 | 49 (0.1%) | 1 (0.1%) | 0.00 | 72 (0.1%) | 1 (0.0%) | 0.04 |
| Lower/ unspecified GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Urogenital bleed; n (%) | 108 (0.9%) | 4 (1.0%) | -0.01 | 187 (1.0%) | 7 (1.0%) | 0.00 | 748 (1.1%) | 11 (0.7%) | 0.04 | 1043 (1.1%) | 22 (0.8%) | 0.03 |
| Other bleeds; n (%) | 98 (0.8%) | 0 (0.0%) | 0.13 | 144 (0.8%) | 2 (0.3%) | 0.07 | 359 (0.5%) | 6 (0.4%) | 0.01 | 601 (0.6%) | 8 (0.3%) | 0.04 |
| Prior cancer; n (%) | 1,312 (10.4%) | 46 (11.5%) | -0.04 | 1,457 (7.7%) | 68 (9.4%) | -0.06 | 8,553 (13.1%) | 279 (17.5%) | -0.12 | 11322 (11.7%) | 393 (14.5%) | -0.08 |
| Antibiotics; n (%) | 5,047 (40.2%) | 180 (45.0%) | #DIV/0! | 7,975 (42.3%) | 325 (44.7%) | -0.05 | 30,154 (46.1%) | 839 (52.7%) | | 7,975 (42.3%) | 325 (44.7%) | -0.05 |
| Aspirin; n (%) | 71 (0.6%) | 6 (1.5%) | -0.09 | 251 (1.3%) | 21 (2.9%) | -0.11 | 217 (0.3%) | 8 (0.5%) | -0.03 | 539 (0.6%) | 35 (1.3%) | -0.07 |
| Aspirin/dipyridamole; n (%) | 16 (0.1%) | 2 (0.5%) | -0.07 | 17 (0.1%) | 2 (0.3%) | -0.04 | 140 (0.2%) | 4 (0.3%) | -0.02 | 173 (0.2%) | 8 (0.3%) | -0.02 |
| Other antiplatelet agents; n (%) | 32 (0.3%) | 1 (0.2%) | 0.02 | 43 (0.2%) | 1 (0.1%) | 0.03 | 252 (0.4%) | 12 (0.8%) | -0.05 | 327 (0.3%) | 14 (0.5%) | -0.03 |
| PGP inhibitors; n (%) | 2,599 (20.7%) | 89 (22.2%) | -0.04 | 3,684 (19.5%) | 156 (21.5%) | -0.05 | 16,200 (24.8%) | 444 (27.9%) | -0.07 | 22483 (23.2%) | 689 (25.3%) | -0.05 |
| Other gastroprotective agents; n (%) | 120 (1.0%) | 4 (1.0%) | 0.00 | 192 (1.0%) | 9 (1.2%) | -0.02 | 817 (1.2%) | 28 (1.8%) | -0.05 | 1129 (1.2%) | 41 (1.5%) | -0.03 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.45 (0.70) | 0.48 (0.69) | -0.04 | 0.33 (0.68) | 0.30 (0.61) | 0.05 | 0.51 (0.73) | 0.57 (0.79) | -0.08 | 0.47 (0.72) | 0.48 (0.73) | 0.00 |
| Proton pump inhibitor; n (%) | 2,635 (21.0%) | 69 (17.2%) | 0.10 | 3,554 (18.8%) | 127 (17.5%) | 0.03 | 17,747 (27.1%) | 439 (27.6%) | -0.01 | 23936 (24.7%) | 635 (23.4%) | 0.03 |
| H2 receptor antagonist; n (%) | 428 (3.4%) | 10 (2.5%) | 0.05 | 563 (3.0%) | 24 (3.3%) | -0.02 | 3,668 (5.6%) | 88 (5.5%) | 0.00 | 4659 (4.8%) | 122 (4.5%) | 0.01 |
| Vitamin K therapy; n (%) | 13 (0.1%) | 0 (0.0%) | 0.04 | 23 (0.1%) | 0 (0.0%) | 0.04 | 50 (0.1%) | 1 (0.1%) | 0.00 | 86 (0.1%) | 1 (0.0%) | 0.04 |
| Number of INR (prothrombin) tests ordered | | | | | | | | | | | | |
| mean (sd) | 2.64 (3.88) | 0.47 (0.88) | 0.77 | 1.67 (3.11) | 0.35 (0.78) | 0.58 | 2.46 (4.10) | 0.46 (1.15) | 0.66 | 2.33 (3.90) | 0.43 (1.03) | 0.01 |
| Treating prescriber - Cardiologist; n (%) | 3,970 (31.6%) | 163 (40.8%) | -0.19 | 5,083 (26.9%) | 207 (28.5%) | -0.04 | 18,575 (28.4%) | 621 (39.0%) | -0.23 | 27628 (28.5%) | 991 (36.4%) | -0.17 |
| Treating prescriber - Primary Care Physician; n (%) | 9,946 (79.2%) | 327 (81.8%) | -0.07 | 7,669 (40.6%) | 267 (36.7%) | 0.08 | 22,033 (33.7%) | 596 (37.4%) | -0.08 | 39648 (40.9%) | 1190 (43.8%) | -0.06 |
| Treating prescriber - Other; n (%) | 11,618 (92.5%) | 387 (96.8%) | -0.19 | 17,713 (93.8%) | 696 (95.7%) | -0.09 | 60,900 (93.1%) | 1,563 (98.2%) | -0.25 | 90231 (93.1%) | 2646 (97.3%) | -0.20 |
| Alpha blockers; n (%) | 899 (7.2%) | 27 (6.8%) | 0.02 | 979 (5.2%) | 23 (3.2%) | 0.10 | 6,060 (9.3%) | 159 (10.0%) | -0.02 | 7938 (8.2%) | 209 (7.7%) | 0.02 |
| CHA2DS2 VASc score, 180 days, V | | | | | | | | | | | | |
| mean (sd) | 3.00 (1.87) | 1.87 (1.57) | 0.65 | 2.83 (1.83) | 1.72 (1.69) | 0.63 | 3.54 (1.80) | 2.80 (1.53) | 0.44 | 3.33 (1.82) | 2.37 (1.58) | 0.01 |
| Use of Prasugrel; n (%) | 11 (0.1%) | 1 (0.2%) | -0.03 | 28 (0.1%) | 0 (0.0%) | 0.04 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 39 (0.0%) | 1 (0.0%) | #DIV/0! |
| Use of Loop Diuretics+other diuretics+other | | | | | | | | | | | | |
| hypertension drugs; n (%) | 2,198 (17.5%) | 56 (14.0%) | 0.10 | 2,239 (11.9%) | 67 (9.2%) | 0.09 | 15,727 (24.0%) | 366 (23.0%) | 0.02 | 20164 (20.8%) | 489 (18.0%) | 0.07 |
| Commercial vs Medicare Advantage- Business Type | | | | | | | | | | | | |
| Code - CORRECT ONE - OPTUM | | | | | | | | | | | | |
| Commercial; n (%) | 4,542 (36.2%) | 213 (53.3%) | -0.35 | 5,181 (27.5%) | 164 (22.6%) | 0.11 | - | - | #VALUE! | 9,723 (30.9%) | 377 (33.5%) | -0.06 |
| Medicare Advantage; n (%) | 8,017 (63.8%) | 187 (46.8%) | 0.35 | 13,693 (72.5%) | 563 (77.4%) | -0.11 | | - | #VALUE! | 21,710 (69.1%) | 750 (66.5%) | 0.06 |
| Commercial vs Medicare Advantage- Business Type | | | | | | | | | | | | |
| Code | | | | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 4,542 (36.2%) | 213 (53.2%) | -0.35 | - | - | | - | - | #VALUE! | 4,542 (36.2%) | 213 (53.2%) | -0.35 |
| MCR = MEDICARE; n (%) | 8,017 (63.8%) | 187 (46.8%) | 0.35 | - | - | | - | - | #VALUE! | 8,017 (63.8%) | 187 (46.8%) | 0.35 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n | | | | | | | | | | | | |
| (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | | | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | | 12,101 (64.1%) | 426 (58.6%) | 0.11 | - | - | | 12,101 (64.1%) | 426 (58.6%) | 0.11 |

| 2 - Encounter; n (%) | - | - | 1,592 (8.4%) | 137 (18.8%) | -0.31 | | - | 1,592 (8.4%) | 137 (18.8%) | -0.31 |
|---|---|---|---|---|---|---|---|---|---|---|
| 3 - Medicare; n (%) | - | - | 4,564 (24.2%) | 150 (20.6%) | 0.09 | - | - | 4,564 (24.2%) | 150 (20.6%) | 0.09 |
| 4 - Medicare Encounter; n (%) | - | - | 617 (3.3%) | 14 (1.9%) | 0.09 | - | - | 617 (3.3%) | 14 (1.9%) | 0.09 |
| Metropolitan Statistical Area - Urban (any MSA) vs | | | | | | | | | | |
| Rural (non-MSA) | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | - | 13,765 (72.9%) | 528 (72.6%) | 0.01 | - | - | 13,765 (72.9%) | 528 (72.6%) | 0.01 |
| Rural; n (%) | - | - | 889 (4.7%) | 46 (6.3%) | -0.07 | - | - | 889 (4.7%) | 46 (6.3%) | -0.07 |
| Unknown/Missing; n (%) | - | - | 4,220 (22.4%) | 153 (21.0%) | 0.03 | - | - | 4,220 (22.4%) | 153 (21.0%) | 0.03 |

| March Marc | | | | | | PS-matched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Marche Marche Marche Marche Marche Marche March Marche Ma | | Opti | um | | MarketScan | | | Medicare | | | Reference warfarin | | |
| Part | Variable | WARFARIN Copy | Dabigatran 150mg Copy | St. Diff. Refe | erence - warfarin Copy e - Dal | bigatran 150mg Copy | St. Diff. Refe | rence - warfarin Copy e - Da | bigatran 150mg Copy | St. Diff. | | | St. Dif |
| March Marc | Number of patients | 387 | 387 | | 711 | 711 | | 1,577 | 1,577 | | 2,675 | 2,675 | |
| Marchand material part | 0 | | | | | | | | | | | | |
| 13 1-140-00 | | 61.91 (15.63) | 61.19 (15.85) | 0.05 | 55.73 (15.87) | 55.10 (15.33) | 0.04 | 76.00 (8.02) | 75.81 (7.72) | 0.02 | 68.57 (11.84) | 68.19 (11.57) | 0.03 |
| | | | | | | | | | - // | | | | |
| | | | | | | | | | | | | , | -0.0 |
| Prof. Prof | | | | | | | | | | | | | 0.03<br>-0.03 |
| Marche M | | | | | | | | | | | | | 0.0 |
| Memory M | | 00 (22.7%) | 80 (20.7%) | 0.03 | 33 (13.370) | 03 (11.770) | 0.07 | 788 (30.0%) | 791 (30.2%) | 0.00 | 373 (30.4%) | 554 (55.7%) | 0.0 |
| Part | | 201 (51.9%) | 188 (48.6%) | 0.07 | 385 (54.1%) | 376 (52.9%) | 0.02 | 630 (39.9%) | 629 (39.9%) | 0.00 | 1.216 (45.5%) | 1.193 (44.6%) | 0.0 |
| March Marc | | , | , | | | | | , | , | | | , , | -0.0 |
| | | () | () | | ( | | | (/ | 0 10 (001211) | | -, (, | _, ( , | |
| | White; n (%) | | | | | | | 1,409 (89.3%) | 1,401 (88.8%) | | 1,409 (89.3%) | 1,401 (88.8%) | 0.0 |
| | Black; n (%) | | | | | | | 103 (6.5%) | 105 (6.7%) | | 103 (6.5%) | 105 (6.7%) | 0.0 |
| Second Content | Asian; n (%) | | | | | | | 10 (0.6%) | 9 (0.6%) | | 10 (0.6%) | 9 (0.6%) | 0.0 |
| Second Processes 1985 19 | Hispanic; n (%) | | | | | | | | 22 (1.4%) | | 17 (1.1%) | 22 (1.4%) | 0.0 |
| Marchester Mar | | | | | | | | | | | | | 0.0 |
| Miller M | | | | | | | | 35 (2.2%) | 37 (2.3%) | | 35 (2.2%) | 37 (2.3%) | 0.0 |
| | | 52 (13 4%) | 43 (11.1%) | 0.07 | 162 (22.8%) | 165 (23.2%) | -0.01 | 371 (23.5%) | 379 (24.0%) | -0.01 | 585 (21 9%) | 587 (21 9%) | 0.0 |
| | | () | () | | () | | | () | (=) | | | | 0.0 |
| | | | | | | | | | | | | | -0.0 |
| | | | | -0.02 | | | -0.05 | 306 (19.4%) | 327 (20.7%) | -0.03 | | | -0.0 |
| Note | Unknown+missing; n (%) | | | #VALUE! | | | 0.03 | | | #VALUE! | | | 0.0 |
| March (N) 1 (2) (3) 1 (2) (3) (3) 1 (2) (3) (3) 1 (2) (3) (3 | | | | | , , | , , | | | | | , , | | |
| March Marc | Ischemic heart disease; n (%) | 56 (14.5%) | 42 (10.9%) | 0.11 | 69 (9.7%) | 70 (9.8%) | 0.00 | 314 (19.9%) | 319 (20.2%) | -0.01 | 439 (16.4%) | 431 (16.1%) | 0.01 |
| Clast State | Acute MI; n (%) | 2 (0.5%) | 1 (0.3%) | 0.03 | 5 (0.7%) | 4 (0.6%) | 0.01 | 14 (0.9%) | 12 (0.8%) | 0.01 | 21 (0.8%) | 17 (0.6%) | 0.02 |
| Stable engine (6) (6) (10, 20) | ACS/unstable angina; n (%) | 5 (1.3%) | 4 (1.0%) | 0.03 | 2 (0.3%) | 4 (0.6%) | -0.04 | 15 (1.0%) | 11 (0.7%) | 0.03 | 22 (0.8%) | 19 (0.7%) | 0.0 |
| Contact phenosteroses and other horse of chronic chr | Old MI; n (%) | 10 (2.6%) | 7 (1.8%) | 0.05 | 15 (2.1%) | 15 (2.1%) | 0.00 | 56 (3.6%) | 64 (4.1%) | -0.03 | 81 (3.0%) | 86 (3.2%) | -0.01 |
| Seminary (No. 10. 14. 12. 16. 16 | Stable angina; n (%) | 1 (0.3%) | 3 (0.8%) | -0.07 | 7 (1.0%) | 10 (1.4%) | -0.04 | 34 (2.2%) | 33 (2.1%) | 0.01 | 42 (1.6%) | 046 (1.7%) | -0.01 |
| Chee mentionate control (1940 or (1945 or (194 | | | | | | | | | | | | | |
| Productation procedure (PAG or PTCA or Steel) Product or Steel Product or Steel Procedure (PAG or PTCA or Steel) 13 (2.45) 3 (2.35) | | | , , | | | | | | | | | | 0.01 |
| | | 2 (0.5%) | 2 (0.5%) | 0.00 | 5 (0.7%) | 6 (0.8%) | -0.01 | 25 (1.6%) | 14 (0.9%) | 0.06 | 32 (1.2%) | 22 (0.8%) | 0.04 |
| Nichory (ASA OF PICK - P(K) 13 (4.8%) 91,2%) 12 (3.8%) 1.0 (3.8%) 1.1 (1.5%) 1.1 ( | | 4 (0.20() | 2 (0.50() | 0.00 | 2 (0 20() | 2 (2 20) | | F (0.20() | 0 (0 50) | 0.00 | 0 (0 20() | 43 (0.40() | 0.00 |
| Amy stroken, (nb) (1945) (1945 | | | | | | | | | | | | | -0.02<br>0.00 |
| Schemics stoke for any womention of cerebral infection of no final stoke for any womention of networks (%) (\$1 (4.0%)\$ \$1 (4.0%)\$ \$0 (0.0%)\$ \$0 (0.0%)\$ | | - (- ' / | , | | | | | | - ( , | | | | 0.0 |
| infarction (n (%) 19 (49%) 19 (49%) 10 (48%) 0.06 13 (1.8%) 13 (1.8%) 0.00 74 (47%) 75 (4.8%) 0.00 106 (4.0%) 102 (8.8%) 104 (1.0%) 10 | | 15 (4.570) | 14 (3.0%) | 0.00 | 13 (1.070) | 13 (1.0%) | 0.00 | 74 (4.770) | 73 (4.6%) | 0.00 | 100 (4.0%) | 102 (5.6%) | 0.0. |
| Nemorthage(stroken, Phj 0,00% 0, | | 19 (4.9%) | 14 (3.6%) | 0.06 | 13 (1.8%) | 13 (1.8%) | 0.00 | 74 (4.7%) | 75 (4.8%) | 0.00 | 106 (4.0%) | 102 (3.8%) | 0.01 |
| Tamp 1 | | | | | | | | | | | | | #DIV/0 |
| Ober cerebrowascular disease; n(b) 9(.2 %) 7(1.8 %) 0.04 12 (1.7 %) 13 (1.8 %) 0.03 14 (1.6 %) 10.1 %) 0.04 0.04 % 26.2 %) 47 (1.8 %) 1.0 | | | | | | | | | | | | | 0.03 |
| Cerebrosocalar procedure, (%) 0,00% 0,00 | | | | | | | | | | | | | 0.04 |
| Perplany Vancular Disasse (PVD) or PVD Surgery V2: | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 2 (0.1%) | 0.00 | 001 (0.0%) | 2 (0.1%) | -0.04 |
| 1 1 1 1 1 1 1 1 1 1 | Heart failure (CHF); n (%) | 34 (8.8%) | 28 (7.2%) | 0.06 | 37 (5.2%) | 40 (5.6%) | -0.02 | 181 (11.5%) | 188 (11.9%) | -0.01 | 252 (9.4%) | 256 (9.6%) | -0.01 |
| Arial final | Peripheral Vascular Disease (PVD) or PVD Surgery v2; | | | | | | | | | | | | |
| Other Cardiac orlyshythmin, 1% 76 (19.5%) 72 (18.6%) 0.03 110 (15.5%) 100 (14.1%) 0.04 305 (19.5%) 309 (19.5%) 0.01 315 (6.0%) 313 (6.0% | | | , | | | | | | | | | | 0.02 |
| Cardiac conduction disorders; n(%) 13 (3.4%) 20 (5.2%) 0.09 24 (3.4%) 15 (2.1%) 0.08 88 (6.2%) 39 (6.9%) 0.01 13 (6.0%) 128 (4.8%) 128 (4.8%) 10 (10 CMC VD; n) (6)% 78 (20.2%) 74 (19.1%) 0.03 76 (10.7%) 91 (3.1%) 0.07 278 (17.6%) 304 (19.3%) 0.04 432 (16.1%) 471 (17.6%) 70 (10 CMC VD; n) (6)% 74 (19.1%) 0.03 76 (10.7%) 12 (1.5%) 12 (1 | | 00 (=0,-) | (==, | | ( , - , | () | | () | | | | | 0.01 |
| Chec (CD), n (S) 78 (20.2%) 74 (19.1%) 76 (10.7%) 76 (10.7%) 93 (13.1%) -0.07 278 (17.5%) 304 (19.3%) -0.04 432 (16.1%) 471 (17.6%) -1.0% | | | | | | | | | | | | | 0.01 |
| Data Courrence Of Diabetic Neuropathy v2 Copy; n (%) 12 (3.8) 14 (3.6) | | - (- ' / | - ( / | | | | | , | | | | | 0.0 |
| Cocurrence of Diabetic Neuropathy V2 Copy; n (%) 11 (2.8%) 14 (3.6%) 2.0% 12 (1.7%) 11 (1.5%) 0.02 67 (4.2%) 59 (3.7%) 0.03 90 (3.4%) 84 (3.1%) Cocurrence of Diabetic Neuropathy V3 with ICD1 Copy; n (%) 0 (0.0%) mDiV/Ol 0 (0.0%) mDiV/Ol 10 (0.6%) 17 (1.1%) 0.05 10 (0.4%) 17 (0.6%) 17 (1.1%) 0.05 10 (0.4%) 17 (0.6%) 17 (1.1%) 0.05 10 (0.4%) 17 (1.1%) 0.05 0.04 0.05 0.04 0.05 0.04 0.05 0.04 0.05 0.04 0.05 0.04 0.05 0 | | /8 (20.2%) | 74 (19.1%) | 0.03 | 76 (10.7%) | 93 (13.1%) | -0.07 | 2/8 (17.6%) | 304 (19.3%) | -0.04 | 432 (16.1%) | 4/1 (17.6%) | -0.04 |
| Courrence of diabetic nephropathy V3 with ICD10 Copyr, (%) 0.0 (0.0%) 0.0 (0.0%) 10.0%) 0.0 (0.0%) 10.0%) 10.06% 17 (1.1%) 0.05 10.0.4% 17 (0.6%) 17 | | 44 (2.00() | 44/2 50/1 | 0.05 | 42 (4 70() | 44 (4 50() | 0.00 | 57 (4.20() | 50 (2.70() | | 00 (2.40() | 04 (2.40() | 0.00 |
| Copy, n(s) 0 (0.0%) 0 (0.0%) 1 (0.0%) 1 (0.0%) 1 (0.0%) 1 (0.0%) 0 (0.0%) 1 | | 11 (2.8%) | 14 (3.6%) | -0.05 | 12 (1.7%) | 11 (1.5%) | 0.02 | b/ (4.2%) | 59 (3.7%) | 0.03 | 90 (3.4%) | 84 (3.1%) | 0.0 |
| Hypoglycemia v2; n (%) 1 (0.3%) 1 (0.3%) 1 (0.3%) 1 (0.3%) 1 (0.4%) 0.12 20 (2.8%) 24 (3.5%) 0.02 31 (2.0%) 24 (1.5%) 0.04 35 (1.3%) 27 (1.0%) 1 (0.6%) 1 (0.6%) 1 (0.6%) 1 (0.6%) 1 (0.6%) 1 (0.6%) 1 (0.6%) 1 (0.5%) 1 | | 0 (0 0%) | 0 (0 0%) | #DIV/01 | 0 (0 0%) | 0 (0 0%) | #DIV/01 | 10 (0 69/) | 17 /1 10/\ | 0.05 | 10 (0.49/) | 17 (0 69/) | -0.03 |
| Hyperglycemia; n (%) 28 (7.2%) 17 (4.4%) 0.12 20 (2.8%) 24 (3.4%) -0.03 134 (8.5%) 135 (8.5%) 0.00 182 (6.8%) 176 (6.5%) 10abetic ketoacidosis; n (%) 0.00%) 0.00% | | | | | | | | | | | | | 0.0 |
| Diabetic ketoacidosis; n(%) 0 (0.0%) 0 (0.0%) #DIV/0! 1 (0.1%) 0 (0.0%) 0 ( | | | | | | | | | | 0.04 | | | 0.0: |
| Hypertension: 1 inpatient or 2 outpatient claims within 355 days, n (%) 208 (53.7%) 212 (54.8%) -0.02 271 (38.1%) 259 (36.4%) 0.04 1,224 (77.6%) 1,189 (75.4%) 0.05 1,703 (63.7%) 1,660 (62.1%) Hyperlipidemialy 2'; n (%) 157 (40.6%) 154 (39.8%) 0.02 200 (28.1%) 192 (27.0%) 0.02 758 (48.1%) 765 (48.5%) -0.01 1,115 (41.7%) 1,111 (41.5%) Edema; n (%) 99 (25.6%) 89 (23.0%) 0.06 134 (18.8%) 127 (17.9%) 0.02 376 (23.8%) 355 (22.5%) 0.03 609 (22.8%) 571 (21.3%) Renal Dysfunction (non-diabetic) v2; n (%) 0 (0.0%) 10 (0.0%) 10 (0.0%) 10 (1.1%) 1 (0.1%) 2 (0.3%) -0.04 2 (0.1%) 3 (0.2%) -0.03 3 (0.1%) 5 (0.2%) Occurrence of chronic renal insufficiency; n (%) 0 (0.0%) 10 | | () | () | | == (=:=:-) | ( ) | | (, | () | | | | 0.00 |
| within 365 days, n (%) | | 0 (0.0%) | 0 (0.070) | | 1 (0.170) | 0 (0.070) | 5.04 | 2 (0.170) | 2 (0.1/0) | 0.00 | 3 (0.1/0) | 02 (0.176) | 0.00 |
| Hyperfipidemia v2; n (%) | | 208 (53.7%) | 212 (54.8%) | -0.02 | 271 (38.1%) | 259 (36.4%) | 0.04 | 1,224 (77.6%) | 1,189 (75.4%) | 0.05 | 1,703 (63.7%) | 1,660 (62.1%) | 0.03 |
| Edema; n (%) 99 (25.6%) 89 (23.0%) 0.06 134 (18.8%) 127 (17.9%) 0.02 376 (23.8%) 355 (22.5%) 0.03 609 (22.8%) 571 (21.3%) 8enal Dysfunction (non-diabetic) v2; n (%) 0 (0.0%) 0 (0.0%) #DIV/0! 1 (0.1%) 2 (0.3%) -0.04 2 (0.1%) 3 (0.2%) -0.03 3 (0.1%) 5 (0.2%) 0 (0.0%) 10 (0.0%) | | | | | | | | , , , , , , | | | | | 0.00 |
| Occurrence of acture renal disease v2; n(\$) 0 (0.0%) 0 (0.0%) #DIV/0! 1 (0.1%) 0.00 1 (0.1%) 2 (0.1%) 0.00 2 (0.1%) 3 (0.1%) 3 (0.1%) Courrence of chronic renal insufficiency; n(\$) 0 (0.0%) #DIV/0! | Edema; n (%) | 99 (25.6%) | 89 (23.0%) | 0.06 | 134 (18.8%) | 127 (17.9%) | 0.02 | 376 (23.8%) | 355 (22.5%) | 0.03 | | | 0.04 |
| Occurrence of acture renal disease v2; n(\$) 0 (0.0%) 0 (0.0%) #DIV/0! 1 (0.1%) 0.00 1 (0.1%) 2 (0.1%) 0.00 2 (0.1%) 3 (0.1%) 3 (0.1%) Courrence of chronic renal insufficiency; n(\$) 0 (0.0%) #DIV/0! | Renal Dysfunction (non-diabetic) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 2 (0.3%) | -0.04 | 2 (0.1%) | 3 (0.2%) | -0.03 | 3 (0.1%) | 5 (0.2%) | -0.0 |
| Chronic kidney disease v2; n (%) 0 (0.0%) 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0 | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.1%) | 2 (0.1%) | 0.00 | 2 (0.1%) | 3 (0.1%) | 0.00 |
| CKD Stage 3-4'; n (%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) #DIV/O! 0 (0.0% | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0 |
| Occurrence of hypertensive nephropathy; $n$ (%) $0$ (0.0%) $0$ (0 | | - ( , | | , | , | - ( / | | - () | | | - ( / | , | #DIV/0 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) 0 (0.0%) 0 (0.0%) #DIV/O! 0 (0.0%) 1 (0.1%) -0.04 1 (0.1%) 1 (0.1%) 0.00 1 (0.0%) 2 (0.1%) Other Covariates | | - ( , | | , | , | - ( / | , | , | | | - ( / | , | #DIV/0 |
| $ (\%) \qquad 0 \ (0.0\%) \qquad 0 \ (0.0\%) \qquad \# \text{DIV}/0! \qquad 0 \ (0.0\%) \qquad 1 \ (0.1\%) \qquad -0.04 \qquad 1 \ (0.1\%) \qquad 1 \ (0.1\%) \qquad 0.00 \qquad 1 \ (0.0\%) \qquad 2 \ (0.1\%) $ Other Covariates | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0 |
| Other Covariates | | | | | | | | | | | | | |
| | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 1 (0.1%) | -0.04 | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.0%) | 2 (0.1%) | -0.04 |
| Liver disease; $n(\%)$ 1 (0.3%) 1 (0.3%) 0.00 2 (0.3%) 3 (0.4%) -0.02 6 (0.4%) 7 (0.4%) 0.00 9 (0.3%) 11 (0.4%) | | | | | | | | | | | | | |
| Osteoarthritis; n(%) 100 (25.8%) 93 (24.0%) 0.04 124 (17.4%) 123 (17.3%) 0.00 510 (32.3%) 501 (31.8%) 0.01 734 (27.4%) 717 (26.8%) | | | | | | | | - () | . () | | | | -0.02<br>0.03 |

| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pain: n (%) | 291 (75.2%) | 279 (72.1%) | 0.07 | 502 (70.6%) | 479 (67.4%) | 0.07 | 1,078 (68.4%) | 1.041 (66.0%) | 0.05 | 1871 (69.9%) | 1799 (67.3%) | 0.06 |
| Dorsopathies; n (%) | 132 (34.1%) | 120 (31.0%) | 0.07 | 178 (25.0%) | 178 (25.0%) | 0.00 | 449 (28.5%) | 449 (28.5%) | 0.00 | 759 (28.4%) | 747 (27.9%) | 0.01 |
| Fractures; n (%) | 37 (9.6%) | 37 (9.6%) | 0.00 | 52 (7.3%) | 52 (7.3%) | 0.00 | 145 (9.2%) | 143 (9.1%) | 0.00 | 234 (8.7%) | 232 (8.7%) | 0.00 |
| Falls v2; n (%) | 42 (10.9%) | 33 (8.5%) | 0.08 | 30 (4.2%) | 30 (4.2%) | 0.00 | 74 (4.7%) | 73 (4.6%) | 0.00 | 146 (5.5%) | 136 (5.1%) | 0.02 |
| Osteoporosis; n (%) | 19 (4.9%) | 19 (4.9%) | 0.00 | 18 (2.5%) | 19 (2.7%) | -0.01 | 161 (10.2%) | 160 (10.1%) | 0.00 | 198 (7.4%) | 198 (7.4%) | 0.00 |
| Depression: n (%) | 55 (14.2%) | 51 (13.2%) | 0.03 | 56 (7.9%) | 65 (9.1%) | -0.04 | 217 (13.8%) | 213 (13.5%) | 0.01 | 328 (12.3%) | 329 (12.3%) | 0.00 |
| Anxiety: n (%) | 60 (15.5%) | 60 (15.5%) | 0.00 | 74 (10.4%) | 78 (11.0%) | -0.02 | 209 (13.3%) | 206 (13.1%) | 0.01 | 343 (12.8%) | 344 (12.9%) | 0.00 |
| Sleep_Disorder; n (%) | 8 (2.1%) | 11 (2.8%) | -0.05 | 27 (3.8%) | 28 (3.9%) | -0.01 | 51 (3.2%) | 57 (3.6%) | -0.02 | 86 (3.2%) | 96 (3.6%) | -0.02 |
| Dementia; n (%) | 24 (6.2%) | 22 (5.7%) | 0.02 | 30 (4.2%) | 31 (4.4%) | -0.01 | 196 (12.4%) | 196 (12.4%) | 0.00 | 250 (9.3%) | 249 (9.3%) | 0.00 |
| Delirium; n (%) | 11 (2.8%) | 7 (1.8%) | 0.07 | 12 (1.7%) | 11 (1.5%) | 0.02 | 60 (3.8%) | 60 (3.8%) | 0.00 | 83 (3.1%) | 78 (2.9%) | 0.01 |
| Psychosis; n (%) | 6 (1.6%) | 8 (2.1%) | -0.04 | 3 (0.4%) | 3 (0.4%) | 0.00 | 34 (2.2%) | 33 (2.1%) | 0.01 | 43 (1.6%) | 44 (1.6%) | 0.00 |
| Obesity; n (%) | 99 (25.6%) | 86 (22.2%) | 0.08 | 136 (19.1%) | 132 (18.6%) | 0.01 | 235 (14.9%) | 239 (15.2%) | -0.01 | 470 (17.6%) | 457 (17.1%) | 0.01 |
| Overweight; n (%) | 29 (7.5%) | 22 (5.7%) | 0.07 | 27 (3.8%) | 24 (3.4%) | 0.02 | 62 (3.9%) | 58 (3.7%) | 0.01 | 118 (4.4%) | 104 (3.9%) | 0.03 |
| Smoking; n (%) | 91 (23.5%) | 92 (23.8%) | -0.01 | 82 (11.5%) | 85 (12.0%) | -0.02 | 448 (28.4%) | 442 (28.0%) | 0.01 | 621 (23.2%) | 619 (23.1%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/01 |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| COPD; n (%) | 57 (14.7%) | 48 (12.4%) | 0.07 | 45 (6.3%) | 43 (6.0%) | 0.01 | 292 (18.5%) | 280 (17.8%) | 0.02 | 394 (14.7%) | 371 (13.9%) | 0.02 |
| Asthma; n (%) | 43 (11.1%) | 43 (11.1%) | 0.00 | 35 (4.9%) | 45 (6.3%) | -0.06 | 163 (10.3%) | 134 (8.5%) | 0.06 | 241 (9.0%) | 222 (8.3%) | 0.02 |
| Obstructive sleep apnea; n (%) | 49 (12.7%) | 43 (11.1%) | 0.05 | 47 (6.6%) | 54 (7.6%) | -0.04 | 113 (7.2%) | 118 (7.5%) | -0.01 | 209 (7.8%) | 215 (8.0%) | -0.01 |
| Pneumonia: n (%) | 37 (9.6%) | 37 (9.6%) | 0.00 | 49 (6.9%) | 56 (7.9%) | -0.04 | 152 (9.6%) | 142 (9.0%) | 0.02 | 238 (8.9%) | 235 (8.8%) | 0.00 |
| Other Medications | 37 (3.0%) | 37 (3.0%) | 0.00 | 45 (0.5%) | 30 (7.5%) | -0.04 | 132 (5.0%) | 142 (5.0%) | 0.02 | 230 (0.370) | 233 (0.0%) | 0.00 |
| Use of ACE inhibitors; n (%) | 77 (19.9%) | 75 (19.4%) | 0.01 | 90 (12.7%) | 98 (13.8%) | -0.03 | 381 (24.2%) | 397 (25.2%) | -0.02 | 548 (20.5%) | 570 (21.3%) | -0.02 |
| Use of ARBs: n (%) | 36 (9.3%) | 41 (10.6%) | -0.04 | 88 (12.4%) | 71 (10.0%) | 0.08 | 307 (19.5%) | 304 (19.3%) | 0.01 | 431 (16.1%) | 416 (15.6%) | 0.02 |
| Use of Loop Diuretics - United; n (%) | 36 (9.3%)<br>44 (11.4%) | 41 (10.6%)<br>37 (9.6%) | -0.04 | 88 (12.4%)<br>56 (7.9%) | 71 (10.0%)<br>48 (6.8%) | 0.08 | 307 (19.5%) | 304 (19.3%)<br>292 (18.5%) | 0.01 | 431 (16.1%) 407 (15.2%) | 416 (15.6%)<br>377 (14.1%) | 0.01 |
| | , , , | | | | | | | | | | | |
| Use of other diuretics- United; n (%) | 4 (1.0%) | 8 (2.1%) | -0.09 | 9 (1.3%) | 8 (1.1%) | 0.02 | 38 (2.4%) | 55 (3.5%) | -0.07 | 51 (1.9%) | 71 (2.7%) | -0.05 |
| Use of nitrates-United; n (%) | 2 (0.5%) | 3 (0.8%) | -0.04 | 6 (0.8%) | 10 (1.4%) | -0.06 | 95 (6.0%) | 78 (4.9%) | 0.05 | 103 (3.9%) | 91 (3.4%) | 0.03 |
| Use of other hypertension drugs; n (%) | 16 (4.1%) | 16 (4.1%) | 0.00 | 10 (1.4%) | 13 (1.8%) | -0.03 | 80 (5.1%) | 79 (5.0%) | 0.00 | 106 (4.0%) | 108 (4.0%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 6 (1.6%) | 5 (1.3%) | 0.03 | 14 (2.0%) | 14 (2.0%) | 0.00 | 47 (3.0%) | 42 (2.7%) | 0.02 | 67 (2.5%) | 61 (2.3%) | 0.01 |
| Use of COPD/asthma meds- United; n (%) | 60 (15.5%) | 59 (15.2%) | 0.01 | 102 (14.3%) | 108 (15.2%) | -0.03 | 361 (22.9%) | 330 (20.9%) | 0.05 | 523 (19.6%) | 497 (18.6%) | 0.03 |
| Use of statins; n (%) | 128 (33.1%) | 119 (30.7%) | 0.05 | 155 (21.8%) | 153 (21.5%) | 0.01 | 633 (40.1%) | 638 (40.5%) | -0.01 | 916 (34.2%) | 910 (34.0%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 23 (5.9%) | 20 (5.2%) | 0.03 | 21 (3.0%) | 19 (2.7%) | 0.02 | 88 (5.6%) | 87 (5.5%) | 0.00 | 132 (4.9%) | 126 (4.7%) | 0.01 |
| Use of antiplatelet agents; n (%) | 26 (6.7%) | 20 (5.2%) | 0.06 | 49 (6.9%) | 40 (5.6%) | 0.05 | 163 (10.3%) | 135 (8.6%) | 0.06 | 238 (8.9%) | 195 (7.3%) | 0.06 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | | |
| heparins; n (%) | 79 (20.4%) | 93 (24.0%) | -0.09 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 289 (18.3%) | 297 (18.8%) | -0.01 | 368 (13.8%) | 390 (14.6%) | -0.02 |
| Use of NSAIDs; n (%) | 81 (20.9%) | 76 (19.6%) | 0.03 | 157 (22.1%) | 156 (21.9%) | 0.00 | 266 (16.9%) | 277 (17.6%) | -0.02 | 504 (18.8%) | 509 (19.0%) | -0.01 |
| Use of oral corticosteroids; n (%) | 115 (29.7%) | 94 (24.3%) | 0.12 | 169 (23.8%) | 174 (24.5%) | -0.02 | 455 (28.9%) | 454 (28.8%) | 0.00 | 739 (27.6%) | 722 (27.0%) | 0.01 |
| Use of bisphosphonate (United); n (%) | 6 (1.6%) | 8 (2.1%) | -0.04 | 4 (0.6%) | 9 (1.3%) | -0.07 | 56 (3.6%) | 53 (3.4%) | 0.01 | 66 (2.5%) | 70 (2.6%) | -0.01 |
| Use of opioids- United; n (%) | 148 (38.2%) | 155 (40.1%) | -0.04 | 310 (43.6%) | 295 (41.5%) | 0.04 | 613 (38.9%) | 630 (39.9%) | -0.02 | 1071 (40.0%) | 1080 (40.4%) | -0.01 |
| Use of antidepressants; n (%) | 91 (23.5%) | 90 (23.3%) | 0.00 | 138 (19.4%) | 147 (20.7%) | -0.03 | 458 (29.0%) | 465 (29.5%) | -0.01 | 687 (25.7%) | 702 (26.2%) | -0.01 |
| Use of antipsychotics; n (%) | 10 (2.6%) | 16 (4.1%) | -0.08 | 14 (2.0%) | 15 (2.1%) | -0.01 | 93 (5.9%) | 77 (4.9%) | 0.04 | 117 (4.4%) | 108 (4.0%) | 0.02 |
| Labs | | | | | | | | | | 1,098 | 1,098 | |
| Lab values- HbA1c (%) v3; n (%) | 47 (12.1%) | 40 (10.3%) | 0.06 | 4 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 051 (4.6%) | 043 (3.9%) | 0.03 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 29 (7.5%) | 26 (6.7%) | 0.03 | 2 (0.3%) | 1 (0.1%) | 0.04 | N/A | N/A | #VALUE! | 031 (2.8%) | 027 (2.5%) | 0.02 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 47 (12.1%) | 40 (10.3%) | 0.06 | 4 (0.6%) | 3 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 051 (4.6%) | 043 (3.9%) | 0.03 |
| Lab values- BNP; n (%) | 4 (1.0%) | 8 (2.1%) | -0.09 | 1 (0.1%) | 2 (0.3%) | -0.04 | N/A | N/A | #VALUE! | 5 (0.5%) | 10 (0.9%) | -0.05 |
| Lab values- BNP (within 3 months); n (%) | 4 (1.0%) | 4 (1.0%) | 0.00 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 04 (0.4%) | 05 (0.5%) | -0.01 |
| Lab values- BNP (within 6 months); n (%) | 4 (1.0%) | 8 (2.1%) | -0.09 | 1 (0.1%) | 2 (0.3%) | -0.04 | N/A | N/A | #VALUE! | 5 (0.5%) | 10 (0.9%) | -0.05 |
| Lab values- BUN (mg/dl); n (%) | 94 (24.3%) | 118 (30.5%) | -0.14 | 5 (0.7%) | 6 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 099 (9.0%) | 124 (11.3%) | -0.08 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 68 (17.6%) | 82 (21.2%) | -0.09 | 2 (0.3%) | 4 (0.6%) | -0.04 | N/A | N/A | #VALUE! | 070 (6.4%) | 086 (7.8%) | -0.05 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 94 (24.3%) | 118 (30.5%) | -0.14 | 5 (0.7%) | 6 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 099 (9.0%) | 124 (11.3%) | -0.08 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 98 (25.3%) | 123 (31.8%) | -0.14 | 5 (0.7%) | 6 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 103 (9.4%) | 129 (11.7%) | -0.07 |
| Lab values-Creatinine (mg/dl) (within 3 months) v2; | | | | | | | | | | | | |
| n (%) | 70 (18.1%) | 88 (22.7%) | -0.11 | 2 (0.3%) | 4 (0.6%) | -0.04 | N/A | N/A | #VALUE! | 072 (6.6%) | 092 (8.4%) | -0.07 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | | | | | | | | | | | | |
| n (%) | 98 (25.3%) | 123 (31.8%) | -0.14 | 5 (0.7%) | 6 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 103 (9.4%) | 129 (11.7%) | -0.07 |
| Lab values- HDL level (mg/dl); n (%) | 64 (16.5%) | 72 (18.6%) | -0.06 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 067 (6.1%) | 075 (6.8%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 36 (9.3%) | 43 (11.1%) | -0.06 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 036 (3.3%) | 044 (4.0%) | -0.04 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 64 (16.5%) | 72 (18.6%) | -0.06 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 067 (6.1%) | 075 (6.8%) | -0.03 |
| Lab values- LDL level (mg/dl) v2; n (%) | 69 (17.8%) | 72 (18.6%)<br>75 (19.4%) | -0.04 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A<br>N/A | #VALUE! | 072 (6.6%) | 075 (6.8%) | -0.03 |
| | 09 (17.8%) | 75 (19.4%) | -0.04 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 072 (0.0%) | 078 (7.1%) | -0.02 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n<br>(%) | 39 (10.1%) | 47 (12.1%) | -0.06 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 039 (3.6%) | 048 (4.4%) | -0.04 |
| | 39 (10.1%) | 47 (12.1%) | -0.06 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 039 (3.6%) | 048 (4.4%) | -0.04 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n<br>(%) | 69 (17.8%) | 75 (19.4%) | -0.04 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 072 (6.6%) | 078 (7.1%) | -0.02 |
| . , | | | -0.04<br>0.10 | | | 0.00<br>#DIV/0! | | | #VALUE! | | | |
| Lab values-NT-proBNP; n (%)<br>Lab values-NT-proBNP (within 3 months); n (%) | 2 (0.5%) | 0 (0.0%) | 0.10 | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | N/A | N/A<br>N/A | #VALUE! | 02 (0.2%) | 0 (0.0%) | 0.06 |
| | 2 (0.5%) | 0 (0.0%) | | | , | | N/A | | | 02 (0.2%) | 0 (0.0%) | |
| Lab values- NT-proBNP (within 6 months); n (%) | 2 (0.5%) | 0 (0.0%) | 0.10 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 02 (0.2%) | 0 (0.0%) | |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 68 (17.6%) | 75 (19.4%) | -0.05 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 071 (6.5%) | 078 (7.1%) | -0.02 |
| Lab values-Total cholesterol (mg/dl) (within 3 | 40 (10.3%) | 47 (43 40/) | -0.06 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | 81/8 | #VALUE! | 040/2 (0/) | 049 (4 49/) | -0.04 |
| months) v2; n (%) | 40 (10.5%) | 47 (12.1%) | -U.Ub | u (U.U%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 040 (3.6%) | 048 (4.4%) | -0.04 |
| Lab values-Total cholesterol (mg/dl) (within 6 months) v2; n (%) | 68 (17.6%) | 75 (19.4%) | -0.05 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 071 (6.5%) | 078 (7.1%) | -0.02 |
| Lab values- Triglyceride level (mg/dl); n (%) | 67 (17.3%) | 75 (19.4%) | -0.05 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 070 (6.4%) | 078 (7.1%) | -0.03 |
| Lab values-Triglyceride level (mg/dl) (within 3 | 20 (0.00/) | 47 (12 10() | 0.07 | 0 (0 00/) | 1 (0.181) | 0.04 | N/c | A1/* | 40/011151 | 030/3.50/ | 049 (4.40) | 0.05 |
| months); n (%) | 38 (9.8%) | 47 (12.1%) | -0.07 | 0 (0.0%) | 1 (0.1%) | -0.04 | N/A | N/A | #VALUE! | 038 (3.5%) | 048 (4.4%) | -0.05 |

| Lab colores Taighteenide Level (as a (dl.) (cristina C | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lab values-Triglyceride level (mg/dl) (within 6<br>months): n (%) | 67 (17.3%) | 75 (19.4%) | -0.05 | 3 (0.4%) | 3 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 070 (6.4%) | 078 (7.1%) | -0.03 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | 07 (17.370) | 75 (15.470) | -0.03 | 3 (0.470) | 3 (0.470) | 0.00 | N/A | 19/5 | #VALUE: | 070 (0.470) | 070 (7.170) | -0.03 |
| included) v4 | 46 | 40 | | 4 | 3 | | N/A | N/A | | 50 | 43 | |
| mean (sd) | 6.11 (0.94) | 6.19 (0.74) | -0.09 | 7.34 (2.56) | 5.93 (0.40) | 0.77 | N/A | N/A | #VALUE! | 6.21 (1.12) | 6.17 (0.74) | 0.04 |
| Missing; n (%) | 341 (88.1%) | 347 (89.7%) | -0.05 | 707 (99.4%) | 708 (99.6%) | -0.03 | N/A | N/A | #VALUE! | 1,048 (95.4%) | 1,055 (96.1%) | -0.03 |
| | 341 (00.1/0) | 347 (05.7%) | -0.03 | 707 (55.470) | 708 (55.0%) | -0.03 | N/A | N/A | #VALUE: | 1,040 (55.470) | 1,033 (50.1%) | -0.03 |
| Lab result number- BNP mean v2 | 409.35 (561.34) | 134.34 (166.13) | 0.66 | 205.00 (0.00) | 0.00 (0.00) | #DIV/0! | N/A<br>N/A | N/A<br>N/A | #VALUE! | 368.48 (687.50) | 107.47 (166.13) | 0.52 |
| mean (sd) | | | | | | | | , | | | | |
| Missing; n (%) | 383 (99.0%) | 379 (97.9%) | 0.09 | 710 (99.9%) | 709 (99.7%) | 0.04 | N/A | N/A | #VALUE! | 1,093 (99.5%) | 1,088 (99.1%) | 0.05 |
| Lab result number- BUN (mg/dl) mean v2 | 94 | 118 | | 5 | 6 | | N/A | N/A | | 99 | 124 | |
| mean (sd) | 15.63 (5.02) | 16.18 (5.23) | -0.11 | 13.50 (2.60) | 13.88 (2.72) | -0.14 | N/A | N/A | #VALUE! | 15.52 (4.97) | 16.07 (5.17) | -0.11 |
| Missing; n (%) | 293 (75.7%) | 269 (69.5%) | 0.14 | 706 (99.3%) | 705 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 999 (91.0%) | 974 (88.7%) | 0.08 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | | | | |
| to 15 included) v3 | 97 | 123 | | 5 | 6 | | N/A | N/A | | 102 | 129 | |
| mean (sd) | 0.90 (0.21) | 0.92 (0.19) | -0.10 | 0.97 (0.17) | 0.87 (0.14) | 0.64 | N/A | N/A | #VALUE! | 0.90 (0.21) | 0.92 (0.19) | -0.10 |
| Missing; n (%) | 290 (74.9%) | 264 (68.2%) | 0.15 | 706 (99.3%) | 705 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 996 (90.7%) | 969 (88.3%) | 0.08 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 64 | 72 | | 3 | 3 | | N/A | N/A | | 67 | 75 | |
| mean (sd) | 51.78 (16.46) | 55.23 (14.10) | -0.23 | 49.00 (3.00) | 53.67 (10.26) | -0.62 | N/A | N/A | #VALUE! | 51.66 (16.34) | 55.17 (14.11) | -0.23 |
| Missing; n (%) | 323 (83.5%) | 315 (81.4%) | 0.06 | 708 (99.6%) | 708 (99.6%) | 0.00 | N/A | N/A | #VALUE! | 1,031 (93.9%) | 1,023 (93.2%) | 0.03 |
| Lab result number-LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 68 | 73 | | 3 | 3 | | N/A | N/A | | 71 | 76 | |
| mean (sd) | 102.65 (33.30) | 103.87 (37.38) | -0.03 | 95.00 (38.22) | 104.33 (41.40) | -0.23 | N/A | N/A | #VALUE! | 102.33 (33.70) | 103.89 (37.75) | -0.04 |
| Missing; n (%) | 319 (82.4%) | 314 (81.1%) | 0.03 | 708 (99.6%) | 708 (99.6%) | 0.00 | N/A | N/A | #VALUE! | 1,027 (93.5%) | 1,022 (93.1%) | 0.02 |
| Lab result number-Total cholesterol (mg/dl) mean | 313 (02.470) | 514 (61.176) | 0.05 | 700 (55.0%) | 700 (33.0%) | 0.00 | 14/1 | 14/1 | WWW.COC. | 1,027 (33.370) | 1,022 (55.170) | 0.02 |
| (only =<5000 included) v2 | 68 | 75 | | 3 | 3 | | N/A | N/A | | 71 | 78 | |
| mean (sd) | 178.75 (41.17) | 188.01 (40.02) | -0.23 | 172.33 (50.64) | 187.67 (27.61) | -0.38 | N/A | N/A | #VALUE! | 178.48 (41.78) | 188.00 (40.01) | -0.23 |
| * * | | | | | | 0.00 | | | #VALUE! | | | 0.02 |
| Missing; n (%) | 319 (82.4%) | 312 (80.6%) | 0.05 | 708 (99.6%) | 708 (99.6%) | 0.00 | N/A | N/A | #VALUE! | 1,027 (93.5%) | 1,020 (92.9%) | 0.02 |
| Lab result number-Triglyceride level (mg/dl) mean | | 75 | | | | | *** | **/* | | 70 | 70 | |
| (only =<5000 included) v2 | 67 | 75 | | 3 | 3 | | N/A | N/A | | 70 | 78 | |
| mean (sd) | 130.80 (70.14) | 144.53 (92.96) | -0.17 | 136.33 (91.88) | 147.00 (50.86) | -0.14 | N/A | N/A | #VALUE! | 131.04 (71.40) | 144.63 (92.71) | -0.16 |
| Missing; n (%) | 320 (82.7%) | 312 (80.6%) | 0.05 | 708 (99.6%) | 708 (99.6%) | 0.00 | N/A | N/A | #VALUE! | 1,028 (93.6%) | 1,020 (92.9%) | 0.03 |
| Lab result number-Hemoglobin mean (only >0 | | | | | | | | | | | | |
| included) | 86 | 101 | | 4 | 6 | | N/A | N/A | | 90 | 107 | |
| mean (sd) | 13.61 (1.76) | 13.96 (1.61) | -0.21 | 13.50 (2.64) | 13.42 (1.17) | 0.04 | N/A | N/A | #VALUE! | 13.61 (1.81) | 13.93 (1.60) | -0.19 |
| Missing; n (%) | 301 (77.8%) | 286 (73.9%) | 0.09 | 707 (99.4%) | 705 (99.2%) | 0.02 | N/A | N/A | #VALUE! | 1,008 (91.8%) | 991 (90.3%) | 0.05 |
| Lab result number-Serum sodium mean (only > 90 | | | | | | | | | | | | |
| and < 190 included) | 93 | 117 | | 5 | 6 | | N/A | N/A | | 98 | 123 | |
| mean (sd) | 140.34 (2.66) | 140.63 (2.25) | -0.12 | 139.70 (3.42) | 139.19 (2.10) | 0.18 | N/A | N/A | #VALUE! | 140.31 (2.71) | 140.56 (2.25) | -0.10 |
| Missing; n (%) | 294 (76.0%) | 270 (69.8%) | 0.14 | 706 (99.3%) | 705 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 1,000 (91.1%) | 975 (88.8%) | 0.08 |
| Lab result number- Albumin mean (only >0 and <=10 | | , , | | • | | | | | | . , , | , , | |
| included) | 87 | 117 | | 4 | 3 | | N/A | N/A | | 91 | 120 | |
| mean (sd) | 4.11 (0.38) | 4.20 (0.37) | -0.24 | 4.20 (0.42) | 3.90 (0.35) | 0.78 | N/A | N/A | #VALUE! | 4.11 (0.38) | 4.19 (0.37) | -0.21 |
| Missing; n (%) | 300 (77.5%) | 270 (69.8%) | 0.18 | 707 (99.4%) | 708 (99.6%) | -0.03 | N/A | N/A | #VALUE! | 1,007 (91.7%) | 978 (89.1%) | 0.09 |
| Lab result number- Glucose (fasting or random) mean | | () | | (, | ( , | | | | | -/ (/ | ( | |
| (only 10-1000 included) | 93 | 117 | | 4 | 7 | | N/A | N/A | | 97 | 124 | |
| mean (sd) | 108.39 (28.61) | 102.85 (22.79) | 0.21 | 151.62 (87.96) | 116.12 (16.32) | 0.56 | N/A | N/A | #VALUE! | 110.17 (32.37) | 103.60 (22.61) | 0.24 |
| Missing: n (%) | 294 (76.0%) | 270 (69.8%) | 0.14 | 707 (99.4%) | 704 (99.0%) | 0.04 | N/A | N/A | #VALUE! | 1,001 (91.2%) | 974 (88.7%) | 0.08 |
| Lab result number- Potassium mean (only 1-7 | 254 (70.0%) | 270 (05.6%) | 0.14 | 707 (55.470) | 704 (55.0%) | 0.04 | N/A | N/A | #VALUE: | 1,001 (51.270) | 374 (00.770) | 0.08 |
| included) | 98 | 124 | | - | 6 | | N/A | N/A | | 103 | 130 | |
| mean (sd) | 4.27 (0.40) | 4.34 (0.43) | -0.17 | 4.15 (0.42) | 4.30 (0.28) | -0.42 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 4.26 (0.40) | 4.34 (0.43) | -0.19 |
| Missing; n (%) | 289 (74.7%) | 263 (68.0%) | 0.15 | 706 (99.3%) | 705 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 995 (90.6%) | 968 (88.2%) | 0.08 |
| Comorbidity Scores | | | | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 v2 | | | | | | | | | | | | |
| mean (sd) | 2.03 (2.16) | 1.85 (2.14) | 0.08 | 1.31 (1.94) | 1.38 (1.86) | -0.04 | 260.68 (376.81) | 243.96 (379.78) | 0.04 | 154.32 (289.39) | 144.46 (291.67) | 0.03 |
| Non-Frailty; n (%) | 193 (49.9%) | 182 (47.0%) | 0.06 | 311 (43.7%) | 286 (40.2%) | 0.07 | 35 (2.2%) | 33 (2.1%) | 0.01 | 539 (20.1%) | 501 (18.7%) | 0.04 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | | | | | _ | |
| mean (sd) | 0.18 (0.07) | 0.17 (0.07) | 0.14 | 0.15 (0.06) | 0.15 (0.05) | 0.00 | 0.09 (0.07) | 0.08 (0.07) | 0.14 | 0.12 (0.07) | 0.11 (0.07) | 0.14 |
| Healthcare Utilization | | | | | | | | | | | | |
| Any hospitalization; n (%) | 171 (44.2%) | 195 (50.4%) | -0.12 | 307 (43.2%) | 305 (42.9%) | 0.01 | 745 (47.2%) | 818 (51.9%) | -0.09 | 1,223 (45.7%) | 1,318 (49.3%) | -0.07 |
| Any hospitalization within prior 30 days; n (%) | 149 (38.5%) | 165 (42.6%) | -0.08 | 263 (37.0%) | 261 (36.7%) | 0.01 | 560 (35.5%) | 632 (40.1%) | -0.09 | 972 (36.3%) | 1058 (39.6%) | -0.07 |
| Any hospitalization during prior 31-180 days; n (%) | 39 (10.1%) | 39 (10.1%) | 0.00 | 62 (8.7%) | 62 (8.7%) | 0.00 | 295 (18.7%) | 267 (16.9%) | 0.05 | 396 (14.8%) | 368 (13.8%) | 0.03 |
| Internal medicine/family medicine visits; n (%) | 317 (81.9%) | 322 (83.2%) | -0.03 | 542 (76.2%) | 518 (72.9%) | 0.08 | 1,399 (88.7%) | 1,410 (89.4%) | -0.02 | 2258 (84.4%) | 2250 (84.1%) | 0.01 |
| Internal medicine/family medicine visits (30 days | (/ | () | | () | () | | _,=== (==:::-, | -, ( | | | | |
| prior) v2; n (%) | 272 (70.3%) | 277 (71.6%) | -0.03 | 426 (59.9%) | 412 (57.9%) | 0.04 | 1,152 (73.1%) | 1,210 (76.7%) | -0.08 | 1850 (69.2%) | 1899 (71.0%) | -0.04 |
| Internal medicine/family medicine visits (31 to 180 | (, 0.3,0) | (, 1.0,0) | 3.03 | .== (55.570) | (57.570) | 3.04 | -, (, 3.2,0) | -, (, 0., ,0) | 0.00 | (03.270) | (, 1.0,0) | 0.04 |
| days prior) v2; n (%) | 240 (62.0%) | 237 (61.2%) | 0.02 | 428 (60.2%) | 397 (55.8%) | 0.09 | 1,163 (73.7%) | 1,143 (72.5%) | 0.03 | 1831 (68.4%) | 1777 (66.4%) | 0.04 |
| Cardiologist visit; n (%) | 192 (49.6%) | 194 (50.1%) | -0.01 | 151 (21.2%) | 165 (23.2%) | -0.05 | 831 (52.7%) | 841 (53.3%) | -0.01 | 1174 (43.9%) | 1200 (44.9%) | -0.02 |
| Number of Cardiologist visits (30 days prior); n (%) | 152 (39.3%) | 157 (40.6%) | -0.01 | 105 (14.8%) | 115 (16.2%) | -0.04 | 580 (36.8%) | 612 (38.8%) | -0.01 | 837 (31.3%) | 884 (33.0%) | -0.02 |
| | 132 (33.3 /0) | 137 (40.0%) | -0.03 | 103 (14.070) | 113 (10.2%) | -0.04 | 300 (30.070) | 012 (30.0%) | -0.04 | 03/(31.3%) | 004 (33.0%) | -0.04 |
| Number of Cardiologist visits (31 to 180 days prior); | 97/22 59/\ | 77 (10 00/) | 0.06 | 77 /40 00/\ | 06 (43 40/) | -0.04 | 402 (24 20/) | 472 /20 00/1 | 0.03 | CEC (24 E0/) | 636 (33.00/) | 0.02 |
| n (%) | 87 (22.5%) | 77 (19.9%) | | 77 (10.8%) | 86 (12.1%) | | 492 (31.2%) | 473 (30.0%) | 0.03 | 656 (24.5%) | 636 (23.8%) | |
| Electrocardiogram v2; n (%) | 217 (56.1%) | 217 (56.1%) | 0.00 | 258 (36.3%) | 278 (39.1%) | -0.06 | 930 (59.0%) | 988 (62.7%) | -0.08 | 1405 (52.5%) | 1483 (55.4%) | -0.06 |
| Use of glucose test strips; n (%) | 3 (0.8%) | 5 (1.3%) | -0.05 | 5 (0.7%) | 2 (0.3%) | 0.06 | 21 (1.3%) | 20 (1.3%) | 0.00 | 29 (1.1%) | 27 (1.0%) | 0.01 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| number of different/distinct medication | | | | | | | | | | | | |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 7.87 (4.99) | 7.80 (5.14) | 0.01 | 7.50 (4.78) | 7.33 (4.83) | 0.04 | 9.41 (5.32) | 9.31 (4.98) | 0.02 | 8.68 (5.13) | 8.57 (4.96) | 0.02 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 0.59 (0.86) | 0.59 (0.67) | 0.00 | 0.51 (0.66) | 0.49 (0.64) | 0.03 | 0.64 (0.83) | 0.67 (0.83) | -0.04 | 0.60 (0.79) | 0.61 (0.76) | -0.01 |

| Number of hospital days | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| number of nospital days<br>mean (sd) | 2.26 (3.74) | 2.31 (3.52) | -0.01 | 2.04 (3.34) | 1.95 (4.05) | 0.02 | 2.60 (3.95) | 2.75 (4.26) | -0.04 | 2.40 (3.77) | 2.47 (4.11) | -0.02 |
| Number of Emergency Department (ED) visits v3 | 2.20 (3.74) | 2.51 (5.52) | 0.01 | 2.04 (3.54) | 1.55 (4.05) | 0.02 | 2.00 (3.33) | 2.75 (4.20) | 0.0-1 | 2.40 (3.77) | 2.47 (4.22) | 0.02 |
| mean (sd) | 1.58 (2.00) | 1.50 (2.10) | 0.04 | 1.08 (2.71) | 1.11 (2.83) | -0.01 | 1.68 (2.86) | 1.60 (2.03) | 0.03 | 1.51 (2.71) | 1.46 (2.28) | 0.02 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.75 (4.79) | 5.44 (4.65) | 0.07 | 4.93 (4.40) | 4.74 (4.30) | 0.04 | 13.36 (17.22) | 13.26 (15.82) | 0.01 | 10.02 (13.54) | 9.86 (12.48) | 0.01 |
| Number of internal medicine/family medicine visits | 0.00(44.20) | 0.50 (43.00) | | 5 20 (40 50) | 5 50 (0 54) | 0.07 | 40.45 (40.70) | 0.20 (40.20) | 0.00 | 0.03 (43.00) | 0.42 (40.50) | 0.07 |
| mean (sd) | 8.98 (11.38) | 8.50 (12.80) | 0.04 | 6.20 (10.58) | 5.50 (9.54) | 0.07 | 10.15 (12.72) | 9.20 (10.29) | 0.08 | 8.93 (12.00) | 8.12 (10.50) | 0.07 |
| Number of Cardiologist visits<br>mean (sd) | 1.89 (3.50) | 1.85 (3.24) | 0.01 | 0.71 (2.35) | 0.81 (2.37) | -0.04 | 2.45 (5.12) | 2.49 (4.57) | -0.01 | 1.91 (4.32) | 1.95 (3.92) | -0.01 |
| Number electrocardiograms received v2 | 1.05 (5.50) | 1.03 (3.24) | 0.01 | 0.71 (2.33) | 0.61(2.37) | -0.04 | 2.43 (3.12) | 2.45 (4.57) | -0.01 | 1.51 (4.52) | 1.55 (5.52) | -0.01 |
| mean (sd) | 1.40 (2.09) | 1.35 (1.81) | 0.03 | 0.70 (1.26) | 0.76 (1.18) | -0.05 | 1.53 (2.22) | 1.50 (1.85) | 0.01 | 1.29 (1.99) | 1.28 (1.69) | 0.01 |
| Number of HbA1c tests ordered | | . , | | | | | , , | | | | | |
| mean (sd) | 0.28 (0.57) | 0.29 (0.63) | -0.02 | 0.17 (0.44) | 0.18 (0.46) | -0.02 | 0.38 (0.69) | 0.38 (0.69) | 0.00 | 0.31 (0.62) | 0.31 (0.63) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.10 (0.52) | 0.18 (1.03) | -0.10 | 0.15 (0.75) | 0.12 (0.46) | 0.05 | 0.21 (2.00) | 0.16 (0.60) | 0.03 | 0.18 (1.60) | 0.15 (0.65) | 0.02 |
| Number of lipid tests ordered<br>mean (sd) | 0.45 (0.65) | 0.48 (0.69) | -0.04 | 0.27 (0.56) | 0.30 (0.62) | -0.05 | 0.55 (0.69) | 0.54 (0.72) | 0.01 | 0.46 (0.65) | 0.47 (0.69) | -0.01 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | 0.43 (0.03) | 0.48 (0.05) | -0.04 | 0.27 (0.30) | 0.30 (0.02) | -0.03 | 0.55 (0.05) | 0.34 (0.72) | 0.01 | 0.40 (0.03) | 0.47 (0.03) | -0.01 |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 10.88 (13.19) | 10.12 (11.25) | 0.06 | 5.87 (8.87) | 5.35 (7.73) | 0.06 | 12.82 (13.12) | 12.69 (12.90) | 0.01 | 10.69 (12.15) | 10.37 (11.50) | 0.03 |
| For PS | | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 9 (2.3%) | 7 (1.8%) | 0.04 | 12 (1.7%) | 9 (1.3%) | 0.03 | 42 (2.7%) | 33 (2.1%) | 0.04 | 63 (2.4%) | 49 (1.8%) | 0.04 |
| Major trauma potentially causing prolonged immobili | 32 (8.3%) | 29 (7.5%) | 0.03 | 46 (6.5%) | 49 (6.9%) | -0.02 | 118 (7.5%) | 109 (6.9%) | 0.02 | 46 (6.5%) | 49 (6.9%) | -0.02 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 19 (4.9%) | 31 (8.0%) | -0.13 | 57 (8.0%) | 90 (12.7%) | -0.15 | 132 (8.4%) | 167 (10.6%) | -0.08 | 208 (7.8%) | 288 (10.8%) | -0.10 |
| Occurrence of BUN tests ordered (for PS); n (%) | 7 (1.8%) | 13 (3.4%) | -0.10 | 22 (3.1%) | 37 (5.2%) | -0.11 | 68 (4.3%) | 86 (5.5%) | -0.06 | 97 (3.6%) | 136 (5.1%) | -0.07 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | | , , | | | . , | | | | |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Acute kidney injury; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0!<br>-0.10 | 1 (0.1%) | 1 (0.1%) | 0.00<br>0.02 | 1 (0.1%) | 3 (0.2%) | -0.03<br>0.00 | 1 (0.1%) | 1 (0.1%) | 0.00<br>-0.01 |
| Bladder stones+Kidney stones (for PS); n (%) Alcohol abuse or dependence+Drug abuse or | 6 (1.6%) | 12 (3.1%) | -0.10 | 13 (1.8%) | 11 (1.5%) | 0.02 | 37 (2.3%) | 37 (2.3%) | 0.00 | 56 (2.1%) | 60 (2.2%) | -0.01 |
| dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! |
| Other atherosclerosis+Cardiac conduction | | | | | , , | | | . , | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 86 (22.2%) | 91 (23.5%) | -0.03 | 98 (13.8%) | 107 (15.0%) | -0.03 | 357 (22.6%) | 374 (23.7%) | -0.03 | 541 (20.2%) | 572 (21.4%) | -0.03 |
| Previous cardiac procedure (CABG or PTCA or Stent) + | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 14 (3.6%) | 10 (2.6%) | 0.06 | 11 (1.5%) | 11 (1.5%) | 0.00 | 118 (7.5%) | 120 (7.6%) | 0.00 | 143 (5.3%) | 141 (5.3%) | 0.00 |
| Diabetes with complication; n (%) Delirium + Psychosis (for PS); n (%) | 18 (4.7%)<br>16 (4.1%) | 18 (4.7%)<br>14 (3.6%) | 0.00 | 18 (2.5%)<br>14 (2.0%) | 15 (2.1%)<br>14 (2.0%) | 0.03 | 125 (7.9%)<br>86 (5.5%) | 123 (7.8%)<br>82 (5.2%) | 0.00<br>0.01 | 18 (2.5%)<br>116 (4.3%) | 15 (2.1%)<br>110 (4.1%) | 0.03<br>0.01 |
| Any use of Meglitinides (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 5 (0.3%) | 2 (0.1%) | 0.01 | 5 (0.2%) | 2 (0.1%) | 0.01 |
| Any use of AGIs (for PS): n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 0 (0.0%) | 0.04 | 1 (0.0%) | 0 (0.0%) | #DIV/0! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of thiazide; n (%) | 31 (8.0%) | 36 (9.3%) | -0.05 | 33 (4.6%) | 34 (4.8%) | -0.01 | 179 (11.4%) | 166 (10.5%) | 0.03 | 243 (9.1%) | 236 (8.8%) | 0.01 |
| Use of beta blockers; n (%) | 85 (22.0%) | 86 (22.2%) | 0.00 | 136 (19.1%) | 130 (18.3%) | 0.02 | 607 (38.5%) | 577 (36.6%) | 0.04 | 828 (31.0%) | 793 (29.6%) | 0.03 |
| Use of calcium channel blockers; n (%) | 73 (18.9%) | 66 (17.1%) | 0.05 | 105 (14.8%) | 88 (12.4%) | 0.07 | 353 (22.4%) | 363 (23.0%) | -0.01 | 531 (19.9%) | 517 (19.3%) | 0.02 |
| All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy: n (%) | 30 (7.8%)<br>14 (3.6%) | 27 (7.0%)<br>9 (2.3%) | 0.03 | 61 (8.6%)<br>12 (1.7%) | 58 (8.2%)<br>12 (1.7%) | 0.01<br>0.00 | 208 (13.2%)<br>56 (3.6%) | 228 (14.5%)<br>52 (3.3%) | -0.04<br>0.02 | 299 (11.2%)<br>82 (3.1%) | 313 (11.7%)<br>73 (2.7%) | -0.02<br>0.02 |
| Use of Low Intensity Statins; n (%) | 76 (19.6%) | 70 (18.1%) | 0.08 | 87 (12.2%) | 82 (11.5%) | 0.00 | 408 (25.9%) | 391 (24.8%) | 0.02 | 571 (21.3%) | 543 (20.3%) | 0.02 |
| Use of High Intensity Statins; n (%) | 54 (14.0%) | 49 (12.7%) | 0.04 | 65 (9.1%) | 72 (10.1%) | -0.03 | 235 (14.9%) | 259 (16.4%) | -0.04 | 354 (13.2%) | 380 (14.2%) | -0.03 |
| Malignant hypertension; n (%) | 3 (0.8%) | 3 (0.8%) | 0.00 | 88 (12.4%) | 64 (9.0%) | 0.11 | 191 (12.1%) | 170 (10.8%) | 0.04 | 282 (10.5%) | 237 (8.9%) | 0.05 |
| Cardiovascular stress test; n (%) | 4 (1.0%) | 2 (0.5%) | 0.06 | 4 (0.6%) | 3 (0.4%) | 0.03 | 12 (0.8%) | 14 (0.9%) | -0.01 | 20 (0.7%) | 19 (0.7%) | 0.00 |
| Echocardiogram; n (%) | 121 (31.3%) | 127 (32.8%) | -0.03 | 160 (22.5%) | 167 (23.5%) | -0.02 | 458 (29.0%) | 531 (33.7%) | -0.10 | 739 (27.6%) | 825 (30.8%) | -0.07 |
| Number of BNP tests | | | | | | | | | | | | |
| mean (sd) | 0.14 (0.44) | 0.11 (0.37) | 0.07 | 0.06 (0.28) | 0.09 (0.31) | -0.10 | 0.14 (0.45) | 0.15 (0.50) | -0.02 | 0.12 (0.41) | 0.13 (0.44) | 0.00 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, M | Ivoglobin CDK) | | | | | | | | | | | |
| mean (sd) | 0.38 (1.02) | 0.43 (1.63) | -0.04 | 0.21 (0.80) | 0.25 (0.75) | -0.05 | 0.26 (0.61) | 0.26 (0.59) | 0.00 | 0.26 (0.73) | 0.28 (0.86) | 0.00 |
| • • | | . , | | | | | , , | | | | | |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.01 (0.10) | 0.00 (0.05) | 0.13 | 0.00 (0.04) | 0.00 (0.05) | 0.00 | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.04) | 0.00 (0.03) | 0.00 |
| N of days on antihypertensive medications during baselin | ne. | | | | | | | | | | | |
| mean (sd) | 67.65 (79.23) | 71.62 (80.47) | -0.05 | 55.48 (76.62) | 52.37 (73.66) | 0.04 | 104.43 (78.04) | 104.63 (78.56) | 0.00 | 86.10 (77.84) | 85.96 (77.57) | 0.00 |
| N of days in database anytime prior | 07.03 (73.23) | 71.02 (00.47) | 0.03 | 33.40 (70.02) | 32.37 (73.00) | 0.04 | 104.45 (70.04) | 104.03 (70.30) | 0.00 | 00.10 (77.04) | 03.30 (77.37) | 0.00 |
| mean (sd) | 1,830.11 (1,432.42) | 1,885.97 (1,492.49) | -0.04 | 2,212.30 (1,514.35) | 2,067.60 (1,411.97) | 0.10 | 779.13 (547.37) | 759.93 (521.03) | 0.04 | 1312.11 (1040.43) | 1270.41 (1005.81) | 0.00 |
| | | • | | | | | | | | • | | |
| Mean Copay for per prescription cost (charges in U.S. \$) ( | | | | | | | | | | | | |
| mean (sd) | 25.11 (47.24) | 29.63 (62.90) | -0.08 | 14.39 (27.22) | 14.21 (21.16) | 0.01 | 106.57 (105.54) | 105.71 (103.82) | 0.01 | 70.28 (84.20) | 70.38 (83.95) | 0.00 |
| Missing; n (%) | 29 (7.5%)<br>19 (4.9%) | 31 (8.0%)<br>13 (3.4%) | -0.02<br>0.08 | 66 (9.3%)<br>29 (4.1%) | 71 (10.0%)<br>21 (3.0%) | -0.02<br>0.06 | 75 (4.8%)<br>52 (3.3%) | 65 (4.1%)<br>52 (3.3%) | 0.03 | 170 (6.4%)<br>100 (3.7%) | 167 (6.2%)<br>86 (3.2%) | 0.01 |
| Colonoscopy; n (%) Fecal occult blood (FOB) test; n (%) | 19 (4.9%)<br>9 (2.3%) | 13 (3.4%) | -0.03 | 29 (4.1%)<br>30 (4.2%) | 21 (3.0%) | 0.05 | 52 (3.3%)<br>48 (3.0%) | 52 (3.3%)<br>43 (2.7%) | 0.00 | 87 (3.3%) | 86 (3.2%)<br>77 (2.9%) | 0.03 |
| Flu vaccine: n (%) | 67 (17.3%) | 73 (18.9%) | -0.03 | 71 (10.0%) | 57 (8.0%) | 0.03 | 440 (27.9%) | 449 (28.5%) | -0.01 | 578 (21.6%) | 579 (21.6%) | 0.02 |
| Mammogram; n (%) | 22 (5.7%) | 31 (8.0%) | -0.09 | 59 (8.3%) | 62 (8.7%) | -0.01 | 174 (11.0%) | 173 (11.0%) | 0.00 | 255 (9.5%) | 266 (9.9%) | -0.01 |
| Pap smear; n (%) | 19 (4.9%) | 21 (5.4%) | -0.02 | 41 (5.8%) | 42 (5.9%) | 0.00 | 39 (2.5%) | 42 (2.7%) | -0.01 | 99 (3.7%) | 105 (3.9%) | -0.01 |
| Pneumonia vaccine; n (%) | 78 (20.2%) | 86 (22.2%) | -0.05 | 99 (13.9%) | 81 (11.4%) | 0.08 | 413 (26.2%) | 440 (27.9%) | -0.04 | 590 (22.1%) | 607 (22.7%) | -0.01 |

| PSA test or Prostate exam for DRE; n (%) | 41 (10.6%) | 43 (11.1%) | -0.02 | 58 (8.2%) | 52 (7.3%) | 0.03 | 202 (12.8%) | 205 (13.0%) | -0.01 | 301 (11.3%) | 300 (11.2%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Bone mineral density; n (%) | 4 (1.0%) | 11 (2.8%) | -0.13 | 4 (0.6%) | 6 (0.8%) | -0.02 | 86 (5.5%) | 74 (4.7%) | 0.04 | 94 (3.5%) | 91 (3.4%) | 0.01 |
| ** * * | | | | | | | | | | | | |
| Use of CNS stimulants; n (%) | 5 (1.3%) | 6 (1.6%) | -0.03 | 3 (0.4%) | 9 (1.3%) | -0.10 | 6 (0.4%) | 5 (0.3%) | 0.02 | 14 (0.5%) | 20 (0.7%) | -0.03 |
| Use of estrogens, progestins, androgens; n (%) | 23 (5.9%) | 27 (7.0%) | -0.04 | 84 (11.8%) | 89 (12.5%) | -0.02 | 52 (3.3%) | 62 (3.9%) | -0.03 | 159 (5.9%) | 178 (6.7%) | -0.03 |
| Use of Angiogenesis inhibitors: n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.1%) | 0 (0.0%) | 0.04 | 2 (0.1%) | 0 (0.0%) | 0.04 |
| 0.00 | | | | | | | | | | , | | |
| Use of Oral Immunosuppressants; n (%) | 0 (0.0%) | 1 (0.3%) | -0.08 | 0 (0.0%) | 2 (0.3%) | -0.08 | 1 (0.1%) | 2 (0.1%) | 0.00 | 1 (0.0%) | 5 (0.2%) | -0.06 |
| Use of fondaparinux or Bivalirudin; n (%) | 5 (1.3%) | 4 (1.0%) | 0.03 | 10 (1.4%) | 7 (1.0%) | 0.04 | 7 (0.4%) | 6 (0.4%) | 0.00 | 22 (0.8%) | 17 (0.6%) | 0.02 |
| Use of other direct thrombin inhibitors (lepirudin, des | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 2 (0.5%) | 1 (0.3%) | 0.03 | 3 (0.4%) | 2 (0.3%) | 0.02 | 0 (0.0%) | 1 (0.1%) | -0.04 | 5 (0.2%) | 4 (0.1%) | 0.03 |
| Use of Ticagrelor; n (%) | 2 (0.5%) | 1 (0.3%) | 0.03 | 4 (0.6%) | 4 (0.6%) | 0.00 | 8 (0.5%) | 5 (0.3%) | 0.03 | 14 (0.5%) | 10 (0.4%) | 0.01 |
| Number of D-dimer tests | | | | | | | | | | | | |
| | 0.25 (0.62) | 0.21 (0.52) | 0.07 | 0.13 (0.45) | 0.14 (0.40) | -0.02 | 0.13 (0.40) | 0.14 (0.41) | -0.02 | 0.45 (0.45) | 0.15 (0.43) | 0.00 |
| mean (sd) | 0.25 (0.62) | 0.21 (0.52) | 0.07 | 0.13 (0.45) | 0.14 (0.40) | -0.02 | 0.13 (0.40) | 0.14 (0.41) | -0.02 | 0.15 (0.45) | 0.15 (0.43) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | | |
| mean (sd) | 0.09 (0.37) | 0.10 (0.39) | -0.03 | 0.10 (0.51) | 0.08 (0.34) | 0.05 | 0.12 (0.53) | 0.13 (0.49) | -0.02 | 0.11 (0.50) | 0.11 (0.44) | 0.00 |
| Number of PT or aPTTt tests | (, | (, | | () | (, | | | () | **** | () | (, | |
| mean (sd) | 0.95 (1.85) | 0.83 (1.60) | 0.07 | 0.58 (1.22) | 0.57 (1.18) | 0.01 | 0.54 (1.23) | 0.52 (1.23) | 0.02 | 0.61 (1.34) | 0.58 (1.28) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! |
| | 0.00 (0.00) | 0.00 (0.00) | #D14/0: | 0.00 (0.00) | 0.00 (0.00) | #DIV/O: | 0.00 (0.00) | 0.00 (0.00) | #DIV/0: | 0.00 (0.00) | 0.00 (0.00) | #514/0: |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| mean (sd) | 2.58 (1.08) | 2.53 (1.04) | 0.05 | 2.14 (1.03) | 2.08 (1.00) | 0.06 | 3.32 (0.79) | 3.29 (0.80) | 0.04 | 2.90 (0.90) | 2.86 (0.89) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | | |
| mean (sd) | 14.58 (14.48) | 14.35 (17.58) | 0.01 | 10.92 (10.62) | 10.45 (11.54) | 0.04 | 17.57 (14.96) | 17.16 (15.12) | 0.03 | 15.37 (13.87) | 14.97 (14.66) | 0.00 |
| () | 14.58 (14.48) | 14.35 (17.58) | 0.01 | 10.92 (10.62) | 10.45 (11.54) | 0.04 | 17.57 (14.96) | 17.16 (15.12) | 0.03 | 15.57 (15.67) | 14.97 (14.00) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 3.58 (7.51) | 3.57 (5.26) | 0.00 | 3.14 (5.30) | 3.04 (3.22) | 0.02 | 3.78 (6.68) | 3.73 (4.80) | 0.01 | 3.58 (6.48) | 3.52 (4.51) | 0.00 |
| | 15 (3.9%) | 11 (2.8%) | 0.06 | | 14 (2.0%) | 0.03 | 123 (7.8%) | 99 (6.3%) | 0.06 | 155 (5.8%) | 124 (4.6%) | 0.05 |
| Use of clopidogrel ; n (%) | | | | 17 (2.4%) | | | | | | | | |
| Systemic embolism; n (%) | 6 (1.6%) | 4 (1.0%) | 0.05 | 20 (2.8%) | 16 (2.3%) | 0.03 | 22 (1.4%) | 24 (1.5%) | -0.01 | 48 (1.8%) | 44 (1.6%) | 0.02 |
| DVT; n (%) | 284 (73.4%) | 274 (70.8%) | 0.06 | 539 (75.8%) | 520 (73.1%) | 0.06 | 1,260 (79.9%) | 1,238 (78.5%) | 0.03 | 2083 (77.9%) | 2032 (76.0%) | 0.05 |
| Post-thrombotic syndrome; n (%) | 7 (1.8%) | 4 (1.0%) | 0.07 | 5 (0.7%) | 4 (0.6%) | 0.01 | 6 (0.4%) | 7 (0.4%) | 0.00 | 5 (0.7%) | 4 (0.6%) | 0.01 |
| PE; n (%) | 166 (42.9%) | 183 (47.3%) | -0.09 | 318 (44.7%) | 328 (46.1%) | -0.03 | 559 (35.4%) | 608 (38.6%) | -0.07 | 1043 (39.0%) | 1119 (41.8%) | -0.06 |
| Coagulation defects; n (%) | 22 (5.7%) | 16 (4.1%) | 0.07 | 16 (2.3%) | 20 (2.8%) | -0.03 | 37 (2.3%) | 32 (2.0%) | 0.02 | 16 (2.3%) | 20 (2.8%) | -0.03 |
| Diabetes: 1 inpatient or 2 outpatient claims within 18 | 57 (14.7%) | 47 (12.1%) | 0.08 | 69 (9.7%) | 67 (9.4%) | 0.01 | 356 (22.6%) | 352 (22.3%) | 0.01 | 482 (18.0%) | 466 (17.4%) | 0.02 |
| Diabetes. 1 inpatient of 2 outpatient claims within 10 | 37 (14.770) | 47 (12.170) | 0.00 | 05 (5.770) | 07 (5.470) | 0.01 | 330 (22.0%) | 332 (22.370) | 0.01 | 402 (10.070) | 400 (17.470) | 0.02 |
| Intracranial or retroperitoneal hemorrhage: 1 inpaties | 0 (0.0%) | 1 (0.3%) | -0.08 | 2 (0.3%) | 1 (0.1%) | 0.04 | 3 (0.2%) | 2 (0.1%) | 0.03 | 5 (0.2%) | 4 (0.1%) | 0.03 |
| Peptic Ulcer Disease; n (%) | 68 (17.6%) | 67 (17.3%) | 0.01 | 96 (13.5%) | 95 (13.4%) | 0.00 | 317 (20.1%) | 332 (21.1%) | -0.02 | 481 (18.0%) | 494 (18.5%) | -0.01 |
| Upper GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! |
| Lower/ unspecified GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Urogenital bleed; n (%) | 1 (0.3%) | 2 (0.5%) | -0.03 | 6 (0.8%) | 7 (1.0%) | -0.02 | 14 (0.9%) | 11 (0.7%) | 0.02 | 21 (0.8%) | 20 (0.7%) | 0.01 |
| Other bleeds; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 2 (0.3%) | -0.08 | 8 (0.5%) | 6 (0.4%) | 0.01 | 8 (0.3%) | 8 (0.3%) | 0.00 |
| Prior cancer; n (%) | 49 (12.7%) | 45 (11.6%) | 0.03 | 67 (9.4%) | 65 (9.1%) | 0.01 | 310 (19.7%) | 273 (17.3%) | 0.06 | 426 (15.9%) | 383 (14.3%) | 0.04 |
| Antibiotics; n (%) | 166 (42.9%) | 174 (45.0%) | #DIV/0! | 344 (48.4%) | 315 (44.3%) | #DIV/0! | 838 (53.1%) | 829 (52.6%) | #DIV/0! | 344 (48.4%) | 315 (44.3%) | 0.00 |
| Aspirin: n (%) | 4 (1.0%) | 6 (1.6%) | -0.05 | 26 (3.7%) | 19 (2.7%) | 0.06 | 12 (0.8%) | 7 (0.4%) | 0.05 | 42 (1.6%) | 32 (1.2%) | 0.03 |
| | | - ' - ' ' | | | - ' ' | | , | , | | , | | |
| Aspirin/dipyridamole; n (%) | 2 (0.5%) | 2 (0.5%) | 0.00 | 5 (0.7%) | 2 (0.3%) | 0.06 | 8 (0.5%) | 4 (0.3%) | 0.03 | 15 (0.6%) | 8 (0.3%) | 0.04 |
| Other antiplatelet agents; n (%) | 1 (0.3%) | 1 (0.3%) | 0.00 | 0 (0.0%) | 1 (0.1%) | -0.04 | 6 (0.4%) | 11 (0.7%) | -0.04 | 7 (0.3%) | 13 (0.5%) | -0.03 |
| PGP inhibitors; n (%) | 78 (20.2%) | 86 (22.2%) | -0.05 | 167 (23.5%) | 152 (21.4%) | 0.05 | 446 (28.3%) | 438 (27.8%) | 0.01 | 691 (25.8%) | 676 (25.3%) | 0.01 |
| Other gastroprotective agents; n (%) | 4 (1.0%) | 4 (1.0%) | 0.00 | | 9 (1.3%) | -0.05 | 28 (1.8%) | 28 (1.8%) | 0.00 | 38 (1.4%) | 41 (1.5%) | -0.01 |
| | 4 (1.0%) | 4 (1.0%) | 0.00 | 6 (0.8%) | 9 (1.3%) | -0.05 | 28 (1.8%) | 28 (1.8%) | 0.00 | 38 (1.4%) | 41 (1.5%) | -0.01 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.45 (0.65) | 0.48 (0.69) | -0.04 | 0.27 (0.56) | 0.30 (0.62) | -0.05 | 0.58 (0.77) | 0.57 (0.79) | 0.01 | 0.48 (0.70) | 0.49 (0.73) | 0.00 |
| Proton pump inhibitor; n (%) | 76 (19.6%) | 67 (17.3%) | 0.06 | 138 (19.4%) | 126 (17.7%) | 0.04 | 437 (27.7%) | 435 (27.6%) | 0.00 | 651 (24.3%) | 628 (23.5%) | 0.02 |
| | , | | | | | | | | | | | |
| H2 receptor antagonist; n (%) | 8 (2.1%) | 9 (2.3%) | -0.01 | 25 (3.5%) | 24 (3.4%) | 0.01 | 87 (5.5%) | 87 (5.5%) | 0.00 | 120 (4.5%) | 120 (4.5%) | 0.00 |
| Vitamin K therapy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.1%) | 1 (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! |
| Number of INR (prothrombin) tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.77 (1.61) | 0.47 (0.88) | 0.23 | 0.47 (1.08) | 0.35 (0.78) | 0.13 | 0.51 (1.21) | 0.46 (1.15) | 0.04 | 0.54 (1.24) | 0.43 (1.03) | 0.00 |
| | , | , | | | | | | | | | | |
| Treating prescriber - Cardiologist; n (%) | 152 (39.3%) | 160 (41.3%) | -0.04 | 197 (27.7%) | 201 (28.3%) | -0.01 | 580 (36.8%) | 612 (38.8%) | -0.04 | 929 (34.7%) | 973 (36.4%) | -0.04 |
| Treating prescriber - Primary Care Physician; n (%) | 323 (83.5%) | 315 (81.4%) | 0.06 | 273 (38.4%) | 263 (37.0%) | 0.03 | 610 (38.7%) | 591 (37.5%) | 0.02 | 1206 (45.1%) | 1169 (43.7%) | 0.03 |
| Treating prescriber - Other; n (%) | 377 (97.4%) | 374 (96.6%) | 0.05 | 679 (95.5%) | 680 (95.6%) | 0.00 | 1.544 (97.9%) | 1.549 (98.2%) | -0.02 | 2600 (97.2%) | 2603 (97.3%) | -0.01 |
| Alpha blockers; n (%) | | 26 (6.7%) | 0.00 | 28 (3.9%) | 23 (3.2%) | 0.04 | 146 (9.3%) | 156 (9.9%) | -0.02 | 200 (7.5%) | 205 (7.7%) | -0.01 |
| | 26 (6.7%) | 26 (6.7%) | 0.00 | 28 (3.9%) | 23 (3.2%) | 0.04 | 146 (9.3%) | 156 (9.9%) | -0.02 | 200 (7.5%) | 205 (7.7%) | -0.01 |
| CHA2DS2 VASc score, 180 days, V | | | | | | | | | | | | |
| mean (sd) | 1.92 (1.42) | 1.89 (1.56) | 0.02 | 1.79 (1.72) | 1.73 (1.69) | 0.04 | 2.83 (1.59) | 2.80 (1.53) | 0.02 | 2.42 (1.60) | 2.38 (1.58) | 0.00 |
| Use of Prasugrel; n (%) | 2 (0.5%) | 1 (0.3%) | 0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.1%) | 1 (0.0%) | 0.04 |
| Ose of Frasugrer, if (76) | 2 (0.5%) | 1 (0.3%) | 0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/U: | 0 (0.0%) | 0 (0.0%) | #010/0: | 2 (0.1%) | 1 (0.0%) | 0.04 |
| Use of Loop Diuretics+other diuretics+other hyperten: | 57 (14.7%) | 55 (14.2%) | 0.01 | 68 (9.6%) | 65 (9.1%) | 0.02 | 367 (23.3%) | 362 (23.0%) | 0.01 | 492 (18.4%) | 482 (18.0%) | 0.01 |
| Commercial vs Medicare Advantage- Business Type Code - CO | RRECT ONE - OPTLIM | | | | | | 0 | 0 | | | | |
| | | 204 (71 71) | a | 4551 | 464 ( | | 3 | U | | 0.054/55.550 | 0.000 ( | |
| Commercial; n (%) | 188 (48.6%) | 201 (51.9%) | -0.07 | 166 (23.3%) | 161 (22.6%) | 0.02 | - | - | #VALUE! | 0,354 (32.2%) | 0,362 (33.0%) | -0.02 |
| Medicare Advantage; n (%) | 0,199 (51.4%) | 186 (48.1%) | 0.07 | 545 (76.7%) | 550 (77.4%) | -0.02 | - | - | #VALUE! | #VALUE! | 0,736 (67.0%) | #VALUE! |
| | • | | | | | | | | | | | |
| Commercial vs Medicare Advantage- Business Type Code | | | | | | | | | | | | |
| | 400 (:= ==::) | 204 (71 71) | a | | | m +++ · · · · · | | | | 400 (*** ****) | 204 (2 - 2 - 4) | |
| COM = COMMERCIAL; n (%) | 188 (48.6%) | 201 (51.9%) | -0.07 | - | - | #VALUE! | - | - | #VALUE! | 188 (48.6%) | 201 (51.9%) | -0.07 |
| MCR = MEDICARE; n (%) | 199 (51.4%) | 186 (48.1%) | 0.07 | - | | #VALUE! | - | | #VALUE! | 199 (51.4%) | 186 (48.1%) | 0.07 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | #VALUE! | | | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| co - medicald, ii (/a) | 0 (0.070) | 0 (0.070) | #DIV/0: | , | • | #VALUE: | 1 | • | #VALUE: | 0 (0.070) | 0 (0.070) | #DIV/U! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n ( | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | | | | | | | | | | | | |
| UNK = UNKNOWN (added in 2015); ii (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - 0 | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 | 0 | #VALUE! | - | - | #VALUE! | | | , |
| | 0 (0.0%)<br>-<br>- | 0 (0.0%)<br>-<br>- | #DIV/0! | -<br>0<br>402 (56.5%) | -<br>0<br>422 (59.4%) | #VALUE! | -<br>- | -<br>- | #VALUE! | 0 (0.0%)<br>402 (56.5%) | 0 (0.0%)<br>422 (59.4%) | #DIV/0! |

| 2 - Encounter; n (%) | - | | 143 (20.1%) | 128 (18.0%) | - | - | 143 (20.1%) | 128 (18.0%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| 3 - Medicare; n (%) | - | - | 159 (22.4%) | 147 (20.7%) | - | - | 159 (22.4%) | 147 (20.7%) | 0.00 |
| 4 - Medicare Encounter; n (%) | - | | 7 (1.0%) | 14 (2.0%) | - | - | 7 (1.0%) | 14 (2.0%) | 0.00 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (non- | -MSA) | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | | 494 (69.5%) | 517 (72.7%) | - | - | 494 (69.5%) | 517 (72.7%) | 0.00 |
| Rural; n (%) | - | | 57 (8.0%) | 46 (6.5%) | - | - | 57 (8.0%) | 46 (6.5%) | 0.00 |
| Unknown/Missing: n (%) | - | - | 160 (22.5%) | 148 (20.8%) | | | 160 (22.5%) | 148 (20.8%) | 0.00 |